# **Phase III Study of ASP015K**

-A randomized, double-blind, placebo-controlled confirmatory study of the safety and efficacy of ASP015K in patients with rheumatoid arthritis (RA) who had an inadequate response to DMARDs-

ISN/Protocol 015K-CL-RAJ3

ClinicalTrials.gov Identifier: NCT02308163

Date of Protocol: Version 5.0, dated 03 March 2017

Sponsor: Astellas Pharma Inc. (API)

2-5-1 Nihonbashi-Honcho, Chuo-ku, Tokyo

| Sponsor: Astellas Pharma Inc. | ISN/Protocol <015K-CL-RAJ3> |
|---|---|
| Protocol for Phase III Study of | of ASP015K |
| -A Randomized, Double-Blind, Placebo-Controlled Con<br>Efficacy of ASP015K in Patients with Rheumatoid Arth<br>Response to DMARDs- | ritis (RA) who Had an Inadequate |
| C., | |
| Sponsor: | |
| Astellas Pharma Inc. (AF | PI) |

ISN/Protocol: 015K-CL-RAJ3

Created 3 March 2017 (Ver. 5.0)

This confidential document is the property of the sponsor. No unpublished information contained in this document may be disclosed without prior written approval of the sponsor.

3 March 2017 Astellas 

# **Table of Contents**

| SIG | NATURE ······ | 8 |
|---|---|---|
| I. CONTACT DETAILS OF KEY SPONSOR'S PERSONNEL | | 9 |
| I. LIST OF ABBREVIATIONS AND DEFINITION OF KEY TERMS | | 1 |
| FLO | OW CHART AND SCHEDULE OF ASSESSMENTS | 30 |
| 1.2 | | |
| 1.2.1 | | |
| 1.2.2 | | |
| 1.2 | | |
| 1.2 | | |
| 1.2.3 | <b>.</b> | |
| 1.2.4 | • | |
| 1.3 | Summary of Key Safety Information for Study Drugs · | 44 |
| 1.4 | Risk-Benefit Assessment····· | 46 |
| STU | DY OBJECTIVE(S), DESIGN, AND VARIABLES | 48 |
| 2.1 | Study Objectives ····· | 48 |
| 2.2 | Study Design and Dose Rationale | 48 |
| 2.2.1 | Study Design · | 48 |
| 2.2.2 | | |
| 2.3 | | |
| 2.3.1 | Primary Variables ····· | 51 |
| 2.3.2 | Secondary Variables · | 51 |
| 2.3 | 2.2.1 Secondary Efficacy Variables · | 51 |
| 2.3 | · | |
| | • | |
| 2.3.3 | | |
| STU | DY POPULATION······ | 53 |
| | CON<br>LIS'<br>SYN<br>FLO<br>ACO<br>INT<br>1.1<br>1.2.2<br>1.2.3<br>1.2.4<br>1.3<br>1.4<br>STU<br>2.1<br>2.2<br>2.3.1<br>2.3.2<br>2.3.2<br>2.3<br>2.3.3<br>2.3.3 | CONTACT DETAILS OF KEY SPONSOR'S PERSONNEL LIST OF ABBREVIATIONS AND DEFINITION OF KEY TERMS SYNOPSIS FLOW CHART AND SCHEDULE OF ASSESSMENTS ACCEPTABLE RANGE OF SCHEDULE OF ASSESSMENTS INTRODUCTION 1.1 Background 1.2 Non-clinical and Clinical Data 1.2.1 Nonclinical Pharmacology and Safety Pharmacology 1.2.2 Pharmacokinetics and Pharmacodynamics 1.2.2.1 Nonclinical Pharmacokinetics and Pharmacodynamics 1.2.2.2 Clinical Pharmacokinetics and Pharmacodynamics 1.2.3 Toxicology 1.2.4 Efficacy 1.3 Summary of Key Safety Information for Study Drugs 1.4 Risk-Benefit Assessment STUDY OBJECTIVE(S), DESIGN, AND VARIABLES 2.1 Study Objectives 2.2 Study Design and Dose Rationale 2.2.1 Study Design 2.2.2 Dose Rationale 2.3.1 Primary Variables 2.3.2 Secondary Variables 2.3.2.1 Secondary Efficacy Variables 2.3.2.2 Safety Variables 2.3.2.3 Pharmacodynamics Variables 2.3.2.4 Pharmacodynamics Variables 2.3.2.5 Pharmacogenomics (Bio-Banking) [unique to Japan and Korea] |

| | 3.1 | Selection of Study Population · | 53 |
|---|---|---|---|
| | 3.2 | Inclusion Criteria · | 53 |
| | 3.3 | Exclusion Criteria · | 54 |
| | 3.4 | Discontinuation Criteria for Individual Subjects · | 58 |
| | 3.4.1 | Suspension, Interruption, and Resumption of the Study Drug or Reference Drug····· | 59 |
| | 3.4 | .1.1 Criteria for Suspension or Interruption of the Study Drug or Reference Drug · | 60 |
| 4 | STU | DY DRUGS OR REFERENCE DRUGS ······ | 61 |
| | 4.1 | Description of Study Drugs or Reference Drugs ····· | 61 |
| | 4.1.1 | Test Drug(s)····· | 61 |
| | 4.1.2 | Comparative Drug(s)····· | 61 |
| | 4.1.3 | Reference Drug(s) · | 61 |
| | 4.2 | Packaging and Labeling · | 62 |
| | 4.3 | Study/Reference Drug Handling · | 63 |
| | 4.4 | Blinding ····· | 63 |
| | 4.4.1 | Blinding Method····· | 63 |
| | 4.4.2 | Confirmation of the Indistinguishability of the Study Drugs | 64 |
| | 4.4.3 | Retention of the Assignment Schedule and Procedures for Treatment Code | |
| | | Breaking | |
| | 4.4.4 | Breaking the Treatment Code for Emergency ····· | |
| | 4.4.5 | Breaking the Treatment Code by the Sponsor · | |
| | 4.5 | Assignment and Allocation ····· | 65 |
| 5 | TRE | ATMENTS AND EVALUATION | 66 |
| | | Dosing and Administration of Study Drugs or Reference Drugs and Other Medications | 66 |
| | 5.1.1 | Dose/Dose Regimen and Administration Period ······ | |
| | 5.1.2 | Previous and Concomitant Medication (Drugs and Therapies) · | |
| | | .2.1 Previous Medication (Drugs and Therapies) | |
| | | .2.2 Concomitant Medication (Drugs and Therapies) | |
| | 5.1.3 | Treatment Compliance | |
| | 5.1.4 | Emergency Procedures and Management of Overdose ······ | |
| | 5.1.5 | Criteria for Continuation of Treatment ······ | |
| | 5.1.6 | Compliance Rules to be Observed by Subjects throughout the Study ······· | 76 |

| 5.2 | Demographics and Baseline Characteristics · | 77 |
|---|---|---|
| 5.2.1 | Demographics · | |
| 5.2.2 | Medical History····· | 77 |
| 5.2.3 | Diagnosis of the Target Disease, Severity, and Duration of Disease | 78 |
| 5.3 | Efficacy, Pharmacodynamics, and Pharmacokinetics Assessments······ | 78 |
| 5.3.1 | Efficacy Assessments · | 78 |
| 5.3 | .1.1 Tender and Swollen Joint Counts | 78 |
| 5.3 | .1.2 Assessment of Pain and Overall Assessment of Disease Activity · · · · | 79 |
| 5.3 | .1.3 Acute Phase Reactants (CRP and ESR) | 79 |
| 5.3 | .1.4 EULAR Response Criteria ······ | 79 |
| 5.3 | .1.5 DAS28 ····· | 80 |
| 5.3 | .1.6 SDAI Score | 80 |
| 5.3 | .1.7 ACR Response Criteria Assessment ····· | 81 |
| 5.3 | .1.8 Patient Reported Outcomes/Assessments······ | 81 |
| 5.3.2 | Pharmacodynamic Assessments · | 81 |
| 5.3 | .2.1 Lymphocyte Subsets · | 81 |
| 5.3 | .2.2 Biomarkers for Efficacy and Safety Assessments | 82 |
| 5.3.3 | Pharmacokinetic Assessments · | 82 |
| 5.4 | Safety Assessment · | 82 |
| 5.4.1 | Vital Signs····· | 82 |
| 5.4.2 | Body Weight ···· | 83 |
| 5.4.3 | Adverse Events · | 83 |
| 5.4 | .3.1 Adverse Events of Possible Hepatic Origin · | 83 |
| 5.4.4 | Laboratory Assessments · | 83 |
| 5.4 | .4.1 CPK Monitoring ····· | 85 |
| 5.4 | .4.2 Hepatic Function Abnormal · | 86 |
| 5.4.5 | Physical Examination · | 86 |
| 5.4.6 | 12-lead Electrocardiogram (ECG)····· | 86 |
| 5.4.7 | Radiography····· | 87 |
| 5.4.8 | Central ECG ···· | 87 |
| 5.5 | Adverse Events and Other Safety Aspects ····· | 87 |
| 5.5.1 | Definition of Adverse Events (AEs) ····· | 87 |
| 5.5.2 | Definition of Serious Adverse Events (SAEs) · | 88 |
| 5.5.3 | Criteria for Causal Relationship to the Study Drug ······ | 89 |
| 5.5.4 | Criteria for Defining the Severity of an Adverse Event ····· | 89 |

| | 5.5.5 | Reporting of Serious Adverse Events (SAEs) · | |
|---|---|---|---|
| | 5.5.6 | Follow-up of Adverse Events ····· | |
| | 5.5.7 | Procedure in Case of Pregnancy ····· | 91 |
| | 5.5.8 | Supply of New Information Affecting the Conduct of the Study · | 92 |
| | 5.5.9 | Deviations from the Protocol and Other Actions Taken to Avoid | |
| | | Life-Threatening Risks to Subjects····· | |
| | 5.6 | Test Drug Concentration · | |
| | 5.7 | Other Measurements, Assessments, or Methods · | 94 |
| | 5.7.1 | Pharmacodynamic Measurements · | 94 |
| | 5.7.2 | Purposes of Pharmacogenomics · | 94 |
| | 5.7.3 | Handling and Storage for Samples Used for Pharmacogenomics ······ | 95 |
| | 5.7.4 | Disposal of Pharmacogenomics Samples · | 95 |
| | 5.7.5 | Disclosure of Genetic Information · | 96 |
| | 5.8 | Total Amount of Blood····· | 96 |
| 6 | TEI | RMINATION OF THE CLINICAL STUDY | 98 |
| 7 | STA | ATISTICAL METHODOLOGY ······ | 99 |
| | 7.1 | Sample Size ····· | 99 |
| | 7.2 | Analysis Set····· | 100 |
| | 7.2.1 | Full Analysis Set (FAS) ····· | 100 |
| | 7.2.2 | Per Protocol Set (PPS) ····· | 100 |
| | 7.2.3 | Safety Analysis Set (SAF)····· | 101 |
| | 7.2.4 | Pharmacokinetic Analysis Set (PKAS) ······ | 101 |
| | 7.2.5 | Pharmacodynamics Analysis Set (PDAS)······ | 101 |
| | 7.3 | Demographics and Other Baseline Characteristics····· | 101 |
| | 7.4 | Analysis of Efficacy ····· | 101 |
| | 7.4.1 | Analysis of Primary Variable · | 101 |
| | 7.4 | 4.1.1 Primary Analysis····· | 101 |
| | 7.4 | 4.1.2 Secondary Analysis ····· | 102 |
| | 7.4 | 4.1.3 Subgroup Analysis····· | 102 |
| | 7.4.2 | Analysis of Secondary Variables · | 102 |
| | 7.5 | Analysis of Safety · | 102 |
| | 7.5.1 | Adverse Events ····· | 103 |
| | 7.5.2 | Laboratory Assessments · | 103 |
| | 7.5.3 | Vital Signs····· | 103 |

| | 7.5.4 | 12-lead ECG ····· | 103 |
|---|---|---|---|
| | 7.5.5 | QT assessment · | 103 |
| | 7.5.6 | Body Weight ····· | 103 |
| | 7.6 | Analysis of Pharmacokinetics · | 103 |
| | 7.7 | Other Analyses ····· | 104 |
| | 7.7.1 | Analysis of Pharmacodynamics · | 104 |
| | 7.7.2 | Analysis of Pharmacogenomics · | 104 |
| | 7.8 | Interim Analysis (and Early Discontinuation of the Clinical Study)······ | 104 |
| | 7.9 | Handling of Missing Data, Outliers, Visit Windows, and Other Information · · · · | 104 |
| | 7.9.1 | Handling of Schedule of Assessments of Efficacy Variables · | 104 |
| | 7.9.2 | Handling of Schedule of Assessments of Safety Variables ····· | 105 |
| | 7.9.3 | Handling of Schedule of Assessments of Pharmacodynamic Variables · · · · | 107 |
| | 7.9.4 | Handling of Schedule of Assessments of Pharmacokinetic Variables · · · · · · | 108 |
| 8 | OP | ERATIONAL AND ADMINISTRATIVE CONSIDERATIONS | 109 |
| | 8.1 | Procedure for Clinical Study Quality Control · | 109 |
| | 8.1.1 | Data Collection · | 109 |
| | 8.1.2 | Specification of Source Documents · | 109 |
| | 8.1.3 | Clinical Study Monitoring····· | |
| | 8.1.4 | Direct Access to Source Data/Documents · | |
| | 8.1.5 | Data Management · | |
| | 8.2 | Ethics and Protection of Subject Confidentiality · | ··· 111 |
| | 8.2.1 | Institutional Review Board (IRB)/ Independent Ethic Committee (IEC)···· | ··· 111 |
| | 8.2.2 | Ethical Conduct of the Study····· | |
| | 8.2.3 | Informed Consent of Subjects · | ··· 111 |
| | 8.2 | 2.3.1 Subject Information and Consent ····· | |
| | 8.2 | Subject Information and Consent for PGx Research | 112 |
| | 8.2 | 2.3.3 Supply of New and Important Information Influencing the Subject's Consent and Revision of the Written Information | 112 |
| | 8.2.4 | Subject Confidentiality · | 113 |
| | 8.3 | Administrative Matters | 113 |
| | 8.3.1 | Arrangement for Use of Information and Publication of the Clinical Study | 113 |
| | 8.3.2 | Documents and Records Related to the Clinical Study ······ | 114 |
| | 8.3.3 | Protocol Amendment and/or Revision · | |
| | 8.3.4 | Insurance of Subjects and Others ····· | 116 |
| | 8.3.5 | Signatory Investigator for Clinical Study Report····· | 117 |

| 9 | <b>Q</b> UA | ALITY A | SSURANCE 11 | 8 |
|---|---|---|---|---|
| 10 | STU | DY ORG | GANIZATION 11 | 9 |
| 10.1 | 1 | Independ | ent Data and Safety Monitoring Board (DSMB) · · · · · 11 | 9 |
| 10.2 | 2 | Other Eva | aluation Committee(s) · · · · · 11 | 9 |
| 10.3 | 3 | Other Stu | ndy Organization · · · · · 11 | 9 |
| 10.4 | 4 | Registrati | ion of Subjects · · · · · 12 | 20 |
| 11 | REF | FERENC | ES 12 | 22 |
| 12 | APP | PENDICE | 2S | 25 |
| APPE | NDIX | <1>: | LIST OF PROHIBITED CONCOMITANT MEDICATION ······· 12 | 25 |
| APPE | NDIX | <2>; | LABORATORY TESTS · · · · · 12 | 26 |
| APPE | NDIX | <3>; | EVENTS ALWAYS CONSIDERED SERIOUS 12 | 28 |
| APPE | NDIX | <4>; | LIVER SAFETY MONITORING AND ASSESSMENT 12 | 29 |
| APPE | NDIX | <5>: | 1987 ACR CRITERIA FOR THE CLASSIFICATION OF RA······ 13 | 32 |
| APPE | NDIX | <6>; | 2010 ACR-EULAR CLASSIFICATION CRITERIA FOR RA ······ 13 | 33 |
| APPE | | | CRITERIA FOR THE CLASSIFICATION OF GLOBAL<br>AL STATUS IN RA (1991 REVISED CRITERIA)13 | 34 |
| APPE | NDIX<br>RA | | CLASSIFICATION OF DISEASE STAGE/PROGRESSION OF 134 | |

# I. SIGNATURE

# AGREEMENT BETWEEN THE SPONSOR'S RESPONSIBLE PERSON AND THE INVESTIGATOR

This clinical study will be conducted in adherence to GCP, ICH Guidelines and applicable laws and regulatory requirements, as well as this study protocol. As the evidence of the agreement, the investigator (CHIKEN SEKININ ISHI) and responsible person of the Sponsor (CHIKEN IRAI SEKININSHA) inscribe in the bipartite agreement.

# II. CONTACT DETAILS OF KEY SPONSOR'S PERSONNEL

| Coı | ntact Information for the Sponsor |
|---|---|
| Coı | rporate Name: |
| Loc | cation: |
| Pho | one No.: |
| Fax | |
| Spo | onsor's personnel: |
| [Co | ontact numbers during non-business hours and for emergency]: |
| Co <sub>1</sub> | ntact Information for the Contract Research Organization (CRO) Japan |
| | Corporate name: |
| | Location: |
| | Phone No.: |
| | Fax: |
| | CRO's personnel: |
| | [Contact numbers during non-business hours and for emergency]: |
| > | Korea |
| | Corporate name: |
| | Location: |
| | Phone No.: |
| | Fax: |
| | CRO's personnel: |
| | [Contact numbers during non-husiness hours and for emergency]. |

| Taiwan |
|----------------------------------------------------------------|
| Corporate name: |
| Location: |
| Phone No.: |
| Fax: |
| CRO's personnel: |
| [Contact numbers during non-business hours and for emergency]: |

# III. LIST OF ABBREVIATIONS AND DEFINITION OF KEY TERMS

# **List of Abbreviations**

| Abbreviations | Description of abbreviations |
|---|---|
| ACR | American College of Rheumatology |
| AE | Adverse event |
| ALP | Alkaline phosphatase |
| ALT | Alanine aminotransferase (GPT) |
| AST | Aspartate aminotransferase (GOT) |
| ASP015K | Astellas Pharmaceuticals Compound 015K |
| AUC | |
| AUC | Area under the plasma concentration—time curve AUC from the time of dosing up to infinity with extrapolation of the |
| AUCinf | |
| ALIC | ALIC from the time of desired to the left management a concentration |
| AUC <sub>last</sub> | AUC from the time of dosing to the last measurable concentration |
| BUN | Blood urea nitrogen |
| anti-CCP antibody | anti-cyclic citrullinated peptide antibody |
| C <sub>max</sub> | Maximum concentration |
| Ctrough | Trough concentration |
| CK/CPK | Creatine kinase/creatine phosphokinase |
| CK-MB | Creatine kinase MB isozyme |
| CRF | Case report form |
| CRO | Contract research organization |
| CRP | C-reactive protein |
| CYP | Cytochrome P450 |
| DAS | Disease activity score |
| DIP | Distal interphalangeal joint |
| DILI | Drug-induced liver injury |
| DMARD | Disease-modifying antirheumatic drug |
| DNA | Deoxyribonucleic acid |
| DSMB | Data and safety monitoring board |
| ECG | Electrocardiogram |
| eCRF | Electronic case report form |
| EDC | Electronic data capture |
| EDTA | Ethylenediaminetetraacetic acid |
| ESR | Erythrocyte sedimentation rate |
| EU | European Union |
| EULAR | European League Against Rheumatism |
| FAS | Full analysis set |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| GFR | Glomerular filtration rate |
| GMP | Good Manufacturing Practice |
| γ-GTP | γ-Glutamyl transpeptidase (GGT) |
| HAQ-DI | Health Assessment Questionnaire - Disability Index |
| HBc antibody | Hepatitis B core antibody |
| HBs antigen/antibody | Hepatitis B surface antigen/antibody |
| HBV | Hepatitis B virus |
| HCV | Hepatitis C virus |
| 110 1 | 110puning C virus |

| Abbreviations | Description of abbreviations |
|---|---|
| HDL | High-density lipoprotein |
| hERG | Ether-a-go-go related gene |
| HIV | Human immunodeficiency virus |
| HSA | Human serum albumin |
| | International Conference on Harmonization of Technical Requirements for |
| ICH | Registration of Pharmaceuticals for Human Use |
| IEC | Independent Ethic Committee |
| IL | Interleukin |
| IND | Investigational new drug |
| INR | International normalized ratio |
| IP | International normanized ratio Interphalangeal joint |
| IR | 1 - 1 |
| IRB | Inadequate response Institutional review board |
| ISN | International study number |
| JAK | Janus kinase |
| LA-CRF | Liver abnormality - CRF |
| LC-MS | Liquid chromatography- mass spectrometry |
| LDL | Low-density lipoprotein |
| LOCF | Last observation carried forward |
| MCP | Metacarpophalangeal joint |
| MDRD | Modification of diet in renal disease |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MMF | Mycophenolate mofetil |
| MMP-3 | Matrix metalloproteinase 3 |
| MPA | Mycophenolic acid |
| MPAG | Mycophenolic acid glucuronide |
| MTP | Metatarsophalangeal joint |
| MTX | Methotrexate |
| NCI-CTCAE | National Cancer Institute Common Terminology Criteria for Adverse |
| NCI-CICAE | Events |
| NDA | New drug application |
| NK | Natural killer |
| NOAEL | No observed adverse effect level |
| NSAIDs | Non-steroidal anti-inflammatory drugs |
| NYHA | New York Heart Association |
| PASI | Psoriasis Area and Severity Index |
| PD | Pharmacodynamic |
| PDAS | Pharmacodynamic analysis set |
| PGA | Physician's Global Assessment of Arthritis |
| PGx | Pharmacogenomics |
| PIP | Proximal interphalangeal joint |
| PK | Pharmacokinetic |
| PKAS | Pharmacokinetic analysis set |
| PPS | Per protocol set |
| QOL | Quality of life |
| RA | Rheumatoid arthritis |
| RF | Rheumatoid factor |
| SAE | Serious adverse event |
| SAF | Safety analysis set |
| SAI | Sately analysis set |

| Abbreviations | Description of abbreviations |
|------------------|---------------------------------------------------------|
| SDAI | Simplified Disease Activity Index |
| SF-36v2® | Short Form Health Survey – 36 questions, version 2 |
| SFL | Screening failure log |
| SGA | Subject's Global Assessment of Arthritis |
| SJC | Swollen joint count |
| SOP | Standard operating procedure |
| STAT5 | Signal transducers and activators of transcription 5 |
| SUSAR | Suspected unexpected serious adverse reactions |
| TBL | Total bilirubin |
| TEAE | Treatment emergent adverse event |
| TJC | Tender joint count |
| TNF | Tumor necrosis factor |
| t <sub>1/2</sub> | Apparent terminal elimination half-life |
| t <sub>max</sub> | Time to attain C <sub>max</sub> |
| TYK | Tyrosine kinase |
| ULN | Upper limit of normal |
| VAS | Visual analog scale |
| VEGF | Vascular endothelial growth factor |
| WBC | White blood cell |
| WPAI | Work Productivity and Activity Impairment Questionnaire |

# **Definition of Key Study Terms**

| Terms | Definition of terms |
|---|---|
| Adverse event | An adverse event is defined as any untoward medical occurrence in a |
| | subject administered a study drug or reference drug that does not |
| | necessarily have a causal relationship with this treatment. |
| Baseline | 1) Values/findings observed prior to the initiation of study treatment, |
| | which are regarded as the starting point for comparison. |
| | 2) The time point at which those reference values/findings were observed. |
| Study discontinuation | The act of concluding participation, prior to completion of all |
| | protocol-required elements, in a study by an enrolled subject. Four |
| | categories of discontinuation are distinguished: a) dropout: Active |
| | discontinuation by a subject (also a noun referring to such a discontinued |
| | subject); b) discontinuation initiated by the investigator or other |
| | responsible personnel (e.g., for cause); c) loss to follow-up: |
| | discontinuation of participation without notice or action by the subject; d) |
| | sponsor-initiated discontinuation. |
| | Note that subject discontinuation does not necessarily imply exclusion of |
| | subject data from analysis. |
| Enroll | To register or enter into a clinical study; transitively and intransitively. |
| Linon | Informed consent precedes enrollment, which precedes or is |
| | contemporaneous with randomization. |
| Investigational period | The period of time where major interests of protocol objectives are |
| mvestigational period | observed. In general, the subject will receive a test drug, comparative |
| | drug, or reference drug (possibly without randomization) during this |
| | period, which extends until the last post-treatment assessment is |
| | completed. |
| Follow-up period | The follow-up period will be 4 weeks (on a per-protocol basis) starting |
| ronow-up penou | after the early-termination visit for withdrawn subjects and after the Week |
| | 52 visit for subjects who completed the study but are not willing to enroll |
| | into the extension study or those in the reference group who completed the |
| | study. For subjects who completed the study and wish to enroll into the |
| | extension study, the follow-up period will last for a maximum of 4 weeks |
| | starting after the Week 52 visit and ending at the initiation of the extension |
| | study treatment. |
| Randomization | |
| Kangonnzanon | Action to allocate a subject to the treatment group or treatment cohort. |
| | Depending on the type of rules for handling for study drugs, 'Randomization' is usually executed just before entering the |
| | 'investigational period.' |
| Caraanina | |
| Screening | 1) Process of searching for candidates for the study 2) Process of shaeking the eligibility of subjects, usually done during the |
| | 2) Process of checking the eligibility of subjects, usually done during the "pro-investigational period" |
| Caraaning failum | "pre-investigational period" Saragnad subject, but did not fulfill protocol inclusion and/or evaluation |
| Screening failure | Screened subject, but did not fulfill protocol inclusion and/or exclusion |
| | criteria and failed to receive randomized or open label study treatment, or |
| | decided not to participate anymore (withdrew consent) prior to completing |
| | pre-investigational period. |

| Terms | <b>Definition of terms</b> |
|---|---|
| Serious adverse event | Any adverse event that is judged "serious" by the |
| | investigator/sub-investigator or the sponsor and results in any of the |
| | following outcomes: death, a life-threatening condition, persistent or |
| | significant disability/incapacity or substantial disruption of the ability to |
| | conduct normal life functions, congenital anomaly/birth defect, |
| | hospitalization or prolongation of hospitalization, and other medically |
| | significant occurrences. |
| Study period | The period of time from obtaining informed consent from the subject to |
| | the end of the final evaluation/observation specified in the protocol. |
| Subject | An individual who participates in a clinical study as a recipient of either |
| | the test drug(s) or reference drug(s), or as a control. |
| Subject ID | A unique identifier code assigned to each subject signing the informed |
| | consent. |
| Variable | A characteristic under study that varies: any attribute, phenomenon, or |
| | event that can have different qualitative or quantitative values. |

# IV. SYNOPSIS

| Till COLL | N HI C. 1 CACROLOU |
|---|---|
| Title of Study: | Phase III Study of ASP015K |
| | A randomized, double-blind, placebo-controlled confirmatory study of the |
| | safety and efficacy of ASP015K in patients with rheumatoid arthritis (RA) who |
| | had an inadequate response to DMARDs— |
| | (Protocol No.: 015K-CL-RAJ3) |
| Planned Study Period: | From July 2014 to December 2017 |
| Study Objectives: | The objectives of the study are as follows: |
| | To verify the superiority of ASP015K alone or in combination with |
| | disease-modifying antirheumatic drugs (DMARDs) over placebo in terms of |
| | efficacy, at doses of 100 mg/day and 150 mg/day, in patients with rheumatoid |
| | arthritis (RA) who had an inadequate response to DMARDs, as measured by |
| | the ACR20 response rate at Week 12, which is the primary variable; |
| | To evaluate the pharmacokinetics, pharmacodynamics, and safety of ASP015K; |
| | To evaluate the efficacy and safety of long-term treatment with ASP015K (52 weeks); and |
| | To use open-label etanercept, an existing anti-TNF agent, as the reference |
| | drug. |
| <b>Planned Total Number of</b> | Approximately 160 centers |
| Study Centers and | Japan, Korea, and Taiwan |
| Locations: | |
| Design and Methodology: | This is a multi-center, randomized, placebo-controlled, double-blind, |
| | parallel-group, confirmatory study to evaluate the efficacy and safety of |
| | ASP015K alone or in combination with DMARDs, at doses of 100 mg and |
| | 150 mg, in patients with RA who had an inadequate response to DMARDs. |
| | Etanercept will also be administered as the reference drug. In the study, |
| | ASP015K (test drug) and placebo (comparative drug) will be given as study |
| | drugs, and etanercept will be given as a separate reference drug. After |
| | screening, subjects will be randomized at baseline in a 1:1:1:2 ratio to the |
| | ASP015K 100 mg group, ASP015K 150 mg group, placebo group, or reference |
| | group in each study region. The study drug will be orally administered once |
| | daily (QD) after breakfast for 52 weeks. Etanercept will be administered |
| | subcutaneously once weekly for 52 weeks (the last dose will be given at Week |
| | 51). At Week 12, subjects in the placebo group will be switched to either |
| | ASP015K 100 mg or ASP015K 150 mg, and the dose will be maintained until |
| | the end of treatment. The dose of ASP015K (100 or 150 mg) to be started at |
| | Week 12 for the placebo group will be determined randomly at baseline in |
| | advance and switched in a blinded manner. |
| | Dynamic allocation procedures in each study region (Japan, Korea and |
| | Taiwan) will be used at randomization at baseline, with the study center, prior |
| | biologic-DMARD-IR, and concomitant DMARD use at the initiation of |
| | treatment with the study drug or reference drug as covariates. |
| | An anti-TNF agent, etanercept, will be administered as the reference drug in an |
| | open-label manner. |
| | Subjects in the ASP015K 100 mg, ASP015K 150 mg, or placebo groups who |
| | have completed the study will be eligible for participation in an open-label |
| | extension study (015K-CL-RAJ2). Subjects will make a follow-up visit after |
| | the Week 52 visit if they do not enroll into the extension study on the day of |
| | the Week 52 visit. |
| Number of Subjects to Be | One-hundred subjects per group will receive the study drug and 200 subjects |
| Enrolled/Randomized: | the reference drug (a total of 500 subjects). |
| | 1 |

# Inclusion/Exclusion Criteria:

<Inclusion Criteria>

Subject is eligible for the study if all of the following apply:

- 1. Subject has received a full explanation of the study drug and this study in advance, and written informed consent to participate in the study has been obtained from the subject himself/herself.
- 2. Subject is a man or woman aged  $\geq 20$  years at the time of informed consent.
- 3. Subject has RA diagnosed according to the 1987 American College of Rheumatology (ACR) criteria or the 2010 American College of Rheumatology/European League against Rheumatism (ACR/EULAR) criteria.
- 4. Subject who did not receive the following drugs, or received the drugs with stable dosage for at least 28 days prior to the baseline (start of treatment) for RA treatment:

Non-steroidal anti-inflammatory drugs (NSAIDs; excluding topical formulations), oral morphine or equivalent opioid analgesics (≤ 30 mg/day), acetaminophen, or oral corticosteroids (≤ 10 mg/day in prednisolone equivalent).

- 5. At screening subject has active RA as evidenced by both of the following:
  - $\geq$  6 tender/painful joints (using 68-joint assessment)
  - $\geq$  6 swollen joints (using 66-joint assessment)
- 6. CRP > 0.50 mg/dL at screening
- 7. Subject meets the ACR 1991 Revised Criteria for the Classification of Global Functional Status in RA Class I, II, or III at screening.
- 8. Inadequate responder to (including subjects who were intolerant of) at least one DMARD administered for at least 90 days prior to screening
- 9. When the following DMARDs are concomitantly administered to subject, the drugs must be administered for at least 90 days prior to screening, and must be stable from at least 28 days prior to screening until the end of the administration period of study drug or reference drug.
  - Methotrexate (MTX)
  - Hydroxychloroquine
  - Salazosulfapyridine
  - Gold
  - D-penicillamine
  - Lobenzarit
  - Actarit
  - Bucillamine
  - Iguratimod

10. Subject must be willing and able to comply with the study requirements.

# Inclusion/Exclusion Criteria:

#### <Exclusion Criteria>

Subject will be excluded from participation if any of the following applies:

- 1. Subject has received a biologic DMARD within the specified period:
  - Anakinra: within 28 days prior to baseline
  - Adalimumab, infliximab: within 56 days prior to baseline
  - Golimumab, certolizumab pegol: within 70 days prior to baseline
  - Abatacept, tocilizumab: within 84 days prior to baseline
  - Denosumab: within 150 days prior to baseline
  - Rituximab: within 180 days prior to baseline
- 2. Subject has received etanercept.
- 3. Inadequate responder to at least 3 biologic DMARDs as determined by investigator/sub-investigator.
- 4. Subject has received a non-biologic DMARD listed below or other drugs used in the treatment of RA within 28 days prior to baseline. Leflunomide is prohibited within 180 days prior to baseline. Alternatively, leflunomide is prohibited within 28 days prior to baseline if washout with cholestyramine for at least 17 days is completed at least 28 days prior to baseline. However, topical drugs other than those for the treatment of RA may be used concomitantly.
  - Leflunomide
  - Tacrolimus
  - Cyclosporine
  - Cyclophosphamide
  - Azathioprine
  - Minocycline
  - Mizoribine
- 5. Subject has received to facitinib or other JAK inhibitor (including other investigational drugs).
- 6. Subject has received intra-articular, intravenous, intramuscular, or endorectal (excluding suppositories for anal diseases) corticosteroid within 28 days prior to baseline.
- 7. Subject has participated in any study of ASP015K and has received ASP015K or placebo.
- 8. Subject has received other investigational drugs within 90 days or within 5 half-lives, whichever is longer, prior to baseline.
- 9. Subject has received plasma exchange therapy within 60 days prior to baseline.
- 10. Subject has undergone joint drainage, has received local anesthesia and nerve block, or has received articular cartilage protectant at the assessed joint within 28 days prior to baseline.
- 11. Subject has undergone surgery and has residual effects in the assessed joints at the discretion of investigator/sub-investigator, or is scheduled to undergo surgery that may affect the study evaluation of the assessed joints at the discretion of investigator/sub-investigator.
- 12. A diagnosis of inflammatory arthritis (psoriatic arthritis, ankylosing spondylitis, SLE, sarcoidosis, etc.) other than RA.
- 13. Any of the following laboratory values during the screening test period:
  - Hemoglobin < 9.0 g/dL
  - Absolute neutrophil count  $< 1000/\mu L$
  - Absolute lymphocyte count < 800/µL
  - Platelet count < 75000/μL

# Inclusion/Exclusion Criteria:

- ALT  $\geq 2 \times ULN$
- AST  $> 2 \times ULN$
- Total bilirubin (TBL)  $\geq 1.5 \times ULN$
- Estimated GFR ≤ 40 mL/min as measured by the MDRD method
- $\beta$ -D-glucan > ULN [in case of Japan:  $\geq 11$  pg/mL]
- Positive HBs antigen, HBc antibody, HBs antibody, or HBV-DNA quantitation (However, subject with negative HBs antigen and HBV-DNA quantitation, and positive HBc antibody and/or HBs antibody is eligible if HBV-DNA is monitored by HBV-DNA quantitation at every scheduled visit after initiation of study drug or reference drug administration.)
- Positive HCV antibody
- 14. Subject has a history of or concurrent active tuberculosis (TB). Eligibility criteria for TB are tabulated below:

| | 1 | | 1 | |
|---|---|---|---|---|
| History of | Chest x-ray (for TB) | TB | Exposure to | Eligibility |
| active TB | | infection <sup>b)</sup> | patients | |
| | | | with | |
| | | | infective TB | |
| | | | (interview) | |
| Present | - | - | - | Not eligible |
| Absent | Abnormal (active) | =. | - | Not eligible |
| | | | Eligible | Eligible if |
| | Abnormal (old) <sup>a)</sup> | _ | | prophylaxis is |
| | 7 tonormar (old) | | | given <sup>c)</sup> |
| | Normal | Positive | Eligible | Eligible if |
| | | | | prophylaxis is |
| | | | | given <sup>c)</sup> |
| | | Negative | Exposed | Eligible if |
| | | | _ | prophylaxis is |
| | | | | given <sup>c)</sup> |
| | | | Not exposed | Eligible |

- a) Old TB is evidenced if chest x-ray reveals pleural thickening, band-like shadow, and calcification  $\geq$  5 mm. Chest x-ray within 90 days prior to baseline may substitute the screening test.
- b) T-spot or Quantiferon Gold test is of first priority. When the result is equivocal or invalid, retest including other test methods may be allowed. If a retest is not performed, criteria for positive results will be followed. When T-spot or Quantiferon Gold test is not feasible, tuberculin test will be performed. Tuberculin is defined as positive with a red spot covering an area of 20 mm or more or induration. Tests conducted within 90 days prior to baseline may be used for diagnosis.
- c) Subject must receive or have received prophylaxis with isoniazid or rifampicin. Prophylaxis will be administered for 6 to 9 months, starting from at least 21 days prior to baseline.
- 15. Subject meets any of the following in terms of infections except for TB:
  - History of or concurrent severe herpes zoster (associated with Hunt syndrome or having ulcerative lesions) or disseminated herpes zoster
  - History of multiple recurrences (at least twice) of localized herpes zoster
  - Serious infection requiring hospitalization within 90 days prior to baseline
  - Subject has received intravenous antibiotics within 90 days prior to baseline. (However, prophylactic antibiotics are allowed.)
  - Subject with high risk of infection (e.g., subject with urinary catheter) at the discretion of investigator/sub-investigator

# Inclusion/Exclusion Criteria:

- 16. Subject has a history of or concurrent interstitial pneumonia and investigator/sub-investigator judges that it is inappropriate for the subject to participate in this study.
- 17. Subject has a history of or concurrent malignant tumor (except for successfully treated basal cell carcinoma).
- 18. Subject has received live or live attenuated virus vaccination within 56 days prior to baseline. (Inactivated vaccines including influenza and pneumococcal vaccines are allowed.)
- 19. Subject has a history of or concurrent demyelinating disorders.
- 20. Subject has any ongoing severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, metabolic, endocrine, pulmonary, cardiac, neurological, infectious, or autoimmune disease except for RA (excluding Sjogren's syndrome and chronic thyroiditis), or any ongoing illness which would make the subject unsuitable for the study as determined by the investigator/sub-investigator.
- 21. Subject has a history of clinically significant allergy. (Clinically significant allergy includes allergies such as systemic urticaria induced by specific antigens and drugs, anaphylaxis, and allergy associated with shock necessitating hospitalized treatment.)
- 22. Subject has received medications that are CYP3A substrates with narrow therapeutic range within 14 days prior to baseline. These medications include: dihydroergotamine, ergotamine, fentanyl, pimozide, quinidine, temsirolimus, and disopyramide.
- 23. Subject has concurrent cardiac failure, defined as NYHA classification Class III or higher, or a history of it.
- 24. Subject has concurrent prolonged QT syndrome or a history of it. Subject has prolonged QT interval (defined as QTc ≥ 500 msec. Subject has QTc ≥ 500 msec at retest will be excluded) at screening.
- 25. Subject has a history of positive HIV infection.
- 26. Subject is a woman who is pregnant or might be pregnant, is nursing, wishes to conceive for a period running from the time informed consent is given within 60 days after end of treatment (including reference drug), or for whom the possibility of pregnancy cannot be ruled out as a result of the serum pregnancy test given at the time of screening.
- 27. Subject is a man who cannot practice at least 2 types of contraception from the time of informed consent to 90 days after end of treatment (including reference drug), or subject is a woman with childbearing potential who cannot practice at least 2 types of contraception from the time of informed consent to 60 days after end of treatment (including reference drug).
- 28. Male subject who do not agree not to donate sperm starting at informed consent and through the treatment period and for at least 90 days after final study drug (or reference drug) administration. Female subject who do not agree not to donate ova starting at informed consent through the treatment period and for 60 days after final study drug (or reference drug) administration.
- 29. The subject has been judged unsuitable to participate in the study for other reasons by the investigator/sub-investigator.
- 30. The subject has a history or complication of lymphatic diseases such as lymphoproliferative disorder, lymphoma, and leukemia.
- 31. Subject has congenital short QT syndrome or a history of it. Subject has shortened QT interval (defined as QTc < 330 msec. Subject has QTc < 330 msec at retest will be excluded) at screening.

#### **Discontinuation Criteria:**

The investigator/sub-investigator should discontinue the study if any of the following occurs:

- 1. The subject withdraws consent.
- 2. The investigator/sub-investigator judges that the study drug or reference drug is not sufficiently effective and the treatment method needs to be changed.
- 3. Symptomatic CPK elevation (> 1.5 × ULN accompanied with severe and unusual episodes of myalgia, muscular weakness, or muscle twitching).
- 4. Any case of myopathy involving severe and unusual episodes of myalgia, muscular weakness, or muscle twitching that persists for no less than, or aggravates rapidly within, 2 weeks, regardless of the CPK level.
- 5. A previously HBV-infected patient with positive HBc antibody, positive HBs antibody, or both has been shown positive for HBV-DNA during the study.
  - Attention should be paid that abrupt discontinuation of immunotherapy may cause fulminant or severe liver failure. Therefore, if the subject manifests HBV reactivation, the investigator/sub-investigator will administer nucleoside analogs without delay [unique to Japan: according to the "Proposal for Management of Rheumatic Disease Patients with Hepatitis B Virus Infection Receiving Immunosuppressive Therapy" (Japan College of Rheumatology)]. The investigator/sub-investigator will carefully decide whether to continue or discontinue the study drug, reference drug, and concomitant DMARDs in consultation with the hepatology specialist.
- 6. Malignant tumor
- 7. The subject develops a serious infection or other adverse events (AEs), and continued administration of the study drug is not deemed appropriate in the subject's best interest by the investigator/sub-investigator.
- 8. The subject has been treated with a prohibited concomitant drug or therapy (including another investigational product) that may impact efficacy evaluation. The subject has been, or needs to be, treated with a rescue medication for a period extending beyond its allowable time. Otherwise, the subject has been, or needs to be, treated with a live or live attenuated vaccine.
- 9. The subject has been judged by the investigator/sub-investigator to be non-compliant to the medication requirements for treatment with the study drug, concomitant DMARDs, or reference drug injection.
- 10. The subject is deemed incapable of continuing the follow-up based on the opinion of the investigator/sub-investigator (subject can no longer come to the study center; subject can no longer be contacted, etc.).
- 11. It comes to light after the administration of the first dose of study drug or reference drug that inclusion criteria were not met at the time of case enrollment or that criteria for exclusion were met. It comes to light that there was some other major deviation from the protocol.
- 12. The subject needs the study drug or reference drug to be interrupted beyond its allowable time limit.
- 13. Investigator/sub-investigator decides it is in the subject's best interest.
- 14. The sponsor has requested that the study be discontinued because of a safety concern in a particular subject, or the sponsor has decided to discontinue the study altogether.
- 15. The Subject shows QTc interval < 300 msec at central ECG, or the subject shows QTc interval < 300 msec at the study site's ECG and also shows QTc interval < 300 msec at retest of study site's ECG.

# Suspension, Interruption, and Resumption of the Study Drug or Reference Drug:

During treatment with the study drug or reference drug, if the subject meets any of the criteria provided in "Criteria for Suspension or Interruption of the Study Drug or Reference Drug," the investigator/sub-investigator will immediately suspend or interrupt the study drug or reference drug. The investigator/sub-investigator can resume treatment with the study drug or reference drug only if re-examinations and other assessments performed after the suspension or interruption confirm that none of the conditions listed below are applicable to the subject and the investigator/sub-investigator considers it desirable for the interest of the subject on the basis of risk-benefit analysis.

The maximum allowable time for "suspension" is 7 days for the study drug and a week (1 dose per week) for the reference drug. If the treatment is halted beyond the suspension period, i.e., longer than 7 days for the study drug or skipping more than 1 dose for the reference drug, the period of no treatment is categorized as an "interruption."

Upper limits have been set to the number of interruptions 1 subject can have and to the duration of 1 interruption. One interruption period may last for 28 days for the study drug and 4 weeks (i.e., 4 consecutive doses) for the reference drug. One subject is allowed to have a maximum of 2 interruptions, which must be separated by 16 or more weeks.

The investigator will consult the sponsor regarding the handling of a subject who repeatedly requires treatment suspension.

The subject must be withdrawn from the study, if he or she requires either a third interruption or a second interruption within less than 16 weeks from the first one.

Criteria for Suspension or Interruption of the Study Drug or Reference Drug The investigator/sub-investigator will suspend or interrupt the study drug or reference drug if any of the following becomes applicable during treatment with the study drug or reference drug:

- 1. Clinical laboratory tests yielded any of the following results:
  - Hemoglobin < 8.0 g/dL
  - Absolute neutrophil count  $< 500/\mu L$
  - Absolute lymphocyte count  $< 500/\mu L$
  - Platelet count  $< 50000/\mu L$
  - Creatinine (serum) levels measured at 2 consecutive hospital visits: above 150% of the baseline level
  - $CPK > 10 \times ULN$
- 2.  $\beta$ -D-glucan > ULN [in case of Japan:  $\geq 11 \text{ pg/mL}$ ]
- 3. The subject requires a medication whose concomitant administration is prohibited in the protocol because of possible drug-drug interaction.
- 4. The subject is suspected to be pregnant.
- 5. The investigator/sub-investigator judged it appropriate in the interest of the subject to suspend or interrupt the study drug or reference drug.
- 6. The sponsor made a request to suspend or interrupt the study drug or reference drug out of safety concerns for the subject.

## Participation in an Open-Label Extension Study:

Subjects in the ASP015K 100 mg group, ASP015K 150 mg group, or placebo group who have completed the study will be eligible for participation in the open-label extension study (Protocol No.: 015K-CL-RAJ2).

| Test Drugs: | Test drugs: ASP015K 1 | 00 mg and 150 mg tablets |
|---|---|---|
| Mode of Administration: | Dose: 100 mg/day, 150 | |
| Dose: | | : To be orally administered QD after breakfast. The first |
| Duration of Treatment: | dose should be given at each study center on the day | |
| Duration of Treatment. | of the baseline visit after all the necessary assessm | |
| | | and tests have been completed. |
| | Duration of treatment: | - |
| Commonstino Dungo | | - 11 - 1 |
| Comparative Drugs: | ASP015K placebo table | |
| Mode of Administration: | Mode of administration | : To be orally administered QD after breakfast. The first |
| Dose: | | dose should be given at each study center on the day |
| <b>Duration of Treatment:</b> | of the baseline visit after all the necessary assessme | |
| | | and tests have been completed. |
| | Duration of treatment: | 52 weeks (placebo will be administered for a |
| | | maximum of 12 weeks. Subjects in the placebo group |
| | | will be switched to either ASP015K 100 mg or |
| | | ASP015K 150 mg at Week 12.) |
| Reference Drugs: | Etanercept: 50 mg for s | ubcutaneous injection, syringe: 1.0 mL |
| Mode of Administration: | Mode of administration | : To be subcutaneously administered once weekly. The |
| Dose: | | first dose should be given at each study center on the |
| <b>Duration of Treatment:</b> | | day of the baseline visit after all the necessary |
| | | assessments and tests have been completed. |
| | | Subsequent doses may be given at the study center or |
| | | self-administered. Subjects who receive etanercept at |
| | | the study center will be required to visit the site in |
| | | addition to the scheduled visits. |
| | Duration of treatment: | 52 weeks (the last dose will be given at Week 51) |
| | Duration of fleatifient. | 32 weeks (the last dose will be given at week 31) |

# Concomitant Medication:

- 1) Prohibited concomitant medications and therapies
- Biologic DMARDs

Administration of the biologic DMARDs below will be prohibited for a specified period of time (stated below) and during treatment with the study drug or reference drug. Etanercept given as the reference drug will be excluded.

- > Etanercept: after informed consent is obtained
- Anakinra: within 28 days prior to baseline
- Adalimumab, infliximab: within 56 days prior to baseline
- ➤ Golimumab, certolizumab pegol: within 70 days prior to baseline
- Abatacept, tocilizumab: within 84 days prior to baseline
- > Denosumab: within 150 days prior to baseline
- Rituximab: within 180 days prior to baseline

#### • Non-biologic DMARDs

Administration of non-biologic DMARDs other than those listed below will be prohibited within 28 days prior to baseline and during treatment with the study drug or reference drug.

Subjects who continue receiving the drugs described below during treatment with the study drug or reference drug should follow regulations for restricted concomitant medications.

The use of leflunomide is prohibited within 180 days prior to baseline. However, if washout with cholestyramine for at least 17 days is completed before 28 days prior to baseline, the use of leflunomide will be prohibited within 28 days prior to baseline and during treatment with the study drug or reference drug.

When subjects discontinue receiving the drugs listed below before the initiation of treatment with the study drug or reference drug, their use will be prohibited within 28 days prior to baseline and during treatment with the study drug or reference drug. However, topical drugs other than those for the treatment of RA may be used concomitantly.

- ➤ Methotrexate (MTX)
- > Hydroxychloroquine
- > Salazosulfapyridine
- ➢ Gold
- ➤ *D*-penicillamine
- ➤ Lobenzarit
- Actarit
- ➤ Bucillamine
- > Iguratimod

# Concomitant Medication:

- Other drugs to be used in the treatment of RA
   Cyclosporine, cyclophosphamide, azathioprine, minocycline, and other
   drugs indicated for the treatment of RA will be prohibited within 28 days
   prior to baseline and during treatment with the study drug or reference
   drug.
- Corticosteroids

Oral corticosteroids at doses exceeding 10 mg per day in the prednisolone equivalent will be prohibited within 28 days prior to baseline and during treatment with the study drug or reference drug.

The intra-articular, intravenous, intramuscular, and endorectal corticosteroid administration will also be prohibited within 28 days prior to baseline and during treatment with the study drug or reference drug. However, suppositories for anal diseases may be used concomitantly.

Oral morphine

Oral morphine at doses exceeding 30 mg per day (or equivalent doses of other opioid analgesics) will be prohibited within 28 days prior to baseline and during treatment with the study drug or reference drug.

• Other study drugs

Other study drugs will be prohibited within 90 days or 5 half-lives, whichever is longer, prior to baseline. In addition, the use of other study drugs will be prohibited during the study period.

CYP3A substrates

The following CYP3A substrate drugs with a narrow therapeutic range will be prohibited within 14 days prior to baseline, during treatment with the study drug or reference drug, and during the follow-up period: dihydroergotamine, ergotamine, fentanyl, pimozide, quinidine, temsirolimus, disopyramide, etc.

Vaccines

Live or live attenuated vaccinations will be prohibited within 56 days prior to baseline, during treatment with the study drug or reference drug, and during the follow-up period. Inactivated vaccines may be administered (influenza, pneumococcal vaccines, etc.).

- Plasma exchange therapy
   Plasma exchange therapy will be prohibited within 60 days prior to baseline and during treatment with the study drug or reference drug.
- Surgical treatment methods
   Surgery involving the target joint will be prohibited from the time of informed consent to the end of treatment with the study drug or reference drug.
- Effusion drainage, local anesthesia, and nerve block of the target joint Effusion drainage, local anesthesia, and nerve block of the target joint will be prohibited within 28 days prior to baseline and during treatment with the study drug or reference drug.
- Articular cartilage protective agents
   The use of articular cartilage protective agents in the target joint will be prohibited within 28 days prior to baseline and during treatment with the study drug or reference drug.
- 2) Restricted concomitant medications

<Concomitant DMARDs>

• If any (some) of the following DMARDs are administered concomitantly with the study drug or reference drug, they should be given for at least 90 days prior to screening, and the same dosage and administration schedule must be maintained from at least 28 days prior to screening to the end of treatment with the study drug or reference drug.

# Concomitant Medication:

- Changes to the dosage, administration schedule, or route of administration will not be allowed within 28 days prior to baseline and during treatment with the study drug or reference drug.
- If a DMARD is temporarily interrupted or its dose is reduced within 28 days prior to the baseline visit in a subject eligible at screening for the study based on inclusion and exclusion criteria, the screening period will be extended to allow for the same dosage and administration schedule to be observed for 28 days prior to the baseline visit.
- In the case of AEs, administration may be temporarily interrupted, or the dose may be temporarily reduced. When resuming administration, the baseline dose is the upper limit. The period of interruption is up to 28 days and interruption is allowed only once.
- If MTX is administered with study drug or reference drug concurrently, the concomitant use of folic acid should be considered whenever possible. The dose of folic acid during the study period will, in principle, be within 10 mg per week, but it may be adjusted. If MTX is administered and ALT/AST becomes ≥ 3 × ULN, MTX must be interrupted, or the dose must be reduced, and daily administration of folic acid should be considered.
  - ➤ Methotrexate (MTX)
  - > Hydroxychloroquine
  - > Salazosulfapyridine
  - ➤ Gold
  - ➤ *D*-penicillamine
  - ➤ Lobenzarit
  - > Actarit
  - ➤ Bucillamine
  - > Iguratimod

#### <Other restricted concomitant medications>

Regarding the drugs listed below, changes to the dosage, administration schedule, or route of administration will not be allowed within 28 days prior to baseline and during treatment with the study drug or reference drug, unless the specific conditions for the change are met.

- The drugs listed below will be prohibited within 28 days prior to baseline
  and during treatment with the study drug or reference drug if they are to be
  discontinued before the initiation of treatment with the study drug or
  reference drug [except in cases where NSAIDs and non-NSAID analgesics
  (e.g., acetaminophen, opioid analgesics, all-in-one flu and cold
  medications) are used as rescue medication].
- In the case of AEs, administration of drugs below may be temporarily interrupted, or the dose may be temporarily reduced. The period of interruption is up to 28 days. When resuming administration, the baseline dose is the upper limit.
- During treatment with the study drug or reference drug from Week 12, the
  drugs below may be discontinued, new drugs may be used, and the dosage,
  administration schedule, or route of administration of the concomitant
  drugs may be changed. However, with the exception of oral corticosteroids,
  after changing the conditions, administration must be continued under the
  same conditions for 12 weeks or longer.
  - ➤ NSAIDs (excluding topical drugs)
  - ➤ Oral morphine (not more than 30 mg per day, or equivalent doses of other opioid analgesics)
  - > Acetaminophen

| Composition 4 | Outloomiogramaid- (I |
|---|---|
| Concomitant<br>Medication: | ➤ Oral corticosteroids (however, at 10 mg per day or less in the prednisolone equivalent and from the visit at Week 12, the dose may be reduced or increased within the range not exceeding the baseline dose.) |
| | 3) Rescue medications |
| | The drugs listed below may be administered only if they are necessary for |
| | treating an untoward medical occurrence, AEs, comorbid conditions, or |
| | acute aggravation of the primary disease within 28 days prior to baseline |
| | and during treatment with the study drug or reference drug. However, these |
| | medications may not be taken within 24 hours before joint assessment at |
| | each visit. ➤ NSAIDs: For 3 days or less |
| | Analgesics other than NSAIDs (acetaminophen, opioid analgesics, |
| | all-in-one flu and cold medications, etc.): For 7 consecutive days or less |
| Major Outcome | <primary variables=""></primary> |
| Variables | ACR20 response rate at Week 12 |
| Efficacy | <secondary variables=""></secondary> |
| | • ACR20 response rate |
| | <ul> <li>ACR50 response rate</li> <li>ACR70 response rate</li> </ul> |
| | <ul> <li>Change from baseline in DAS28-CRP and DAS28-ESR scores</li> </ul> |
| | • Change from baseline in Tender Joint Count (TJC) (68 joints) |
| | • Change from baseline in Swollen Joint Count (SJC) (66 joints) |
| | <ul> <li>Percentage of subjects achieving DAS28-CRP and DAS28-ESR scores for</li> </ul> |
| | remission |
| | <ul> <li>Percentage of subjects achieving low disease activity by DAS28-CRP and<br/>DAS28-ESR</li> </ul> |
| | Change from baseline in CRP and ESR |
| | <ul> <li>Percentage of subjects with good EULAR response</li> <li>Percentage of subjects with good or moderate EULAR response</li> </ul> |
| | <ul> <li>Percentage of subjects with good or moderate EULAR response</li> <li>Percentage of subjects achieving ACR/EULAR remission</li> </ul> |
| | If all of the following 4 parameters are fulfilled, it is defined as remission: |
| | > TJC ≤ 1 |
| | SJC ≤ 1 |
| | $ ightharpoonup CRP \le 1 \text{ mg/dL}$ |
| | Subject's Global Assessment of Arthritis (SGA) ≤ 1 cm (on a VAS of 0–100 mm) |
| | <ul> <li>Percentage of subjects achieving SDAI remission (SDAI score ≤ 3.3)</li> <li>Change from baseline in SDAI score</li> </ul> |
| | • Change from baseline in Physician's Global Assessment of Arthritis (PGA) (VAS) |
| | • Change from baseline in SGA (VAS) |
| | Change from baseline in subject's assessment of pain (VAS) Incidence of subject with drawed due to the leaf of officery. |
| | <ul> <li>Incidence of subject withdrawal due to the lack of efficacy</li> <li>Change from baseline in HAQ-DI score</li> </ul> |
| | <ul> <li>Change from baseline in FF-36v2® score</li> </ul> |
| | <ul> <li>Change from baseline in WPAI score</li> </ul> |
| Variables | • AEs |
| (Safety): | • Vital signs (body temperature, pulse rate, and blood pressure in a sitting |
| | position) |
| | Body weight 12 In the transport (FCC) |
| | 12-lead electrocardiogram (ECG) Control electrocardiogram |
| | <ul><li>Central electrocardiogram</li><li>Chest radiography</li></ul> |
| | Cnest radiography Laboratory assessments |
| | - Emotimory moderoniems |

| Variables | Plasma ASP015K concentration on each day of the study visit |
|---|---|
| (Pharmacokinetics): | - 1 month 1101 01012 concentration on each day of the study visit |
| Variables | Change from baseline in VEGF level |
| (Pharmacodynamics): | • Change from baseline in MMP-3 level |
| | • Change from baseline in lymphocyte subset assays (CD3, CD4, CD8, |
| | CD16, CD19, CD56, CD56/16) |
| | Additional analysis may be performed for biomarkers for efficacy and safety |
| | assessments based on study results using blood samples that have been |
| | collected during the study and biobanked (i.e., residual sample stored for retrospective analysis). These could include biomarkers of inflammation, bone |
| | or cartilage metabolism, or inhibitory activity of JAK, but other biomarkers |
| | may also be subject to analysis. |
| Pharmacogenomics | [Unique to Japan and Korea: To prepare for future research to analyze the |
| (Bio-Banking): | relationship between genes and the efficacy, safety, or pharmacokinetics of the |
| | study drug, blood samples will be collected and stored with the consent of the |
| | subject in Japan and Korea.] |
| Statistical Methods: | [Target Sample Size Calculation] |
| | The target sample size for placebo and each ASP015K treatment group was set |
| | at 100 subjects. The target sample size for the reference group was set at 200 subjects. |
| | Based on 015K-CL-RAJ1 result and efficacy result from other RA drugs |
| | [XELJANZ®, tablet, 5 mg, CTD (2013)] [CIMZIA, sc, 200 mg, Syringe, CTD |
| | (2012)], 62 subjects per group will provide 90% power to detect a difference |
| | assumed in the Step 2 in the closed testing procedure (described in Primary |
| | Efficacy Variable Analysis) under the following assumptions. In addition, it is |
| | assumed that ACR20 response rate of each region is similar: |
| | o ACR 20% response rate at Week12 in the placebo group: 25% |
| | o ACR 20% response rate at Week12 in the ASP015K 100 mg group: 54.5% |
| | o ACR 20% response rate at Week12 in the ASP015K 150 mg group: 65.5% |
| | o Two-sided significance level of 0.05 |
| | On the other hand, according to the Extent of Population Exposure to Assess |
| | Clinical Safety for Drugs Intended for Long-term Treatment of |
| | Non-life-threatening Conditions (PAB/PCD Notification No. 592, dated 24 |
| | May 1995) ("the long-term treatment guideline") and "Guidelines on |
| | methodology for clinical assessment of antirheumatic drugs" (PFSB/ELD |
| | Notification No. 0217001, dated 17 February 2006), to collect data for 300 |
| | subjects for 6 month period, and for 100 subjects for 1 year period in both |
| | ASP015K 100 mg and 150 mg groups among 015K-CL-RAJ2/RAJ3/RAJ4 |
| | studies as long term treatment data, approximately 80 subjects per treatment group are necessary to be enrolled in Japan. In addition, the target sample size |
| | for Taiwan is set at 10 subjects per treatment group in consideration of the |
| | requirement of regulatory authority in Taiwan (10% or more Taiwan subjects) |
| | and target sample size for Korea is also set at 10 subjects per treatment group. |
| | Therefore, the target sample size per treatment group is set at 100 subjects in |
| | total for 3 regions. |
| | In addition to ASP015K and Placebo group, etanercept was set as open-label |
| | reference group and its target sample size is 200 subjects, considering the |
| | followings. |
| | O Incidence rates for serious infections from post marketing studies for |
| | approved biologic drugs [ACTEMRA®, drip infusion, 80 mg, 200 mg, 400 mg, final reports for all patients ] [ORENCIA®, drip infusion, |
| | 250 mg, information for appropriate drug usage] [HYUMIRA®, sc, |
| | 40 mg, Syringe 0.8 mL, information for appropriate drug usage] |
| | [XELJANZ®, tablet, 5 mg, CTD (2013)] |
| L | [12201112 , words, 5 mg, 612 (2013)] |

| | o Operational feasibility |
|---|---|
| Statistical Methods: | Setting the sample size of reference group as 200, it can be detectable at least 1 subject with 95% confidence probability for AE which occurs at 1.5% incidence rate. |
| | [Primary Efficacy Variable Analysis] For the ACR20 response at Week 12/ET as primary efficacy variable, pairwise comparisons to placebo will be performed at each ASP015K dose level using logistic regression model with treatment group (Placebo, ASP015K 100 mg, and ASP015K 150 mg) as the factor and the prior biologic-DMARD-IR, concomitant DMARD use during the study period, and study region (Japan, Korea and Taiwan) as the covariates. For multiplicity adjustment, following closed testing procedure will be done. Step 1.ACR20 response at Week 12/ET: ASP015K 150 mg vs. Placebo Step 2.ACR20 response at Week 12/ET: ASP015K 100 mg vs. Placebo The null hypotheses will be tested at a significance level of 0.05. For the missing data imputation of ACR20 at Week 12/ET, Last Observation Carried Forward (LOCF) methodology will be used. |
| | [Secondary Efficacy Variable Analysis] For secondary efficacy endpoints, binary variables such as Percentage of subjects achieving ACR50 response at Week 12/ET, and Percentage of subjects achieving ACR70 response at Week 12/ET will be analyzed using logistic regression model as described in the primary analysis with treatment group as the factor, and the prior biologic-DMARD-IR, concomitant DMARD use during the study period and study region (Japan, Korea and Taiwan) as the covariates. Continuous variables, such as Change from baseline/Day 1 to Week 12/ET in DAS28-CRP and DAS28-ESR scores, will be analyzed using analysis of covariance (ANCOVA) with treatment group as factor, and the prior biologic-DMARD-IR, concomitant DMARD use, study region (Japan, Korea and Taiwan) and baseline value as the covariates. Each ASP015K group will be compared with placebo group and multiplicity for the secondary efficacy variables will not be adjusted. [Safety and Other Variables Analyses] Summary statistics will be calculated for trough levels and biomarker concentrations by dose and time point. AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). The incidence of AEs, serious AEs (SAEs), AEs leading to |
| | discontinuation, and AEs related to study drug will be summarized. All AEs will be listed. Descriptive statistics for laboratory values, vital signs, body weight, 12-lead ECG results, QT variables (including QTc) and their changes from baseline over time will be provided. |

# V. FLOW CHART AND SCHEDULE OF ASSESSMENTS

#### Flow Chart





Sponsor: Astellas Pharma Inc.

ISN/Protocol <015K-CL-RAJ3>

**Table 1: Schedule of Assessment** 

| Visit | Initiation<br>of<br>Screening <sup>1)</sup> | Screening<br>Test<br>Period | 0<br>W | 4<br>W | 8<br>W | 12<br>W | 16<br>W | 20<br>W | 24<br>W | 28<br>W | 32<br>W | 36<br>W | 40<br>W | 44<br>W | 48<br>W | 52<br>W | Early<br>Termination | Follow-up <sup>2)</sup> | Unscheduled<br>Visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit day | -1 at latest | -28 to -1 | 1 | 29 | 57 | 85 | 113 | 141 | 169 | 197 | 225 | 253 | 281 | 309 | 337 | 365 | Within 2<br>days of<br>withdrawal | 28 days after<br>Week 52 or<br>early<br>termination<br>visit | - |
| Allowable range from specified date | | | | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | +2 | ±7 | - |
| Informed consent | 0 | | | | | | | | | | | | | | | | | | |
| Inclusion/exclusion<br>criteria | 0 | 0 | 0 | | | | | | | | | | | | | | | | |
| Subject registration | 0 | | 0 | | | 0 | | | | | | | | | | 0 | 0 | 0 | |
| Confirmation of<br>DMARD-IR | 0 | | 0 | | | | | | | | | | | | | | | | |
| Demographics | 0 | 0 | 0 | | | | | | | | | | | | | | | | |
| Medical history | 0 | 0 | 0 | | | | | | | | | | | | | | | | |
| Height | | 0 | | | | | | | | | | | | | | | | | |
| Tuberculin test | | 0 | | | | | | | | | | | | | | | | | |
| Safety | | | | | | | | | | | | | | | | | | | |
| Physical examination | | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | <b>A</b> |
| Body weight | | 0 | | | | 0 | | | | 0 | | | 0 | | | 0 | 0 | 0 | <b>A</b> |
| Vital signs | | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | <b>A</b> |
| Hepatitis examination | | 0 | | | | | | | | | | | | | | | | | <b>A</b> |
| Hematology <sup>3)</sup> | | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | <b>A</b> |
| Biochemistry <sup>3)</sup> | | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | <b>A</b> |
| Urinalysis <sup>3)</sup> | | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | <b>A</b> |
| Fasting lipid profile test | | | 0 | | | 0 | | 0 | | 0 | | | 0 | | | 0 | 0 | 0 | <b>A</b> |
| Chest radiography | | 0 | | | | | | | | 0 | | | | | | 0 | <b>A</b> | | <b>A</b> |
| 12-lead ECG | | 0 | | | | | | | | 0 | | | | | | 0 | 0 | | <b>A</b> |
| Central ECG <sup>4)</sup> | | | 0 | С | 6) | | | | | | | | | | | | | | |
| Pregnancy test <sup>5)</sup> | | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | <b>A</b> |

| Visit | Initiation<br>of<br>Screening <sup>1)</sup> | Screening<br>Test<br>Period | 0<br>W | 4<br>W | 8<br>W | 12<br>W | 16<br>W | 20<br>W | 24<br>W | 28<br>W | 32<br>W | 36<br>W | 40<br>W | 44<br>W | 48<br>W | 52<br>W | Early<br>Termination | Follow-up <sup>2)</sup> | Unscheduled<br>Visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit day | -1 at latest | -28 to -1 | 1 | 29 | 57 | 85 | 113 | 141 | 169 | 197 | 225 | 253 | 281 | 309 | 337 | 365 | Within 2<br>days of<br>withdrawal | 28 days after<br>Week 52 or<br>early<br>termination<br>visit | - |
| Allowable range from specified date | | | | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | +2 | ±7 | - |
| Adverse events | | | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | <b>A</b> |
| Efficacy | | | | | | | | | | | | | | | | | | | |
| CRP and ESR | | O<br>(CRP<br>only) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | <b>A</b> |
| TJC/SJC (68/66 joints) | | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | <b>A</b> |
| PGA (VAS), SGA<br>(VAS), and<br>subject's assessment of<br>pain (VAS) | | | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | <b>A</b> |
| SF-36 v2® | | | 0 | 0 | 0 | 0 | | | | 0 | | | | | | 0 | 0 | 0 | <b>A</b> |
| WPAI | | | 0 | 0 | 0 | 0 | | | | 0 | | | | | | 0 | 0 | 0 | <b>A</b> |
| HAQ-DI | | | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | <b>A</b> |
| PK/PD | | | | | | | | | | | | | | | | | | | <b>A</b> |
| Blood sampling for trough concentration <sup>4)</sup> | | | 0 | 0 | 0 | 0 | | | | 0 | | | | | | 0 | 0 | | |
| Blood sampling for<br>post-dose drug<br>concentration <sup>4)</sup> | | | | ( | ) | | | | | | | | | | | | | | |
| Blood sampling for PD (biomarkers) | | | 0 | 0 | 0 | 0 | | | | 0 | | | | | | 0 | 0 | 0 | <b>A</b> |
| Blood sampling for PD (lymphocyte subset) | | | 0 | 0 | 0 | 0 | | | | 0 | | | | | | 0 | 0 | 0 | <b>A</b> |
| Informed consent for PGx research (relevant sites only) <sup>4)</sup> | | | 0 | | | | | | | | | | | | | | | | |
| Blood sampling for PGx (relevant sites only) <sup>4)</sup> | | | 0 | | | | | | | | | | | | | | | | |

| Visit | Initiation<br>of<br>Screening <sup>1)</sup> | Screening<br>Test<br>Period | 0<br>W | 4<br>W | 8<br>W | 12<br>W | 16<br>W | 20<br>W | 24<br>W | 28<br>W | 32<br>W | 36<br>W | 40<br>W | 44<br>W | 48<br>W | 52<br>W | Early<br>Termination | Follow-up <sup>2)</sup> | Unscheduled<br>Visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit day | -1 at latest | -28 to -1 | 1 | 29 | 57 | 85 | 113 | 141 | 169 | 197 | 225 | 253 | 281 | 309 | 337 | 365 | Within 2<br>days of<br>withdrawal | 28 days after<br>Week 52 or<br>early<br>termination<br>visit | - |
| Allowable range from specified date | | | | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | +2 | ±7 | - |
| Study drug/reference drug | | | | | | | | | | | | | | | | | | | |
| Confirmation of remaining unused drugs | | | | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | | |
| Prescription | | | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | | | | |

The symbol "○" designates mandatory items, whereas the symbol "▲" denotes the optional items to be investigated on the basis of the clinical judgment of the investigator/sub-investigator.

For details, see the respective sections of the protocol.

- 1) Subjects who have signed the informed consent will undergo evaluation of DMARD response at the screening visit.
- 2) Follow-up will not be performed for subjects starting the extension study immediately after the Week 52 visit.
- 3) For details of the test parameters, refer to Section 5.4.4.
- 4) Subjects in the reference group will not undergo these procedures.
- 5) For pregnancy tests, serum samples will be used at the screening visit, and urine samples will be used at and after the baseline visit.
- 6) Central ECG should be performed on the same day as blood sampling for post-dose drug concentration at Week 4 or Week 8 before and after study drug administration.

# VI. ACCEPTABLE RANGE OF SCHEDULE OF ASSESSMENTS

The paragraphs that follow describe the allowable time windows on scheduled test and observation dates.

Reasonable efforts must be made to perform the tests and observations specified for early termination and follow-up, even if they cannot be conducted within the allowable time frame.

# [Acceptable Time Ranges for Efficacy Tests]

TJC/SJC (68/66 joints) and CRP

| Screening | From 1 to 28 days prior to the baseline visit. |
|---|---|
| Baseline | Before the initiation of treatment with the study |
| Basefille | drug or reference drug on the baseline visit day. |
| Study visits from West 1 to | Within $\pm$ 7 days of the protocol-specified date |
| Study visits from Week 4 to Week 48 | <b>AND</b> before the initiation of treatment with the |
| Week 46 | study drug or reference drug on the visit day. |
| Week 52 | Within $\pm$ 7 days of the protocol-specified date. |
| Early termination | Within 2 days of withdrawal. |
| Follow-up | Within $\pm$ 7 days of the date 28 days after the Week |
| Follow-up | 52 <b>OR</b> early termination visit. |

# PGA (VAS), SGA (VAS), Subject's Assessment of Pain (VAS), HAQ-DI, and ESR

| Baseline | Before the initiation of treatment with the study drug or reference drug on the baseline visit day. |
|---|---|
| Study visits from Week 4 to<br>Week 48 | Within ± 7 days of the protocol-specified date <b>AND</b> before the initiation of treatment with the study drug or reference drug on the visit day. |
| Week 52 | Within $\pm$ 7 days of the protocol-specified date. |
| Early termination | Within 2 days of withdrawal. |
| Follow-up | Within ± 7 days of the date 28 days after the Week 52 <b>OR</b> early termination visit. |

## Sponsor: Astellas Pharma Inc.


SF-36 v2<sup>®</sup>, WPAI

| Baseline | Before the initiation of treatment with the study drug or reference drug on the baseline visit day. |
|---|---|
| Weeks 4, 8, 12, and 28 | Within ± 7 days of the protocol-specified date <b>AND</b> before the initiation of treatment with the study drug or reference drug on the visit day. |
| Week 52 | Within $\pm$ 7 days of the protocol-specified date. |
| Early termination | Within 2 days of withdrawal. |
| Follow-up | Within ± 7 days of the date 28 days after the Week 52 <b>OR</b> early termination visit. |

# [Acceptable Time Ranges for Safety Tests]

Physical Examination, Vital Signs, Laboratory Tests [Hematology, Serum Biochemistry, Urinalysis, Pregnancy Test (serum/urine)]

| Screening | From 1 to 28 days prior to the baseline visit. |
|---|---|
| Baseline | Before the initiation of treatment with the study |
| | drug or reference drug on the baseline visit day. |
| Study visits from Week 4 to Week 48 | Within $\pm$ 7 days of the protocol-specified date |
| | <b>AND</b> before the initiation of treatment with the |
| | study drug or reference drug on the visit day. |
| Week 52 | Within $\pm$ 7 days of the protocol-specified date. |
| Early termination | Within 2 days of withdrawal. |
| Follow-up | Within $\pm$ 7 days of the date 28 days after the Week |
| | 52 <b>OR</b> early termination visit. |

# Body Weight

| Screening | From 1 to 28 days prior to the baseline visit. |
|---|---|
| Weeks 12, 28, and 40 | Within ± 7 days of the protocol-specified date <b>AND</b> before the initiation of treatment with the study drug or reference drug on the visit day. |
| Week 52 | Within $\pm$ 7 days of the protocol-specified date. |
| Early termination | Within 2 days of withdrawal. |
| Follow-up | Within ± 7 days of the date 28 days after the Week 52 <b>OR</b> early termination visit. |
# Sponsor: Astellas Pharma Inc.


# Fasting Lipid Profile Test

| | Before the initiation of treatment with the study |
|---|---|
| Baseline | drug or reference drug on the baseline visit day |
| | <b>AND</b> 8 or more hours after the last meal. |
| | Within $\pm$ 7 days of the protocol-specified date |
| Weeks 12, 20, 28, and 40 | Before the initiation of treatment with the study |
| Weeks 12, 20, 28, and 40 | drug or reference drug on the study visit day <b>AND</b> |
| | 8 or more hours after the last meal. |
| Wools 52 | Within $\pm$ 7 days of the protocol-specified date |
| Week 52 | <b>AND</b> 8 or more hours after the last meal. |
| | Within 2 days after withdrawal <b>AND</b> 8 or more |
| Early termination | hours after the last meal (the nutritional condition |
| | is recommended but not compulsory). |
| Follow-up | Within $\pm$ 7 days of the date 28 days after the Week |
| | 52 <b>OR</b> early termination visit. |

# Chest Radiography

| Screening | From 1 to 28 days prior to the baseline visit. Radiographs taken before the informed consent will be acceptable as long as they were taken within 90 days before the baseline visit. |
|---|---|
| Weeks 28 and 52 | Within $\pm$ 7 days of the protocol-specified date. |
| Early termination | Within 2 days of withdrawal. Not mandatory; may be required at the discretion of the investigator/sub-investigator. |

# 12-lead ECG

| Screening | From 1 to 28 days prior to the baseline visit. |
|---|---|
| Week 28 | Within ± 7 days of the protocol-specified date <b>AND</b> before the initiation of treatment with the study drug or reference drug on the visit day. |
| Week 52 | Within $\pm$ 7 days of the protocol-specified date. |
| Early termination | Within 2 days of withdrawal. |

## Sponsor: Astellas Pharma Inc.


# Central ECG (except for the reference group)

| Baseline | Before the initiation of treatment with the study drug on the baseline visit day |
|---|---|
| Week 4 or 8 | |
| | Within $\pm$ 7 days of the protocol-specified date |
| (before study drug | AND before the initiation of treatment with the |
| administration) | study drug on the visit day. |
| Week 4 or 8<br>(after study drug<br>administration) | Within $\pm$ 7 days of the protocol-specified date |
| | AND 2-hour post-dose on the visit day |
| | (Recommended time point. Sampling from 1 hour |
| | to 4 hours post-dose will be acceptable.) |

[Acceptable Time Ranges for PD Tests: Biomarker and Lymphocyte Subset

**Measurements**]

| Baseline | Before the initiation of treatment with the study drug or reference drug on the baseline visit day. |
|---|---|
| Weeks 4, 8, 12, and 28 | Within ± 7 days of the protocol-specified date <b>AND</b> before the initiation of treatment with the study drug or reference drug on the visit day. |
| Week 52 | Within $\pm$ 7 days of the protocol-specified date. |
| Early termination | Within 2 days of withdrawal. |
| Follow-up | Within ± 7 days of the date 28 days after the Week 52 <b>OR</b> early termination visit. |

# [Acceptable Time Ranges for Blood Sampling for Plasma Drug Concentration]

Trough Concentration (except the reference group)

| Baseline | Before the initiation of treatment with the study drug on the baseline visit day. |
|---|---|
| | • |
| Weeks 4, 8, 12, 28, and 52 | Within $\pm$ 7 days of the protocol-specified date |
| | <b>AND</b> within 19 to 29 hours between the time of |
| | treatment with the study drug before blood |
| | collection and the time of blood collection. |
| Early termination | Within 2 days after withdrawal. |

Post-Dose Drug Concentration (except the reference group)

| Week 4 or 8 | The recommended time point is 2 hours post-dose. Sampling from 1 hour to 4 hours post-dose will be |
|---|---|
| | acceptable. |

## 1 INTRODUCTION

## 1.1 Background

Rheumatoid arthritis (RA) is a chronic systemic inflammatory autoimmune disease that targets the synovial tissues [O'Dell, 2004]. The synovial inflammation is associated with irreversible cartilage destruction and erosion of bone, which may cause pain as well as decreased activity of daily living (ADL) due to functional impairment, and therefore reduce quality of life (QOL). The goal of RA treatment is to control the disease activity and achieve remission by preventing or controlling joint destruction, preventing loss of function, and relieving pain, thereby improving patient QOL.

Conventional RA treatments have been based on pain control with nonsteroidal anti-inflammatory drugs and inflammation control with corticosteroids, with which disease-modifying antirheumatic drugs (DMARDs) have been combined [Nakajima, 2009]. After the approval of methotrexate (MTX) and biologics, RA treatment improved greatly, shifting its goal from pain control to induction and maintenance of remission. In more recent years, the ultimate goal of RA therapy evolved to include clinical, structural, and functional remission. Now, researchers are attempting to achieve drug-free remission.

In Japan, MTX has been established as the standard first-line therapy for RA. The combination of tumor necrosis factor (TNF) inhibitors and other biological agents with MTX has paved the way for the treat-to-target (T2T) approach aimed at clinical and structural remission.

However, it has been that such combination therapies induced clinical remission in approximately 30% to 50% of treated patients [Y. Tanaka, 2009; K. Yamaoka, 2008], failing to control disease in most cases. In addition, MTX, a non-specific inhibitor of cellular proliferation, frequently causes adverse drug reactions in proliferative tissues such as the gastrointestinal epithelium and bone marrow, and these reactions lead to premature discontinuation in a certain proportion of patients. TNF inhibitors (e.g., etanercept, infliximab, adalimumab), selective T-cell co-stimulation modulators (e.g., abatacept), and other biologics are very expensive and require intravenous or subcutaneous administration; the issues of cost, cumbersome dosing procedure, and other factors are a hindrance to their application. Under these circumstances, low-molecular-weight DMARDs acting on a novel molecular target have captured increasing interest from drug companies.

ASP015K is an oral Janus kinase (JAK) inhibitor discovered by Astellas Pharma. *In vitro* kinase assays demonstrated that this agent effectively inhibited JAK1, JAK2, JAK3, and tyrosine kinase 2 (TYK2). In particular, JAK3 was suppressed in a relatively selective manner. The binding of the ligand to the cytokine receptor triggers JAK activation, and activated JAK molecules in turn phosphorylate the receptor. The phosphorylation of the cytokine receptor creates a site for interaction with the signal transducer and activator of transcription (STAT). Upon JAK-induced phosphorylation, STAT forms a dimer complex and enters into the nucleus, where the STAT dimer binds with DNA to regulate gene

transcription. Because JAK3 expression is restricted to primarily hematopoietic cells, JAK3 inhibition is a desirable therapeutic target for immunosuppression in human organ transplantation and immunomodulation in autoimmune disorders [Papageorgiou and Wikman, 2004], without significantly affecting other organ systems [Kremer et al, 2009].

Xeljanz® (tofacitinib) 5 mg is a JAK inhibitor approved by the US FDA in 2012 for the treatment of adult patients with moderate to severe RA who had an inadequate response to or are intolerant of MTX. In Japan, this drug was approved in March 2013 for treating RA patients who had an inadequate response to conventional therapies.

Astellas Pharma is pursuing the development program of ASP015K for the indication of RA. In Japan, the Phase IIb dose-finding study (015K-CL-RAJ1) has been completed, and its long-term extension study (015K-CL-RAJ2, or RAJ2) is ongoing. Overseas, 2 Phase II dose-finding studies (1 with MTX and the other without MTX) have been completed, and their follow-up extension study is underway, similar to the situation in Japan. The results of 015K-CL-RAJ1 showed that ASP015K caused a significantly higher improvement in RA than placebo in terms of the ACR response rate, DAS28 score, and other efficacy variables, suggesting its usefulness for treating RA.

## 1.2 Non-clinical and Clinical Data

## 1.2.1 Nonclinical Pharmacology and Safety Pharmacology

ASP015K is a novel oral immunosuppressant that exerts it pharmacological action by relatively selectively inhibiting JAK3, a key enzyme in the IL-2 signaling pathway. *In vitro* kinase studies showed that ASP015K also inhibited JAK1, JAK2, and TYK2, although less potently than it inhibited JAK3. In a study using a rat model of adjuvant-induced arthritis, prophylactic use of ASP015K significantly suppressed the swelling of the injected limb and prevented the worsening of the bone destruction score assessed by radiography. Therapeutic administration of ASP015K in which treatment was initiated after the occurrence of pedal edema also prevented the event and reduced joint destruction scores.

In safety pharmacology studies, ASP015K showed no effect on human ether-a-go-go related gene (hERG) current or action potential duration in isolated guinea pig papillary muscles at clinically relevant concentrations. ASP015K had no effect on the central nervous system (modified Irwin's method) of rats at up to 100 mg/kg orally. In monkeys, loose/watery stools and a tendency towards reduced blood potassium concentrations were observed at 60 mg/kg orally, but there were no effects on the central nervous system, cardiovascular system [electrocardiogram (ECG), blood pressure, or heart rate], or respiratory system of monkeys at up to 60 mg/kg.

## 1.2.2 Pharmacokinetics and Pharmacodynamics

#### 1.2.2.1 Nonclinical Pharmacokinetics

Absolute bioavailability ranged from 39.8% to 46.4% in rats and 18.9% to 19.2% in monkeys. Following a single oral dose of 3 mg/kg <sup>14</sup>C-ASP015K in Sprague-Dawley rats, radioactivity

distributed rapidly into tissues with no long-term tissue retention observed. In a study with pigmented rats, the dosed radioactivity was rapidly excreted within the first 24 hours after administration in almost all tissues with the exception of the eyeball (t<sub>1/2</sub> of 1105.8 hours). No apparent differences were noted in radioactivity concentration-time profiles between nonpigmented and pigmented skin, and the radioactivity was not detected in these skins for a long time. These data suggest that ASP015K-related compounds may have bound to melanin, but binding was likely weak and reversible. In Sprague-Dawley rats orally administered <sup>14</sup>C-ASP015K 3 mg/kg once daily for 21 days, radioactivity was slowly eliminated from the lung, spleen, skin, bone marrow, testis, and thoracic aorta. With the exception of the thoracic aorta, the radioactivity levels 168 hours after the last dose were reduced to 19% or less of the levels measured 0.25 hours after the last dose. The mean radioactivity of the thoracic aorta at 168 hours of the last dose was as low as less than 3 times the lower limit of quantification.

The *in vitro* plasma protein binding rates of ASP015K and its metabolite AS2628528 (H2) were determined in the concentration range of  $0.2–20~\mu g/mL$ . The plasma protein binding rates in mice, rats, rabbits, dogs, monkeys, and humans were in the ranges of 59%–95% for ASP015K and 84%–99% for H2. Among human plasma proteins, human serum albumin (HSA) most preferentially bound to ASP015K and H2.

In pregnant and lactating rats administered a single oral dose of <sup>14</sup>C-ASP015K 3 mg/kg, the radioactivity was distributed widely across different tissues of the dams, although the tissue radioactivity almost completely disappeared within 24 hours. Although the levels of placental radioactivity transfer were low, comparatively higher levels of radioactivity were rapidly transferred to the milk, leading to elevated radioactivity in pups via lactation.

When <sup>14</sup>C-ASP015K was orally administered alone to rats at a dose of 3 mg/kg, 3 radioactivity peaks were detected in plasma on the radiochromatogram, with the main peak being that of the unchanged drug. *In vitro* metabolic profile of <sup>14</sup>C-ASP015K was performed in liver microsomes and cryopreserved hepatocytes from mice, rats, rabbits, dogs, cynomolgus monkeys, and humans. No human-specific metabolites were identified in either assay. In *in vitro* metabolic studies, ASP015K was metabolized to H2 by human sulfotransferase 2A1 (hSULT2A1) and to AS2604202 (H4) by human nicotinamide N-methyltransferase (hNNMT).

In rats orally administered a single <sup>14</sup>C-ASP015K dose, 25.2% and 46.7% of the administered radioactivity was eliminated into urine and bile at 72 hours, respectively, suggesting an excellent oral absorption profile of ASP015K. In monkeys orally administered a single <sup>14</sup>C-ASP015K dose, 22.3% and 26.4% of the administered radioactivity was eliminated into urine and bile at 72 hours, respectively.

#### 1.2.2.2 Clinical Pharmacokinetics and Pharmacodynamics

A total of 17 clinical studies of ASP015K have been completed till date. These studies included 14 pharmacokinetic studies in healthy adult volunteers, 1 pharmacokinetic study in RA patients, 1 efficacy and safety study in patients with psoriasis, and 1 efficacy and safety study in RA patients. More specifically, they were as follows: a single-dose and

repeated-dose study in Japanese and Caucasian subjects conducted in Japan (015K-CL-HV03), an overseas single ascending dose and food effect study (015K-CL-HV01), an overseas repeated-dose study (015K-CL-HV02), a mass balance study using radiolabeled ASP015K (015K-CL-PK03), a regional absorption study (015K-CL-PK15), 4 relative bioavailability and food effect studies (015K-CL-PK09, 015K-CL-PK18, 015K-CL-PK19, 015K-CL-PK51), 5 drug—drug interaction (DDI) studies in healthy adult volunteers (015K-CL-PK01, 015K-CL-PK02, 015K-CL-PK05, 015K-CL-PK16, and 015K-CL-PK26), 1 DDI study in RA patients (015K-CL-PK13), 1 efficacy and safety study in psoriasis patients (015K-CL-PS01), and 1 efficacy and safety study in RA patients (015K-CL-RAJ1).

These completed studies involved 472 healthy adults and 296 RA patients; they received ASP015K doses ranging from 3 to 300 mg/day in single-dose studies and from 10 to 200 mg twice daily (BID) in repeated-dose studies. In addition, 124 patients with psoriasis were enrolled and were administered 10 to 100 mg BID or 50 mg once daily (QD).

After a single dose of 3 to 300 mg/day administered under fasting conditions in Study 015K-CL-HV01, ASP015K was rapidly absorbed with a median t<sub>max</sub> ranging from 1.0 to 1.75 hours across the dose groups. The AUC<sub>inf</sub>, AUC<sub>last</sub>, and C<sub>max</sub> of ASP015K increased dose proportionally. Elimination occurred in a multiphasic manner with a mean t<sub>1/2</sub> value of 2.8 to 18.5 hours. Compared to administration under fasting conditions, the mean C<sub>max</sub> of ASP015K administered under fed conditions increased by 5%. Similarly, the mean AUC<sub>inf</sub> increased by 27% with t<sub>max</sub> being prolonged for approximately 2.5 hours. Urinary excretion of ASP015K accounted for between 9% and 15% of the oral dose. ASP015K inhibited JAK3-mediated phosphorylation of STAT5 dose-dependently. Peak inhibition of JAK3-mediated phosphorylation of STAT5 was observed around 1 to 2 hours (median) following administration of ASP015K under fasting conditions. At a dose of 60 mg, the peak inhibition reached 84% of the maximum. The mean changes from baseline lymphocyte counts and peripheral lymphocyte subsets suggested there were no time- or dose-dependent changes after a single oral dose of ASP015K.

Study 015K-CL-HV02, in which ASP015K was given at doses of 30 mg BID, 100 mg BID, or 200 mg BID for 14 days under non-fasting conditions, demonstrated no clear difference in pharmacokinetics of ASP015K after repeated dosing between the morning and evening doses, although the trough level after the morning dose tended to be lower. Steady state in plasma ASP015K concentrations was achieved by Day 3. The mean accumulation factor on Day 14 was between 1.12 and 1.65 for  $C_{max}$ , 1.38 and 1.65 for  $AUC_{12}$ , and 2.02 and 2.71 for  $C_{trough}$ , PM. At steady state, the peak-trough ratios (peak/trough levels) of ASP015K concentrations were between 8.8 and 18. Overall,  $C_{max}$  and  $AUC_{12}$  values generally increased dose proportionally over the range of 30 to 100 mg BID. There was no sex difference in ASP015K exposure with the 100 mg BID dose.

As a result of metabolite analysis of samples collected in 015K-CL-HV01 and 015K-CL-HV02, 3 metabolites (H1, H2, H4) were identified from plasma samples and 6 metabolites (H1 to H6) were identified from urine samples.

Results from the mass balance study (015K-CL-PK03) indicated that unchanged ASP015K accounted for 36% of the total radioactivity in plasma (metabolites accounted for the remaining 64%). Approximately 36.8% of the total radioactivity was excreted in urine and 56.6% in feces. Unchanged ASP015K accounted for 36% of the total radioactivity in urine.

In Study 015K-CL-HV03, Japanese had greater ASP015K exposure than Caucasian. After adjustment for dose and body weight,  $C_{max}$  was 42.9% to 53.9% higher and AUC<sub>inf</sub> was 22.5% to 44.9% higher in Japanese relative to Caucasian. JAK3 inhibition was dose-dependent in Japanese and Caucasian. Consistent with the generally higher plasma concentrations of ASP015K in Japanese, the peak inhibition of JAK3 following a single dose of ASP015K was also higher in Japanese. Overall, the mean change from baseline for T cell subsets was similar with ASP015K single or repeated dosing, with little variation among ethnicity.

Results from a regional absorption study (015K-CL-PK15) indicated that absorption primarily ( $\geq 50\%$ ) occurred in the proximal small bowel, and the rate and extent of absorption decreased as the delivery site became more distal within the gastrointestinal tract.

In Study 015K-CL-PK19, subjects were administered ASP015K (5 tablets of 30 mg) after a meal (approximately 500 to 600 kcal, with fat accounting for 25% to 35% of the total calories). Compared with fasting conditions, t<sub>max</sub> was extended by 0.5 hours, and C<sub>max</sub> and AUC increased by 34% and 27%, respectively.

In the 6 DDI studies, the pharmacokinetic profile of ASP015K was investigated in the presence of: mycophenolate mofetil (MMF) (015K-CL-PK01), tacrolimus (015K-CL-PK02 and 015K-CL-PK16), midazolam (015K-CL-PK05), MTX (015K-CL-PK13), and rosuvastatin (015K-CL-PK26). MMF, tacrolimus, midazolam, and rosuvastatin were administered in healthy adult volunteers, whereas MTX was used in RA patients.

Administration of ASP015K 100 mg BID had no effect on the pharmacokinetic profile of MTX in patients with RA or the MMF metabolites MPA and MPAG in healthy volunteers. ASP015K 60 mg and 100 mg BID did increase tacrolimus levels in whole blood following oral administration of tacrolimus 5 mg, but not when tacrolimus was administered as a 1 mg intravenous dose. Concomitant use of ASP015K elevated the plasma midazolam concentrations after a single oral dose of midazolam 3 mg. It also raised the plasma rosuvastatin levels following a single oral dose of rosuvastatin 10 mg. However, steady-state pharmacokinetics of ASP015K were not significantly impacted by MTX 15 to 25 mg, MMF 1 g, midazolam 3 mg, oral tacrolimus 5 mg, or intravenous tacrolimus 1 mg doses.

In Study 015K-CL-PS01 that enrolled patients with psoriasis, the administration of ASP015K 10 to 100 mg BID elevated ASP015K exposure (C<sub>max</sub>, AUC<sub>last</sub>, and AUC<sub>6h</sub>) in a dose-dependent manner. The median t<sub>max</sub> values were in the range of approximately 1.0 to 1.8 hours. STAT5 phosphorylation and JAK3 activity were inhibited in a dose-dependent manner. Although no consistent trends were noted for the absolute lymphocyte count, a slight dose-dependent decreasing trend was noted for the proportions and absolute counts of NK and B cells.

In Study 015K-CL-RAJ1 of Japanese patients with RA, matrix metalloproteinase 3 (MMP-3) levels decreased in a dose-dependent manner following the administration of ASP015K 25 to 150 mg QD. Although no consistent trends were noted for the absolute lymphocyte count, NK cell counts decreased and B cell counts increased in a dose-dependent manner.

## 1.2.3 Toxicology

Nonclinical repeated-dose toxicity studies of ASP015K were conducted using rats (up to 26 weeks) and monkeys (up to 52 weeks). Toxicities observed in these studies were mainly related to gastrointestinal, hematopoietic, muscular, and immune systems. All these findings were reversible and resolved upon the withdrawal of ASP015K. Muscle toxicity was observed in monkeys: mild multifocal muscle necrosis in 1 female at 60 mg/kg/day in the 4-week preliminary study; elevation of CPK and LDH without histopathological changes in 2 males at 60 mg/kg/day in the 4-week preliminary study; elevation of CPK and LDH without histopathological changes in 1 male that was sacrificed in extremis in 13-week study, and a transient increase of CPK without histopathological changes observed in another male in the same 13-week study.

Genotoxicity studies were conducted *in vitro* and *in vivo*. ASP015K was negative in the reverse mutation test in bacteria but was positive in an *in vitro* chromosomal aberration test in Chinese hamster lung cells. ASP015K was negative in 2 *in vivo* genotoxicity studies, the unscheduled DNA synthesis test in rats and the micronucleus test in mice. These results suggested that ASP015K had little potential to induce chromosomal aberrations in *in vivo*.

In toxicity studies on the fertility and early embryonic development in rats, the viability of embryos decreased after implantation and the number of live embryos decreased in the 100 mg/kg/day group compared with the control group. ASP015K neither induced general toxicity nor impacted male or female fertility up to the dose of 100 mg/kg/day. In an embryo–fetal development study in rats, increased incidences of skeletal abnormalities and variations and visceral variations were noted at 30 mg/kg/day and higher, while increased incidences of visceral and external abnormalities were observed at 300 mg/kg/day. NOAEL for embryo–fetal development in rats was 10 mg/kg/day. In an embryo–fetal developmental toxicity study in rabbits, no teratogenicity was observed; however, increased postimplantation loss and decreased numbers of live fetuses were noted at 10 mg/kg/day.

Four- and 13-week toxicity studies of ASP015K administered in combination with tacrolimus, MMF, or MTX demonstrated no significant synergistic toxicities.

## 1.2.4 Efficacy

In a double-blind, placebo-controlled study conducted in Japan (015K-CL-RAJ1), the dose response for the efficacy and safety of once-daily oral ASP015K (25, 50, 100, 150 mg) was investigated in 281 patients with moderate to severe RA. Its primary efficacy variable was the ACR20 response rate at Week 12. The ACR20 response rates were 10.7% for placebo, 23.6% for 25 mg, 31.6% for 50 mg, 54.5% for 100 mg, and 65.5% for 150 mg groups. Significant improvements over placebo were noted for 50 mg (P=0.021), 100 mg (P<0.001), and 150 mg groups (P<0.001). In addition, logistic regression analysis demonstrated a

statistically significant dose–response relationship (P<0.001). Secondary efficacy variables, the ACR50 response rate, ACR70 response rate, and DAS28-CRP, exhibited significant improvements for ASP015K over placebo. A long-term extension study (015K-CL-RAJ2) for patients who completed this study is underway to investigate the efficacy and safety of ASP015K administered over an extended period of time.

Overseas, 3 clinical studies of patients with moderate to severe RA have been completed (015K-CL-RA21, 015K-CL-RA22, 015K-CL-RA25). 015K-CL-RA21 and 015K-CL-RA22 were dose-finding studies of ASP015K administered with and without MTX, respectively. 015K-CL-RA25 was a long-term follow-up extension study that enrolled the patients who completed either of the 2 studies.

In a US double-blind, placebo-controlled study in patients with moderate to severe psoriasis vulgaris (015K-CL-PS01), 124 subjects were orally administered ASP015K (10, 25, 60, 100 mg BID or 50 mg QD) over 6 weeks. Compared with placebo, all ASP015K groups showed greater improvements in terms of change from baseline in the PASI score (primary efficacy variable), depicting a statistically significant difference in the overall therapeutic response. For secondary efficacy variables, the treatment success based on Physician's Static Global Assessment (PSGA) and 75% reduction in the PASI score (PASI 75 response) demonstrated the efficacy of ASP015K.

# 1.3 Summary of Key Safety Information for Study Drugs

The safety and tolerability of ASP015K were evaluated in 14 studies in healthy adult volunteers (13 overseas and 1 Japanese), 2 studies in RA patients (1 each overseas and Japanese), and 1 study in patients with psoriasis (overseas). In these studies, a single dose of 3 to 300 mg and repeated doses of 10 to 200 mg BID were administered in 423 healthy adults and 14 RA patients. In addition, 225 RA patients received repeated doses of 25 to 150 mg QD, and 95 psoriasis patients received repeated doses of 10 to 200 mg BID or 50 mg QD.

Treatment emergent adverse events (TEAEs) that occurred relatively frequently in these studies included gastrointestinal disorders (e.g., diarrhoea, nausea, flatulence, vomiting) and nervous system disorders (e.g., headache).

In the overseas single-dose study (015K-CL-HV01), there was no evidence of clinically significant safety findings in subjects who received single oral doses of ASP015K (3, 10, 30, 60, 120, 200 and 300 mg) under fasted conditions or a single 120 mg oral dose in the fed state. The more common TEAEs in this study that occurred in multiple subjects were headache (7 subjects; moderate in 1 subject and mild in 6 subjects); mild, tension headache (3 subjects); flatulence (3 subjects; moderate in 1 subject and mild in 2 subjects); and mild, asymptomatic bradycardia (2 subjects).

In the overseas repeat-dose study (015K-CL-HV02), the more common TEAEs in the 36 subjects receiving ASP015K were neutropenia (14 subjects; severe in 1 subject, moderate in 3 subjects, and mild in 10 subjects); headache (7 subjects; moderate in 2 subjects and mild in 5 subjects); mild, abdominal pain (6 subjects); mild, diarrhoea (4 subjects); and nausea (4

subjects; moderate in 1 subject and mild in 3 subjects). Dose-dependent gastrointestinal disorders (e.g., nausea, diarrhoea, dyspepsia, and abdominal pain) and neutropenia were observed, especially in approximately two-thirds of subjects (6 of 9 subjects) in the highest dose group (ASP015K 200 mg BID). In this repeat-dose study, 2 subjects experienced severe TEAEs and 8 experienced moderate TEAEs. Severe TEAEs included elevated lipase and CPK elevation that occurred in 1 male subject (200 mg BID group) and neutropenia in 1 female subject (100 mg BID group).

In the single-dose and repeated-dose study in Japanese and Caucasian volunteers (015K-CL-HV03), the only TEAE observed in at least 1 subject after a single dose of ASP015K was mild white blood cell count increased in 2 of 6 Japanese subjects receiving ASP015K 60 mg and 1 of 6 Japanese subjects receiving ASP015K 200 mg. TEAEs observed in at least 1 subject who received repeated doses of ASP015K were mild neutrophil count decreased in 3 of 6 Japanese male subjects receiving ASP015K 100 mg BID; mild white blood cell count increased in 2 of 6 Japanese male subjects receiving ASP015K 30 mg BID and 1 of 6 Japanese male subjects receiving ASP015K 10 mg BID; and mild alanine aminotransferase increased in 1 of 6 Japanese male subjects receiving ASP015K 10 mg BID.

There were no vital sign or ECG findings observed in subjects following administration of ASP015K in the previous clinical pharmacology studies that were considered clinically relevant, except mild, asymptomatic bradycardia (possibly related; recovered) in 2 subjects in the overseas single-dose study (015K-CL-HV01), and intermittent, mild arrhythmia (not related; recovered) lasting for approximately 5 hours in 1 subject after a single dose of ASP015K 100 mg in the DDI study of ASP015K with midazolam (015K-CL-PK05).

DDI studies involving MTX, MMF, midazolam, tacrolimus, and rosuvastatin (015K-CL-PK01, 015K-CL-PK02, 015K-CL-PK05, 015K-CL-PK13, 015K-CL-PK16, 015K-CL-PK26) demonstrated that ASP015K administered in combination with these agents was well tolerated, and reported TEAE incidence rates comparable with those documented for ASP015K as single-agent therapy.

In the Japanese clinical trial in RA patients (015K-CL-RAJ1), the incidence rates of AEs in the ASP015K 25 mg, 50 mg, 100 mg, and 150 mg groups were 70.9%, 64.9%, 52.7%, and 67.2%, respectively. These rates were comparable with that of the placebo group (64.3%). The incidence rates of AEs whose relationship to the study drug could not be ruled out for the ASP015K 25 mg, 50 mg, 100 mg, and 150 mg groups were 38.2%, 43.9%, 29.1%, and 55.2%, respectively. These rates were higher than that reported for the placebo group (28.6%). By severity (NCI-CTCAE), most were either Grade 1 or Grade 2. In the placebo and ASP015K 25 mg, 50 mg, 100 mg, and 150 mg groups, the numbers of subjects with serious adverse events (SAEs) were 1 (1.8%), 1 (1.8%), 2 (3.5%), 3 (5.5%), and 0, respectively. Death was reported from 1 subject of the 50 mg group (cerebral haemorrhage). AEs resulted in treatment discontinuation in 10 (17.9%), 7 (12.7%), 5 (8.8%), 6 (10.9%), and 4 (6.9%) subjects of the placebo, ASP015K 25 mg, 50 mg, 100 mg, and 150 mg groups, respectively. The most common reason was rheumatoid arthritis aggravated (21/32).

Rheumatoid arthritis, nasopharyngitis, blood creatine phosphokinase (CPK) increased, diarrhoea, cystitis, constipation, stomatitis, dyspepsia, lipids increased, and blood triglycerides increased were reported at ≥ 5% incidence rates from 1 or more groups. By the MedDRA System Organ Class (SOC), Infections and infestations, Gastrointestinal disorders, Musculoskeletal and connective tissue disorders, and Investigations showed high incidence rates. Blood creatine phosphokinase increased were observed in 0, 2 (3.6%), 1 (1.8%), 1 (1.8%), and 7 (12.1%) subjects of the placebo, ASP015K 25 mg, 50 mg, 100 mg, and 150 mg groups, respectively. Most cases were transient, and all subjects except 1 who prematurely discontinued the study recovered or were recovering. With regard to clinical laboratory testing, compared with the placebo group, the ASP015K groups showed decreased levels of neutrophils, platelets, and estimated glomerular filtration rate (eGFR) and elevated levels of CPK, hemoglobin, lymphocytes, creatinine, total cholesterol, LDL, HDL, and triglycerides. No noteworthy changes were detected in vital signs or ECG recordings.

In the overseas study in psoriasis patients (015K-CL-PS01), none of the AEs observed were apparently dose-dependent, although the overall incidence of AEs in patients receiving ASP015K was higher than in those receiving placebo. No SAEs were reported. However, 1 subject treated with 60 mg BID prematurely discontinued the study owing to mild neutrophil count decreased, and this case was judged possibly related to the study drug. The more common AEs were pharyngitis, diarrhoea, and flatulence, which did not occur more frequently in a specific treatment group including the placebo group. Mild neutrophil count decreased was observed in patients receiving ASP015K, with none having neutrophil count of less than 1000/mm³. The mean CPK level increased with dose. A total of 4 AEs of increased CPK were reported, each in the placebo, 10 mg BID, 25 mg BID, and 100 mg BID groups, none of which were associated with symptoms suggestive of myopathy. During this study, no anaemia occurred. While mild to moderate increases in HDL, triglycerides, and total cholesterol were observed, there was no change from baseline in LDL.

For more information regarding the efficacy and safety of ASP015K, refer to the current version of the Investigator's Brochure.

For more information regarding the efficacy and safety of etanercept, refer to the current version of the package insert.

## 1.4 Risk-Benefit Assessment

Findings from nonclinical studies of ASP015K suggest that the primary areas of toxicity are the gastrointestinal system, hematopoietic system, and muscle tissue. The commonly observed AEs during clinical studies conducted to date included reversible neutrophil count decreased, gastrointestinal disorders (e.g., diarrhoea, nausea, flatulence, vomiting), CPK elevations without evidence of myopathy, and headache. In the clinical trial of ASP015K in Japanese patients with RA (015K-CL-RAJ1), 1 or more groups reported rheumatoid arthritis, nasopharyngitis, blood creatine phosphokinase increased, diarrhoea, cystitis, constipation, stomatitis, dyspepsia, lipids increased, and blood triglycerides increased at incidence rates of

 $\geq$  5%. By the MedDRA System Organ Class (SOC), Infections and infestations, Gastrointestinal disorders, Musculoskeletal and connective tissue disorders, and Investigations showed high incidence rates. Thus, these events may occur in the present study.

In the 015K-CL-QT01 study to evaluate the effect of ASP015K on cardiac function (QT interval), single doses of ASP015K 150 mg and 450 mg shortened the QTcF interval (QT interval corrected using Fridericia's Correction). The maximum decrease in the mean change from placebo- and baseline-adjusted QTcF occurred at 2 and 4 hour post dose with values of -12.0 and -14.7 msec for the 150 mg and 450 mg treatments, respectively. Therefore, shortened QT interval may be observed in the present study. The risk of drug-induced QT shortening is uncertain.

Because ASP015K is an immunosuppressive agent, it may increase the risk of infections and reactivation of latent, chronic infections. In particular, excessive immunosuppression can lead to serious infections. Of note is the fact that Xeljanz<sup>®</sup> (tofacitinib) 5 mg, a member of the class of JAK inhibitors to which ASP015K belongs, has been associated with new onset or aggravation of serious infections such as tuberculosis, pneumonitis, sepsis, viral infections, and opportunistic infectious diseases including fungal infections. In addition, several cases of malignant tumors have been reported, although their causal relation to the agent has not been established. Based on the data pooled from 5 domestic and overseas comparative studies of Xeljanz<sup>®</sup> (tofacitinib) 5 mg, the incidence density of malignancies (excluding non-melanoma skin cancers) among RA patients treated with 5 mg BID for a maximum of 1 year was 0.55/100 person-years (incidence rate 0.5% < 5/1216) [Xeljanz<sup>®</sup> Pharmaceutical Interview Form (in Japanese)].

These findings suggest that investigators pay particular attention to the possible development of infections and malignancies and take appropriate measures. Three cases of malignancies (stomach cancer, uterine sarcoma, chronic myelogenous leukemia) have been reported as of the cut-off date of 5 December 2013, from completed and ongoing national and international studies of ASP015K. Only the case of uterine sarcoma was judged as related to ASP015K.

In the Japanese clinical trial in patients with moderate to severe RA (015K-CL-RAJ1), 50 mg and higher doses of ASP015K significantly improved the ACR20 response rate versus placebo. Xeljanz<sup>®</sup> (tofacitinib) 5 mg, which acts via the same mechanism as ASP015K, was approved by the US FDA in 2012 for the treatment of adult patients with moderate to severe RA who had an inadequate response to or are intolerant of MTX. In March 2013, Xeljanz<sup>®</sup> (tofacitinib) 5 mg tablets was authorized for marketing in Japan for treating RA patients who had an inadequate response to conventional therapies. Therefore, a potential benefit of JAK inhibitor ASP015K is to improve RA.

One can also expect that long-term use of ASP015K will improve QOL of RA patients by successfully controlling the RA disease activity over an extended period.

3 March 2017 Astellas 

## 2 STUDY OBJECTIVE(S), DESIGN, AND VARIABLES

## 2.1 Study Objectives

The objectives of this study are to verify the superiority of ASP015K alone or in combination with DMARDs over placebo in terms of efficacy, at doses of 100 mg/day and 150 mg/day, in patients with rheumatoid arthritis (RA) who had an inadequate response to DMARDs, as measured by the ACR20 response rate at Week 12, which is the primary variable; to evaluate the pharmacokinetics, pharmacodynamics, and safety of ASP015K; and to evaluate the efficacy and safety of long-term treatment with ASP015K (52 weeks).

# 2.2 Study Design and Dose Rationale

## 2.2.1 Study Design

This is a Japanese, Korean and Taiwanese, multi-center, randomized, placebo-controlled, double-blind, parallel-group, confirmatory study to evaluate the efficacy and safety of ASP015K alone or in combination with DMARDs, at doses of 100 mg/day and 150 mg/day, in patients with RA who had an inadequate response to DMARDs. Open-label etanercept will also be administered as the reference drug for 52 weeks (the last dose will be given at Week 51). In the study, ASP015K (test drug) and placebo (comparative drug) will be given as study drugs, and etanercept will be given as a separate reference drug. DMARD response is evaluated at the initiation of screening and then after the screening period, subjects will be randomized in a 1:1:1:2 ratio to the ASP015K 100 mg, ASP015K 150 mg, placebo, or reference groups, and they will receive either the study drug or reference drug for 52 weeks. Subjects in the ASP015K 100 mg, ASP015K 150 mg, and placebo groups will orally receive either ASP015K or placebo once daily after breakfast, while those in the reference group will receive 50 mg of subcutaneous etanercept once weekly.

The planned sample size is 100 subjects each for the ASP015K 100 mg, ASP015K 150 mg, and placebo groups and 200 subjects for the reference group.

Re-screening is allowed only in situations in which a subject underwent the screening procedures (i.e., scans and laboratory work) and owing to logistical circumstances, the allocated time window for these tests has expired. Re-screening is not permitted in cases in which the initial test results do not support eligibility based on inclusion and exclusion criteria. The subject must be classified as a screening failure at that time point.

Any subject found not to meet the inclusion criterion (CRP) is permitted to undergo retest only once during the screening period. This however only applies to cases in which the CRP value measured at screening exceeds 0.30 mg/dL and the most resent CRP value measured at least 28 days before the screening procedures exceeds 0.5 mg/dL.

Based on the consideration of the ethical issues related to long-term placebo use, at Week 12 subjects in the placebo group will be switched to either ASP015K 100 mg or ASP015K 150 mg, and the dosage will be maintained until the end of treatment. The ASP015K dose

that will be started for placebo group subjects at Week 12 (100 or 150 mg) will be randomly chosen at baseline. The dose will be switched under the blinded condition.

Subjects in the ASP015K 100 mg, ASP015K 150 mg, or placebo groups who complete this study will be eligible for participation in the open-label extension study (015K-CL-RAJ2). Subjects will make a follow-up visit after the Week 52 visit if they do not enroll into the extension study on the day of the Week 52 visit.

Safety data obtained from this study will be reviewed by the Independent Data and Safety Monitoring Board (DSMB), which will make recommendations on study continuation, termination, or protocol revision from the safety perspective.

#### [Study Design Rationale]

According to "Guidelines on methodology for clinical assessment of antirheumatic drugs" (PFSB/ELD Notification No. 0217001, dated 17 February 2006), the appropriate treatment period for clinical studies including a group taking a placebo alone is generally held to be 12 weeks or less, and the Guidelines state that the study should be planned so that a sufficient investigation can be performed within this time frame. Taking note that 015K-CL-RAJ1 and clinical trials of similar drugs documented treatment responses sufficient for efficacy evaluation within 12 weeks of treatment, this study was designed to assess the ACR20 response rate, a primary efficacy variable, at 12 weeks of treatment.

After Week 12, all subjects in the placebo group are to receive the active drug, and according to the "Guidelines on methodology for clinical assessment of antirheumatic drugs" (PFSB/ELD Notification No. 0217001, dated 17 February 2006), the efficacy and safety of 1-year treatment with ASP015K are to be assessed as secondary variables. As shown above, the duration of treatment was set at 52 weeks.

#### 2.2.2 Dose Rationale

#### [Dose Rationale]

Study 015K-CL-RAJ1 evaluated the efficacy, safety, and dose response of ASP015K as single-agent therapy in RA patients. This study employed 25, 50, 100, and 150 mg doses. The primary efficacy variable of this study, the ACR20 response rate at Week 12 (or early termination), showed statistically significant improvements for 50 mg and higher doses relative to placebo, and dose-dependent improvements were noted up to 150 mg. Compared with placebo, statistically significant dose-dependent decreases in the DAS28-CRP score were observed for 50 mg, 100 mg, and 150 mg groups at Week 12 (or early termination).

When the effect size between ASP015K versus placebo for the ACR20 response rate was compared with the effect sizes reported from clinical trials of a similar design (12- to 14-week, double-blind, single-agent studies) conducted in Japan for other drugs, ASP015K 100 mg or higher doses were likely to provide levels of efficacy comparable with those of other agents.

AEs reported from 1 or more groups of Study 015K-CL-RAJ1 at  $\geq$  5% incidence rates were nasopharyngitis, rheumatoid arthritis aggravated, diarrhoea, constipation, blood creatine

phosphokinase increased, stomatitis, dyspepsia, lipids increased, and blood triglycerides increased. Compared with placebo, the incidence rates of AEs were not significantly elevated for the ASP015K groups. The reported AEs were mostly Grade 1 or Grade 2 by severity (NCI-CTCAE), involving a high proportion of events known as the class effect of JAK inhibitors. The ASP015K 150 mg group had the highest incidence rate of study-related AEs. This group had a particularly high incidence rate of blood creatine phosphokinase increased, reported in 7 subjects. AEs of increased CPK levels were mostly transient; in all the cases, the subjects recovered completely, including 1 subject who prematurely discontinued the study owing to logistic issues. No collateral symptoms suggestive of rhabdomyolysis or myopathy were detected. Although careful monitoring of CPK levels will be necessary for individual subjects of this Phase III study, currently available data suggest that ASP015K-induced changes in CPK are reversible and that subject safety associated with CPK changes can be properly monitored. The mean changes in CPK levels reported for the ASP015K and placebo groups were comparable with those reported from tofacitinib clinical trials.

Ten SAEs were reported from 7 subjects; there was no characteristic pattern of occurrence, and no dose—response relationship was noted.

Thus, the results of Study 015K-CL-RAJ1 raised no safety concerns with the use of 100 and 150 mg/day doses in this Phase III study.

With regard to efficacy, ACR20 response rate and DAS28 score, the primary variables of the Phase II study, showed dose-dependent improvements up to 150 mg, and the observed effects were statistically significant in comparison with placebo for 50 mg and higher doses. Comparison of published data [Enbrel® Pharmaceutical Interview Form, Simponi® Pharmaceutical Interview Form, Xeljanz® Pharmaceutical Interview Form, Humira® Pharmaceutical Interview Form] showed that 100 mg and higher doses of ASP015K could provide efficacy comparable with that of the approved doses of similar drugs, supporting the validity of using 100 mg and higher doses in this Phase III study. From the safety perspective, the results of Study 015K-CL-RAJ1 confirmed the tolerability of ASP015K doses up to 150 mg.

Based on the abovementioned discussion, 100 and 150 mg/day doses were selected for this Phase III clinical trial.

The dose of etanercept was set at 50 mg/week, which is commonly used in Japan and recommended in the US package insert.

[Rationale for the Mode of Administration]

Nonclinical study results showed that AUC was the most important pharmacokinetic parameter for characterizing the therapeutic effect of ASP015K. While admitting that 015K-CL-PS01 focused on a clinical condition different from that of this Phase III study, this clinical trial conducted in patients with psoriasis demonstrated no significant differences between 50 mg QD and 25 mg BID doses of ASP015K.

In Study 015K-CL-RAJ1, ASP015K was administered once daily after breakfast. This method of administration was based on the idea that the desired efficacy could be achieved regardless of the differences in the mode of administration, as long as the target AUC is attained. In addition, this method of administration was favorable from the view point of subject convenience, medication adherence, and other aspects of study implementation. Study 015K-CL-RAJ1 showed excellent medication adherence and demonstrated the efficacy of ASP015K in terms of the ACR20 response rate and other outcome measures. Therefore, administration once daily after breakfast was also adopted in this clinical trial.

# 2.3 Variables

## 2.3.1 Primary Variables

• ACR20 response rate at Week 12

[Rationale]

Taking note of the "Guidelines on methodology for clinical assessment of antirheumatic drugs," and "Guidance for Industry Rheumatoid Arthritis: Developing Drug Products for Treatment", the ACR20 response rate, an indicator of RA disease activity and response to treatment, was chosen as a primary variable. The evaluation time point was set at Week 12 of treatment on the basis of the guidelines.

## 2.3.2 Secondary Variables

#### 2.3.2.1 Secondary Efficacy Variables

- ACR20 response rate
- ACR50 response rate
- ACR70 response rate
- Change from baseline in DAS28-CRP and DAS28-ESR scores
- Change from baseline in TJC (68 joints)
- Change from baseline in SJC (66 joints)
- Percentage of subjects achieving DAS28-CRP and DAS28-ESR scores for remission
- Percentage of subjects achieving low disease activity by DAS28-CRP and DAS28-ESR
- Change from baseline in CRP and ESR
- Percentage of subjects with good EULAR response
- Percentage of subjects with good or moderate EULAR response
- Percentage of subjects achieving ACR/EULAR remission

If all of the following 4 parameters are fulfilled, it is defined as remission:

- **>** TJC ≤ 1
- **>** SJC ≤ 1
- $ightharpoonup CRP \le 1 \text{ mg/dL}$
- Subject's Global Assessment of Arthritis (SGA)  $\leq 1$  cm (on a VAS of 0-100 mm)
- Percentage of subjects achieving SDAI remission (SDAI score  $\leq 3.3$ )
- Change from baseline in SDAI score
- Change from baseline in Physician's Global Assessment of Arthritis (PGA) (VAS)

- Change from baseline in SGA (VAS)
- Change from baseline in subject's assessment of pain (VAS)
- Incidence of subject withdrawal due to the lack of efficacy
- Change from baseline in HAQ-DI score
- Change from baseline in SF-36v2<sup>®</sup> score
- Change from baseline in WPAI score

## 2.3.2.2 Safety Variables

- AEs
- Vital signs (body temperature, pulse rate, and blood pressure in sitting a position)
- Body weight
- 12-lead ECG
- Central ECG
- Chest radiography
- Laboratory assessments

#### 2.3.2.3 Pharmacokinetics Variables

Plasma ASP015K concentration

#### 2.3.2.4 Pharmacodynamics Variables

- Change from baseline in MMP-3 level
- Change from baseline in VEGF level
- Change from baseline in lymphocyte subset assays (CD3, CD4, CD8, CD16, CD19, CD56, CD56/16)

## 2.3.2.5 Pharmacogenomics (Bio-Banking) [unique to Japan and Korea]

To prepare for future research to analyze the relationship between genes and the efficacy, safety, or pharmacokinetics of the study drug, blood sample will be collected and stored with the consent of the subject in Japan and Korea.

#### 2.3.3 Other Variables

Not applicable.

## 3 STUDY POPULATION

# 3.1 Selection of Study Population

The target population for this study is patients with RA who had an inadequate response to DMARDs.

## 3.2 Inclusion Criteria

Subject is eligible for the study if all of the following apply:

- 1. Subject has received a full explanation of the study drug and this study in advance, and written informed consent to participate in the study has been obtained from the subject himself/herself.
- 2. Subject is a man or woman aged  $\geq 20$  years at the time of informed consent.
- 3. Subject has RA diagnosed according to the 1987 American College of Rheumatology (ACR) criteria or the 2010 American College of Rheumatology/European League against Rheumatism (ACR/EULAR) criteria.
- 4. Subject who did not receive the following drugs, or received the drugs with stable dosage for at least 28 days prior to the baseline (start of treatment) for RA treatment: Non-steroidal anti-inflammatory drugs (NSAIDs; excluding topical formulations), oral morphine or equivalent opioid analgesics (≤ 30 mg/day), acetaminophen, or oral corticosteroids (≤ 10 mg/day in prednisolone equivalent).
- 5. At screening subject has active RA as evidenced by both of the following:
  - $\geq$  6 tender/painful joints (using 68-joint assessment)
  - $\geq$  6 swollen joints (using 66-joint assessment)
- 6. CRP > 0.50 mg/dL at screening.
- 7. Subject meets the ACR 1991 Revised Criteria for the Classification of Global Functional Status in RA Class I, II, or III at screening.
- 8. Inadequate responder to (including subjects who were intolerant of) at least one DMARD administered for at least 90 days prior to screening.
- 9. When the following DMARDs are concomitantly administered to subject, the drugs must be administered for at least 90 days prior to screening, and must be stable from at least 28 days prior to screening until the end of the administration period of study drug or reference drug.
  - Methotrexate (MTX)
  - Hydroxychloroquine
  - Salazosulfapyridine
  - Gold
  - *D*-penicillamine
  - Lobenzarit
  - Actarit
  - Bucillamine
  - Iguratimod

- 10. Subject must be willing and able to comply with the study requirements.

[Rationale for Inclusion Criteria]

- 1: Established with consideration for ethics of conducting the study.
- 2: Established to ensure ethical and safe conduct of the study.
- 3: Established to select RA patients relevant for this study. Taking note of the recent changes in RA diagnostic criteria and current practices in clinical settings, patients conforming to either the 1987 ACR or the 2010 ACR/EULAR criteria have been defined eligible for inclusion.
- 4: Established because these drugs are used to improve QOL of RA patients and may possibly impact the efficacy evaluation of ASP015K.
- 5 and 6: Established to define the range of RA disease activity pertinent to this study.
- 7: Established to identify patients appropriate for evaluation using the classification criteria for functional status.
- 8: Established to select patients who had an inadequate response to the protocol-specified DMARDs.
- 9: Established to choose patients who can maintain the same dosage and administration schedule for the specified concomitant DMARDs from before baseline and throughout the treatment period.
- 10: Established to ensure the integrity of the study evaluation.

## 3.3 Exclusion Criteria

Subject will be excluded from participation if any of the following applies:

- 1. Subject has received a biologic DMARD within the specified period:
  - Anakinra: within 28 days prior to baseline
  - Adalimumab, infliximab: within 56 days prior to baseline
  - Golimumab, certolizumab pegol: within 70 days prior to baseline
  - Abatacept, tocilizumab: within 84 days prior to baseline
  - Denosumab: within 150 days prior to baseline
  - Rituximab: within 180 days prior to baseline
- 2. Subject has received etanercept.
- 3. Inadequate responder to at least 3 biologic DMARDs as determined by investigator/sub-investigator.
- 4. Subject has received a non-biologic DMARD listed below or other drugs used in the treatment of RA within 28 days prior to baseline. Leflunomide is prohibited within 180 days prior to baseline. Alternatively, leflunomide is prohibited within 28 days prior to baseline if washout with cholestyramine for at least 17 days is completed at least 28 days

prior to baseline. However, topical drugs other than those for the treatment of RA may be used concomitantly.

- Leflunomide
- Tacrolimus
- Cyclosporine
- Cyclophosphamide
- Azathioprine
- Minocycline
- Mizoribine
- 5. Subject has received to facitinib or other JAK inhibitor (including other investigational drugs).
- 6. Subject has received intra-articular, intravenous, intramuscular, or endorectal (excluding suppositories for anal diseases) corticosteroid within 28 days prior to baseline.
- 7. Subject has participated in any study of ASP015K and has received ASP015K or placebo.
- 8. Subject has received other investigational drugs within 90 days or within 5 half-lives, whichever is longer, prior to baseline.
- 9. Subject has received plasma exchange therapy within 60 days prior to baseline.
- 10. Subject has undergone joint drainage, has received local anesthesia and nerve block, or has received articular cartilage protectant at the assessed joint within 28 days prior to baseline.
- 11. Subject has undergone surgery and has residual effects in the assessed joints at the discretion of investigator/sub-investigator, or is scheduled to undergo surgery that may affect the study evaluation of the assessed joints at the discretion of investigator/sub-investigator.
- 12. A diagnosis of inflammatory arthritis (psoriatic arthritis, ankylosing spondylitis, SLE, sarcoidosis, etc.) other than RA.
- 13. Any of the following laboratory values during the screening test period:
  - Hemoglobin < 9.0 g/dL
  - Absolute neutrophil count < 1000/μL
  - Absolute lymphocyte count < 800/μL
  - Platelet count < 75000/μL
  - ALT  $\geq 2 \times ULN$
  - $AST > 2 \times ULN$
  - Total bilirubin (TBL)  $\geq 1.5 \times ULN$
  - Estimated GFR  $\leq$  40 mL/min as measured by the MDRD method
  - $\beta$ -D-glucan > ULN [in case of Japan:  $\geq 11 \text{ pg/mL}$ ]
  - Positive HBs antigen, HBc antibody, HBs antibody or HBV-DNA quantitation (However, subject with negative HBs antigen and HBV-DNA quantitation, and positive HBc antibody and/or HBs antibody is eligible if HBV-DNA is monitored by HBV-DNA quantitation at every scheduled visit after initiation of study drug or reference drug administration.)
  - Positive HCV antibody

| 14. | ubject has a history of or concurrent active tuberculosis (TB). Eligibility criteria for TE | 3 |
|---|---|---|
| | re tabulated below: | |

| History of active<br>TB | Chest x-ray<br>(for TB) | TB infection <sup>b)</sup> | Exposure to patients with infective TB (interview) | Eligibility |
|---|---|---|---|---|
| Present | - | - | - | Not eligible |
| | Abnormal (active) | - | - | Not eligible |
| | Abnormal (old) <sup>a)</sup> | - | Eligible | Eligible if |
| | | | _ | prophylaxis is given <sup>c)</sup> |
| Absent | | Positive | Eligible | Eligible if |
| Aosent | | | _ | prophylaxis is given <sup>c)</sup> |
| | Normal | | Exposed | Eligible if |
| | | Negative | _ | prophylaxis is given <sup>c)</sup> |
| | | | Not exposed | Eligible |

- a) Old TB is evidenced if chest x-ray reveals pleural thickening, band-like shadow, and calcification  $\geq 5$  mm. Chest x-ray within 90 days prior to baseline may substitute the screening test.
- b) T-spot or Quantiferon Gold test is of first priority. When the result is equivocal or invalid, retest including other test methods may be allowed. If a retest is not performed, criteria for positive results will be followed. When T-spot or Quantiferon Gold test is not feasible, tuberculin test will be performed. Tuberculin is defined as positive with a red spot covering an area of 20 mm or more or induration. Tests conducted within 90 days prior to baseline may be used for diagnosis.
- c) Subject must receive or have received prophylaxis with isoniazid or rifampicin. Prophylaxis will be administered for 6 to 9 months, starting from at least 21 days prior to baseline.
- 15. Subject meets any of the following in terms of infections except for TB:
  - History of or concurrent severe herpes zoster (associated with Hunt syndrome or having ulcerative lesions) or disseminated herpes zoster
  - History of multiple recurrences (at least twice) of localized herpes zoster
  - Serious infection requiring hospitalization within 90 days prior to baseline
  - Subject has received intravenous antibiotics within 90 days prior to baseline. (However, prophylactic antibiotics are allowed.)
  - Subject with high risk of infection (e.g., subject with urinary catheter) at the discretion of investigator/sub-investigator
- 16. Subject has a history of or concurrent interstitial pneumonia and investigator/sub-investigator judges that it is inappropriate for the subject to participate in this study.
- 17. Subject has a history of or concurrent malignant tumor (except for successfully treated basal cell carcinoma).
- 18. Subject has received live or live attenuated virus vaccination within 56 days prior to baseline. (Inactivated vaccines including influenza and pneumococcal vaccines are allowed.)
- 19. Subject has a history of or concurrent demyelinating disorders.
- 20. Subject has any ongoing severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, metabolic, endocrine, pulmonary, cardiac, neurological, infectious, or autoimmune disease except for RA (excluding Sjogren's syndrome and chronic thyroiditis), or any ongoing illness which would make the subject unsuitable for the study as determined by the investigator/sub-investigator.

- 21. Subject has a history of clinically significant allergy. (Clinically significant allergy includes allergies such as systemic urticaria induced by specific antigens and drugs, anaphylaxis, and allergy associated with shock necessitating hospitalized treatment.)
- 22. Subject has received medications that are CYP3A substrates with narrow therapeutic range within 14 days prior to baseline. These medications include: dihydroergotamine, ergotamine, fentanyl, pimozide, quinidine, temsirolimus, and disopyramide.
- 23. Subject has concurrent cardiac failure, defined as NYHA classification Class III or higher, or a history of it.
- 24. Subject has concurrent prolonged QT syndrome or a history of it. Subject has prolonged QT interval (defined as QTc ≥ 500 msec. Subject has QTc ≥ 500 msec at retest will be excluded) at screening.
- 25. Subject has a history of positive HIV infection.
- 26. Subject is a woman who is pregnant or might be pregnant, is nursing, wishes to conceive for a period running from the time informed consent is given within 60 days after end of treatment (including reference drug), or for whom the possibility of pregnancy cannot be ruled out as a result of the serum pregnancy test given at the time of screening.
- 27. Subject is a man who cannot practice at least 2 types of contraception from the time of informed consent to 90 days after end of treatment (including reference drug), or subject is a woman with childbearing potential who cannot practice at least 2 types of contraception from the time of informed consent to 60 days after end of treatment (including reference drug).
- 28. Male subject who do not agree not to donate sperm starting at informed consent and through the treatment period and for at least 90 days after final study drug (or reference drug) administration. Female subject who do not agree not to donate ova starting at informed consent through the treatment period and for 60 days after final study drug (or reference drug) administration.
- 29. The subject has been judged unsuitable to participate in the study for other reasons by the investigator/sub-investigator.
- 30. The subject has a history or complication of lymphatic diseases such as lymphoproliferative disorder, lymphoma, and leukemia.
- 31. Subject has congenital short QT syndrome or a history of it. Subject has shortened QT interval (defined as QTc < 330 msec. Subject has QTc < 330 msec at retest will be excluded) at screening.

#### [Rationale for exclusion criteria]

- 1, 4, 5, 6, 7, 8: Established to eliminate confounding factors affecting evaluation.
- 2: Established in consideration of the efficacy of etanercept.
- 3, 9, 10, 11, 12: Established to eliminate confounding factors affecting efficacy evaluation.
- 13, 14, 15, 16, 17, 18, 20, 21, 22, 23, 24, 25, 26, 27, 28, 30, 31: Established out of safety concerns.

- 19: Established in consideration of the safety of subjects, because etanercept is contraindicated in patients who previously had or currently have demyelinating disorders.
- 29: Established in anticipation for a case where the investigator/sub-investigator judges a patient to be inappropriate for participation in the study.
- 31: The QTc criterion is quoted from Expert Consensus [Silvia G. Priori, 2014] of HRS/EHRA/APHRS.

# 3.4 Discontinuation Criteria for Individual Subjects

A discontinuation is a subject who enrolled in the study and for whom study treatment is permanently prematurely discontinued for any reason.

The subject is free to withdraw from the study treatment and/or study for any reason and at any time without giving reason for doing so and without penalty or prejudice. The investigator is also free to terminate a subject's involvement in the study at any time if the subject's clinical condition warrants it.

The Appendix 4 entitled "Liver Safety Monitoring and Assessment" describes liver function tests raised that provide grounds for discontinuation. Refer to Appendix 4 concerning the measures to take for increases in liver function test parameters.

The investigator/sub-investigator should discontinue the study if any of the following occurs:

- 1. The subject withdraws consent.
- 2. The investigator/sub-investigator judges that the study drug or reference drug is not sufficiently effective and the treatment method needs to be changed.
- 3. Symptomatic CPK elevation (> 1.5 × ULN accompanied with severe and unusual episodes of myalgia, muscular weakness, or muscle twitching).
- 4. Any case of myopathy involving severe and unusual episodes of myalgia, muscular weakness, or muscle twitching that persists for no less than, or aggravates rapidly within, 2 weeks, regardless of the CPK level.
- 5. A previously HBV-infected patient with positive HBc antibody, positive HBs antibody, or both has been shown positive for HBV-DNA during the study.

  Attention should be paid that abrupt discontinuation of immunotherapy may cause fulminant or severe liver failure. Therefore, if the subject manifests HBV reactivation, the investigator/sub-investigator will administer nucleoside analogs without delay [unique to Japan: according to the "Proposal for Management of Rheumatic Disease Patients with Hepatitis B Virus Infection Receiving Immunosuppressive Therapy" (Japan College of Rheumatology)]. The investigator/sub-investigator will carefully decide whether to continue or discontinue the study drug, reference drug, and concomitant DMARDs in consultation with the hepatology specialist.
- 6. Malignant tumor

- 7. The subject develops a serious infection or other AEs, and continued administration of the study drug is not deemed appropriate in the subject's best interest by the investigator/sub-investigator.
- 8. The subject has been treated with a prohibited concomitant drug or therapy (including another investigational product) that may impact efficacy evaluation. The subject has been, or needs to be, treated with a rescue medication for a period extending beyond its allowable time. Otherwise, the subject has been, or needs to be, treated with a live or live attenuated vaccine.
- 9. The subject has been judged by the investigator/sub-investigator to be non-compliant to the medication requirements for treatment with the study drug, concomitant DMARDs, or reference drug injection.
- 10. The subject is deemed incapable of continuing the follow-up based on the opinion of the investigator/sub-investigator (subject can no longer come to the study center; subject can no longer be contacted, etc.).
- 11. It comes to light after the administration of the first dose of study drug or reference drug that inclusion criteria were not met at the time of case enrollment or that criteria for exclusion were met. It comes to light that there was some other major deviation from the protocol.
- 12. The subject needs the study drug or reference drug to be interrupted beyond its allowable time limit.
- 13. Investigator/sub-investigator decides it is in the subject's best interest.
- 14. The sponsor has requested that the study be discontinued because of a safety concern in a particular subject, or the sponsor has decided to discontinue the study altogether.
- 15. The Subject shows QTc interval < 300 msec at central ECG, or the subject shows QTc interval < 300 msec at the site's ECG and also shows QTc interval < 300 msec at retest.

Subjects who discontinue early from the study should be given the necessary tests and assessments specified for early termination within 2 days of withdrawal. They should also undergo follow-up tests and assessments. Subjects with early termination will be treated as discontinuations, and the investigator/sub-investigator must make clear the reason for discontinuation and the day of early termination (the date on which the investigator/sub-investigator has decided to discontinue the subject) as well as retain all clinical study data on the discontinuations and submit them to the sponsor in eCRF, etc.

# 3.4.1 Suspension, Interruption, and Resumption of the Study Drug or Reference Drug

During treatment with the study drug or reference drug, if the subject meets any of the criteria provided in Section 3.4.1.1 Criteria for Suspension or Interruption of the Study Drug or Reference Drug, the investigator/sub-investigator will immediately suspend or interrupt the study drug or reference drug. The investigator/sub-investigator can resume treatment with the study drug or reference drug only if re-examinations and other assessments performed after the suspension or interruption confirm that none of the conditions listed below are

3 March 2017 Astellas 

applicable to the subject and the investigator/sub-investigator considers it desirable for the interest of the subject on the basis of risk-benefit analysis.

The maximum allowable time for "suspension" is 7 days for the study drug and a week (1 dose per week) for the reference drug. If the treatment is halted beyond the suspension period, i.e., longer than 7 days for the study drug or skipping more than 1 dose for the reference drug, the period of no treatment is categorized as an "interruption."

Upper limits have been set to the number of interruptions 1 subject can have and to the duration of 1 interruption. One interruption period may last for 28 days for the study drug and 4 weeks (i.e., 4 consecutive doses) for the reference drug. One subject is allowed to have a maximum of 2 interruptions, which must be separated by 16 or more weeks.

The investigator will consult the sponsor regarding the handling of a subject who repeatedly requires treatment suspension.

The subject must be withdrawn from the study, if he or she requires either a third interruption or a second interruption within less than 16 weeks from the first one.

### 3.4.1.1 Criteria for Suspension or Interruption of the Study Drug or Reference Drug

The investigator/sub-investigator will immediately suspend or interrupt the study drug or reference drug if any of the following becomes applicable during treatment with the study drug or reference drug:

- 1. Clinical laboratory tests yielded any of the following results:
  - Hemoglobin < 8.0 g/dL
  - Absolute neutrophil count < 500/μL
  - Absolute lymphocyte count < 500/μL
  - Platelet count < 50000/μL
  - Creatinine (serum) levels measured at 2 consecutive hospital visits: above 150% of the baseline level
  - CPK > 10 × ULN
- 2.  $\beta$ -D-glucan > ULN [in case of Japan:  $\geq 11 \text{ pg/mL}$ ]
- 3. The subject requires a medication whose concomitant administration is prohibited in the protocol because of possible drug-drug interaction.
- 4. The subject is suspected to be pregnant.
- 5. The investigator/sub-investigator judged it appropriate in the interest of the subject to suspend or interrupt the study drug or reference drug.
- 6. The sponsor made a request to suspend or interrupt the study drug or reference drug out of safety concerns for the subject.

## 4 STUDY DRUGS OR REFERENCE DRUGS

# 4.1 Description of Study Drugs or Reference Drugs

The test drugs for this study are ASP015K tablets of 100 mg and 150 mg. The comparative drugs are ASP015K tablet placebos of 100 mg and 150 mg. The reference drug is an etanercept (recombinant) 50 mg syringe (1.0 mL).

## **4.1.1 Test Drug(s)**

| Code name | ASP015K |
|---|---|
| Generic name | Peficitinib hydrobromide |
| Chemical name | 4-{[(1 <i>R</i> ,2 <i>S</i> ,3 <i>S</i> ,5 <i>S</i> ,7 <i>S</i> )-5-hydroxy-2-adamantyl]amino}-1 <i>H</i> -pyrrolo[2,3- <i>b</i> ] pyridine-5-carboxamide monohydrobromide |
| Molecular formula<br>(molecular weight) | $C_{18}H_{22}N_4O_2 \cdot HBr (407.30)$ |
| Content and dosage form | ASP015K tablet 100 mg: An elliptical, pale-red film coated tablet containing the ASP015K drug substance at 100 mg (as free form) ASP015K tablet 150 mg: An elliptical, yellow, film-coated tablet containing the ASP015K drug substance at 150 mg (as free form) |
| Manufacturer | Astellas Pharma Inc. (API) |
| Lot No. | Noted in SOP for handling of study drugs |
| Storage method | Store at room temperature |
| Expiration date | Noted in SOP for handling of study drugs |

# 4.1.2 Comparative Drug(s)

| | 807 |
|---|---|
| Code name | ASP015K |
| | ASP015K tablet 100 mg placebo: An elliptical, pale-red film coated |
| Content and dosage form | tablet indistinguishable from the ASP015K tablet 100 mg |
| | ASP015K tablet 150 mg placebo: An elliptical, yellow, film-coated |
| | tablet indistinguishable from the ASP015K tablet 150 mg |
| Manufacturer | Astellas Pharma Inc. (API) |
| Lot No. | Noted in SOP for handling of study drugs |
| Storage method | Store at room temperature |
| Expiration date | Noted in SOP for handling of study drugs |

# 4.1.3 Reference Drug(s)

| Generic name | Etanercept (recombinant) |
|---|---|
| Generic name | 1 \ |
| Chemical name | 1-235-Tumor necrosis factor receptor(human)fusion protein with |
| | 236-467-immunoglobulin G1(humany1-chain Fc fragment),dimer |
| Molecular formula | Molecular weight: approximately 150,000 |
| (molecular weight) | Total number of amino acids: 934 |
| Content and dosage form | Etanercept 50 mg syringe (1.0 mL) |
| Manufacturer | |
| Lot No. | Noted in SOP for handling of study drugs |
| Storage method | Do not freeze and store at 2°C to 8°C protected from light. |
| Expiration date | Noted in SOP for handling of study drugs |

# 4.2 Packaging and Labeling

All medications used in this study will be manufactured, packaged, and labeled under the responsibility of the Quality Assurance Manager in accordance with sponsor's Standard Operating Procedures (SOP), GMP guidelines, GCP and applicable local laws/regulations. (Refer to the study drug handling manual for details)

(Packaging form)

The study drugs will be packaged in a small box containing 28 day's worth of medication and 7 day's worth of spare medication. One PTP sheet (aluminium/aluminium) holds a total of 14 tablets: 7 tablets of ASP015K at 100 mg or placebo for ASP015K at 100 mg and 7 tablets of ASP015K at 150 mg or placebo for ASP015K at 150 mg. Five PTP sheets (including 1 spare sheet) will be packaged in the small box.

Reference drugs will be supplied in 2 commercially available cartons containing 2 syringes each.

In case of Japan (Package design of study drug and reference drug for Korea and Taiwan is described in the study drug handling manual):

(Study drug)



## (Reference drug)



Lot No. is noted in SOP for handling of study drugs.

# 4.3 Study/Reference Drug Handling

Japan:

The head of the study center or the study drug storage manager should take accountability of the study drugs or reference drugs as following issues.

- The study drug storage manager should store and take accountability of the study drugs or reference drugs in conforming to the procedures for handling the study drugs written by the sponsor.
- The study drug storage manager should prepare and retain records of the study drug's receipt, the inventory at the study center, the use by each subject, and the return to the sponsor or alternative disposal of unused study drugs or reference drugs. These records should include dates, quantities, batch/serial numbers, expiration dates (if applicable), and the subject identification codes.
- The study drug storage manager should prepare and retain records that document adequately that the subjects were provided the doses specified by the protocol, and reconcile all the study drugs or reference drugs supplied from the sponsor.

#### Korea and Taiwan:

The procedures will be specified separately in the study drug handling manual in accordance with the local requirements.

# 4.4 Blinding

## 4.4.1 Blinding Method

Treatment allocation to the ASP015K 100 mg, ASP015K 150 mg, or placebo groups is double-blinded. The ASP015K tablet 100 mg, ASP015K tablet 100 mg placebo, or ASP015K

tablet 150 mg, ASP015K tablet 150 mg placebo are indistinguishable from each other in appearance, and the packaging for each treatment group (100 mg, 150 mg, and placebo) is also indistinguishable from that for other groups in appearance. The treatment code will only be known to the person responsible for assigning study drugs, person appointed at the institution performing measurements of plasma drug concentrations, persons in the Safety Control Division when necessary for Suspected Unexpected Serious Adverse Reaction (SUSAR) handling, and independent Data and Safety Monitoring Board (DSMB).

No blinding will be performed for the reference group.

## 4.4.2 Confirmation of the Indistinguishability of the Study Drugs

The appearance and the form of both the drug and packaging of the ASP015K tablet 100 mg and ASP015K tablet 150 mg are identical to those of their matching placebo. [unique to Japan: The person responsible for assigning study drugs will confirm the indistinguishability of the study drugs and their packaging in appearance before the assignment of the study drugs and during the period from collection of the study drugs to the breaking of the treatment code].

# 4.4.3 Retention of the Assignment Schedule and Procedures for Treatment Code Breaking

The person responsible for assigning study drugs will create a randomization list (original document) plus 3 copies (reproductions) for Japan and Korea/Taiwan separately in advance of the assignment of the study drug and seal each separately. The person responsible for assigning study drugs will retain the original randomization list. One copy of the randomization list (reproduction) will be retained by the sponsor in a sealed state even after the breaking of the treatment code, one copy will be prepared for use by DSMB, and the third copy will be provided to the institution performing measurements of plasma drug concentrations by the person responsible for assigning study drugs to be used as a sample measurement instruction sheet bearing treatment code information.

The person responsible for assigning study drugs will also create a treatment code for emergency and provide it to the person responsible for managing the treatment code for emergency. The person responsible for managing the treatment code for emergency will manage individual treatment code for emergency with code breaking permission in the web-based system. The web treatment code system can only be accessed by the person responsible for managing treatment code for emergency, the sponsor's responsible personnel (or sponsor), and the person in charge of the Safety Control Division when necessary for SUSAR handling. The "SOPs for the Phase III Study of ASP015K DSMB" should be followed for treatment code retention, breaking, and code information conservation at the time of safety data review and safety evaluation.

## 4.4.4 Breaking the Treatment Code for Emergency

In the event of a medical emergency requiring knowledge of the treatment assigned to the subject, the investigator/sub-investigator can ask the sponsor to break the treatment code for emergency for the subject in question. The sponsor will make the decision as to whether or

not to break the treatment code for emergency. The "SOPs for breaking the treatment code for emergency in Phase III study of ASP015K (015K-CL-RAJ3)" should be followed when the treatment code is broken. The investigator/sub-investigator, sponsor, and the person responsible for managing the treatment code for emergency should maintain contact so that the treatment code can be broken immediately in an emergency. When a sub-investigator requests that the treatment code be broken in an emergency, the consent of the investigator should in principle be obtained in advance. However, in cases where it is difficult to obtain the understanding of the investigator in advance, the sub-investigator should immediately report the request to break the treatment code for an emergency to investigator after the fact. After the treatment code has been broken by the investigator or other responsible personnel, the study center must report the breaking of the treatment code and the reason for doing so to the contacts listed in the "Section II CONTACT DETAILS OF KEY SPONSOR'S PERSONNEL."

## 4.4.5 Breaking the Treatment Code by the Sponsor

The sponsor may break the treatment code for subjects who experience SUSAR if regulatory reporting is considered necessary. An individual emergency code will be provided to the limited staff who are empowered to break the code for all SUSAR cases for reporting purposes.

# 4.5 Assignment and Allocation

The person responsible for assigning study drugs will randomly assign the study drugs and retain the treatment code under secrecy until the breaking of the treatment code.

The Case Registration Center will assign subjects who have been found to be eligible for enrollment in accordance with the case registration procedures to 1 of the following groups: ASP015K 100 mg, ASP015K 150 mg, placebo, or reference groups at baseline in 1:1:1:2 ratio. At Week 12, subjects in the placebo group will be switched to receiving either ASP015K at a dose of 100 mg or ASP015K at a dose of 150 mg. The dose of ASP015K (100 mg or 150 mg) to be administered to the placebo group from Week 12 will be determined in advance randomly at baseline, and study drugs must be switched under double-blind conditions.

To minimize potential bias in this study, dynamic allocation procedures in each study region (Japan, Korea, and Taiwan) will be used by biased-coin minimization with the following 1 to 3 as factors:

- 1. Study center;
- 2. Prior biologic DMARD-IR at baseline; and
- 3. Concomitant DMARD use at the initiation of treatment with the study drug or reference drug.

All drug numbers are assigned randomly by the Case Registration Center under blind conditions.

## 5 TREATMENTS AND EVALUATION

# 5.1 Dosing and Administration of Study Drugs or Reference Drugs and Other Medications

## 5.1.1 Dose/Dose Regimen and Administration Period

## (1) Dose and administration period

The following 4 treatment groups will be set up: ASP015K 100 mg group, ASP015K 150 mg group, placebo group, and reference group.

The dose for each treatment group is shown in the table below. Two tablets of the drug described in the table below will be administered QD. The administration period will be 52 weeks. At Week 12, subjects in the placebo group will be switched to receiving either ASP015K at a dose of 100 mg or ASP015K at a dose of 150 mg under blind conditions. The dose of ASP015K to be administered to the placebo group from Week 12 will be determined in advance at baseline and will be continued until Week 52.

For the reference group, open-label etanercept will be administered for 52 weeks.

Table Treatment Periods and Doses by Treatment Period (Administered Drug) in Study 015K-CL-RAJ3

| | Baseline–Week 12 <sup>1)</sup> | Week 12–Week 52 |
|---|---|---|
| Placebo group | ASP015K placebo (ASP015K tablet 100 mg placebo and ASP015K tablet 150 mg placebo) | 100 mg/day as ASP015K (ASP015K tablet 100 mg and ASP015K tablet 150 mg placebo) 150 mg/day as ASP015K (ASP015K tablet 100 mg placebo and ASP015K tablet 150 mg) |
| ASP015K 100 mg group | 100 mg/day as ASP015K<br>(ASP015K tablet 100 mg and ASP015K tablet 150 mg placebo) | |
| ASP015K 150 mg group | 150 mg/day as ASP015K<br>(ASP015K tablet 100 mg placebo and ASP015K tablet 150 mg) | |
| Reference group | Etanercept 50 mg/week (the last dose will be given at Week 51.) | |

<sup>1)</sup> At Week 12, subjects in the placebo group will be assigned to receiving either ASP015K 100 mg or ASP015K 150 mg. Subjects will continue receiving the assigned dose thereafter.

#### (2) Mode of administration

[ASP015K 100 mg, ASP015K 150 mg, and placebo groups]

The assigned study drug will be orally administered to subjects under double-blind conditions QD after breakfast. The baseline dose should be given at each study center on the day of the baseline visit after all assessments and tests are completed.

Doses on the day of scheduled visits during treatment with the study drug or reference drug should be given on the day of the visit after all assessments and tests are completed, except for blood sampling for the assessment of post-dose concentrations.

## [Reference group]

The reference drug will be subcutaneously administered to subjects once weekly (the last dose will be given at Week 51). The baseline dose should be given at each study center on the day of the baseline visit after all assessments and tests are completed. After the baseline visit, the reference drug will be given taking the same day of the week at baseline as the reference date. The acceptable time range for administration of the reference drug will be within  $\pm$  6 days of the reference date, and if the reference drug is given beyond the acceptable time range, it will be regarded as unadministered. The reference drug should also be administered at a minimum of 3-day intervals.

Doses on the day of scheduled visits during treatment with the study drug or reference drug should be given on the day of the visit after all assessments and tests are completed.

The reference drug may be given at any time on administration days (in-hospital administration and self-administration), except those of scheduled visits.

Etanercept can be self-administered only by the subject who has been provided with adequate education and training by the study center and who is judged to be capable of injecting etanercept by himself/herself in the opinion of the investigator/sub-investigator.

The investigator/sub-investigator should instruct subjects who will self-administer etanercept to pay close attention to their condition before and after administration on the day of self-administration to assess the condition in a prompt manner. When the investigator/sub-investigator finds problems with the subject's adherence to self-injection treatment regimens and the mode of administration, the investigator/sub-investigator will administer etanercept at the hospital until the subject can learn to inject it by himself/herself.

The subject's condition before and after in-hospital administration should also be closely monitored.

## 5.1.2 Previous and Concomitant Medication (Drugs and Therapies)

The survey period and survey method for previous and concomitant medication (drugs and therapies) will be as follows.

#### (1) Previous medications

Pharmaceutical name, daily dose, route of administration, period of administration, and reason for administration of drugs used within the past 90 days, counting back from before the initiation of treatment with the study drug or reference drug on the day of the baseline visit

> DMARD, prohibited concomitant medications, restricted concomitant medications (taken within 28 days prior to baseline), rescue medications (taken within 28 days prior to baseline)

Medications for the treatment of RA (biologic DMARD, non-biologic DMARD) should be entered separately in the eCRF as the treatment history of the target disease described in Section 5.2.3 Diagnosis of the Target Disease, Severity, and Duration of Disease.

## (2) Previous therapies

None

### (3) Concomitant medications

The survey period will be from the initiation of treatment with the study drug or reference drug on the day of the baseline visit.

Information on pharmaceutical name, daily dose, route of administration, period of administration, and reason for administration of DMARD, prohibited concomitant medication, restricted concomitant medication, and rescue medication will be collected.

In addition, pharmaceutical name, route of administration, period of administration, and reason for administration of medications other than DMARD, prohibited concomitant medication, restricted concomitant medication, rescue medication, and the following will be obtained.

Solution for dissolving or diluting (water for injection, saline), disinfectant, rinsing fluid, surface anesthetic for tests and procedures (such as Xylocaine jelly), contrast media for tests (such as barium, noniodinated contrast media), anticoagulants for use by the IV placement route, foaming agents and laxatives for use during tests, and topical drugs for local effect and for purposes other than RA.

\*However, if such medications are used for the purpose of treating an adverse event, they should be entered in the eCRF.

Medications for the treatment of RA (biologic DMARD, non-biologic DMARD) should be entered separately in the eCRF as the treatment history of the target disease described in Section 5.2.3 Diagnosis of the Target Disease, Severity, and Duration of Disease.

#### (4) Concomitant therapies

The survey period will be from the initiation of study treatment on the day of the baseline visit.

The name, purpose, and duration of therapies performed for RA, and adverse events will be obtained. Procedures (such as gauze replacement) and therapies (such as rehabilitation) performed for surgery will not be considered as concomitant therapies.

#### **5.1.2.1** Previous Medication (Drugs and Therapies)

A period during which a drug cannot be used or a therapy is prohibited will be established as follows before the initiation of treatment with the study drug or reference drug for any previous medication (drugs and therapies) that could affect the evaluation of ASP015K:

- 1) Prohibited concomitant medications and therapies:
- Biologic DMARD

The following biologic DMARDs will be prohibited during the period shown below:

Etanercept: after informed consent is obtained

- Anakinra: within 28 days prior to baseline
- Adalimumab, infliximab: within 56 days prior to baseline
- Golimumab, certolizumab pegol: within 70 days prior to baseline
- Abatacept, tocilizumab: within 84 days prior to baseline
- Denosumab: within 150 days prior to baseline
- Rituximab: within 180 days prior to baseline

## Non-biologic DMARD

Non-biologic DMARDs other than those listed below will be prohibited within 28 days prior to baseline. Subjects who continue receiving the drugs described below during treatment with the study drug or reference drug should follow regulations for restricted concomitant medications. The use of leflunomide will be prohibited within 180 days prior to baseline. However, if washout with cholestyramine for at least 17 days is completed before 28 days prior to baseline, the use of leflunomide is prohibited within 28 days prior to baseline. However, topical drugs other than those for the treatment of RA may be used concomitantly.

- ➤ Methotrexate (MTX)
- > Hydroxychloroquine
- > Salazosulfapyridine
- ➢ Gold
- > D-penicillamine
- Lobenzarit
- Actarit
- Bucillamine
- Iguratimod

#### Other drugs used in the treatment of RA

Cyclosporine, cyclophosphamide, azathioprine, minocycline, and other drugs indicated for the treatment of RA will be prohibited within 28 days prior to baseline.

#### Corticosteroids

Oral corticosteroids at doses exceeding 10 mg per day in the prednisolone equivalent will be prohibited within 28 days prior to baseline.

The intra-articular, intravenous, intramuscular, and endorectal corticosteroid administration will also be prohibited within 28 days prior to baseline. However, suppositories for anal diseases may be used concomitantly.

## Oral morphine

Oral morphine at doses exceeding 30 mg per day (or equivalent doses of other opioid analgesics) will be prohibited within 28 days prior to baseline.

#### Other study drugs

Other study drugs will be prohibited within 90 days or 5 half-lives, whichever is longer, prior to baseline.

#### CYP3A substrates

The following CYP3A substrates with a narrow therapeutic range will be prohibited within 14 days prior to baseline: dihydroergotamine, ergotamine, fentanyl, pimozide, quinidine, temsirolimus, disopyramide, etc.

#### Vaccines

Live or live attenuated virus vaccinations will be prohibited within 56 days prior to baseline. Inactivated vaccines may be administered (influenza, pneumococcal vaccines, etc.).

Plasma exchange therapy

Plasma exchange therapy will be prohibited within 60 days prior to baseline.

Surgical treatment methods

After obtaining informed consent, surgery involving the target joint will be prohibited.

• Effusion drainage, local anesthesia, and nerve block of the target joint

Effusion drainage, local anesthesia, and nerve block of the target joint will be prohibited within 28 days prior to baseline.

Articular cartilage protective agents

The use of articular cartilage protective agents in the target joint will be prohibited within 28 days prior to baseline.

2) Restricted concomitant medications

<Concomitant DMARDs>

- If any (some) of the following DMARDs are administered concomitantly with the study drug or reference drug, they should be given for at least 90 days prior to screening, and the same dosage and administration schedule must be maintained from at least 28 days prior to screening to the end of treatment with the study drug or reference drug.
- Changes to the dosage, administration schedule, or route of administration will not be allowed within 28 days prior to baseline and during treatment with the study drug or reference drug.
- If a DMARD is temporarily interrupted or its dose is reduced within 28 days prior to the baseline visit in a subject eligible at screening for the study based on inclusion and exclusion criteria, the screening period will be extended to allow for the same dosage and administration schedule to be observed for 28 days prior to the baseline visit.
- If MTX is administered with study drug or reference drug concurrently, the concomitant use of folic acid should be considered whenever possible. The dose of folic acid during the study period will, in principle, be within 10 mg per week, but it may be adjusted. If MTX is administered and ALT/AST becomes ≥ 3 × ULN, MTX must be interrupted, or the dose must be reduced, and daily administration of folic acid should be considered.

- ➤ Methotrexate (MTX)
- > Hydroxychloroquine
- > Salazosulfapyridine
- ➢ Gold
- ➤ *D*-penicillamine
- Lobenzarit
- > Actarit
- Bucillamine
- > Iguratimod

#### <Other restricted concomitant medications>

- For subjects who continue receiving the drugs described below during treatment with the study drug or reference drug, changes to the dosage, administration schedule, or route of administration will not be allowed within 28 days prior to baseline.
- The drugs listed below will be prohibited within 28 days prior to baseline if they are to be discontinued before the initiation of treatment with the study drug or reference drug [except in cases where NSAIDs and non-NSAID analgesics (e.g., acetaminophen, opioid analgesics, all-in-one flu and cold medications) are used as rescue medication].
- In the case of a medically unfavourable event during the screening period, administration may be temporarily interrupted, or the dose may be temporarily reduced. The period of interruption is up to 28 days. When resuming administration, the dose prior to interruption/reduction is the upper limit.
  - NSAIDs (excluding topical drugs)
  - ➤ Oral morphine (Not more than 30 mg per day, or equivalent doses of other opioid analgesics)
  - > Acetaminophen
  - ➤ Oral corticosteroids
    (However, at 10 mg per day or less in the prednisolone equivalent and from the visit at Week 12, the dose may be reduced or increased within the range not exceeding the baseline dose.)

#### 3) Rescue medications

The drugs listed below may be used within 28 days prior to baseline only if they are necessary for treating a medically unfavourable event or acute worsening of the primary disease. However, these medications may not be taken within 24 hours before joint assessment at baseline.

- NSAIDs: For 3 days or less
- Analgesics other than NSAIDs (acetaminophen, opioid analgesics, all-in-one cold and flu medications, etc.): For 7 consecutive days or less.
#### 5.1.2.2 Concomitant Medication (Drugs and Therapies)

- 1) Prohibited concomitant medications and therapies:
- Biologic DMARDs

The following biologic DMARDs will be prohibited during treatment with the study drug or reference drug. Etanercept given as the reference drug will be excluded.

Adalimumab, anakinra, infliximab, golimumab, certolizumab pegol, abatacept, tocilizumab, rituximab, etanercept, and denosumab

#### Non-biologic DMARDs

Non-biologic DMARDs other than those listed below will be prohibited during treatment with the study drug or reference drug.

Subjects who continue receiving the drugs described below during treatment with the study drug or reference drug should follow regulations for restricted concomitant medications. Administration of the drugs listed below will be prohibited when subjects do not observe these regulations. However, topial drugs other than those for the treatment of RA may be used concomitantly.

- ➤ Methotrexate (MTX)
- > Hydroxychloroquine
- Salazosulfapyridine
- ➤ Gold
- ➤ *D*-penicillamine
- Lobenzarit
- > Actarit
- Bucillamine
- Iguratimod

#### Other drugs used in the treatment of RA

Cyclosporine, cyclophosphamide, azathioprine, minocycline, and other drugs indicated for the treatment of RA will be prohibited during treatment with the study drug or reference drug.

#### Corticosteroids

Oral corticosteroids at doses exceeding 10 mg per day in the prednisolone equivalent will be prohibited during treatment with the study drug or reference drug.

The intra-articular, intravenous, intramuscular, and endorectal corticosteroid administration will also be prohibited during treatment with the study drug or reference drug. However, suppositories for anal disease may be used concomitantly.

#### Oral morphine

Oral morphine at doses exceeding 30 mg per day (or equivalent doses of other opioid analgesics) will be prohibited during treatment with the study drug or reference drug.

#### Other study drugs

Other study drugs will be prohibited during treatment with the study drug or reference drug and during the follow-up period.

#### CYP3A substrates

The following CYP3A substrates with a narrow therapeutic range will be prohibited during treatment with the study drug or reference drug and during the follow-up period: dihydroergotamine, ergotamine, fentanyl, pimozide, quinidine, temsirolimus, disopyramide, etc.

#### Vaccines

Live or live attenuated virus vaccinations will be prohibited during treatment with the study drug or reference drug and during the follow-up period. Inactivated vaccines may be administered (influenza, pneumococcal vaccines, etc.)

#### Plasma exchange therapy

Plasma exchange therapy will be prohibited during treatment with the study drug or reference drug.

#### Surgical treatment methods

Surgery involving the target joint will be prohibited during treatment with the study drug or reference drug.

• Effusion drainage, local anesthesia, and nerve block of the target joint

Effusion drainage, local anesthesia, and nerve block of the target joint will be prohibited during treatment with the study drug or reference drug.

• Articular cartilage protective agents

The use of articular cartilage protective agents in the target joint will be prohibited during treatment with the study drug or reference drug.

#### 2) Restricted concomitant medications

#### <Concomitant DMARDs>

- If any (some) of the following DMARDs are administered concomitantly with the study drug or reference drug, they should be given for at least 90 days prior to screening, and the same dosage and administration schedule must be maintained from at least 28 days prior to screening to the end of treatment with the study drug or reference drug.
- Changes to the dosage, administration schedule, or route of administration will not be allowed during treatment with the study drug or reference drug.

- In the case of AEs, administration may be temporarily interrupted, or the dose may be temporarily reduced. When resuming administration, the baseline dose is the upper limit. The period of interruption is up to 28 days and interruption is allowed only once.
- If MTX is administered with study drug or reference drug concurrently, the concomitant use of folic acid should be considered whenever possible. The dose of folic acid during the study period will, in principle, be within 10 mg per week, but it may be adjusted. If MTX is administered and ALT/AST becomes ≥ 3 × ULN, MTX must be interrupted, or the dose must be reduced, and daily administration of folic acid should be considered.
  - ➤ Methotrexate (MTX)
  - > Hydroxychloroquine
  - Salazosulfapyridine
  - **➢** Gold
  - ➤ D-penicillamine
  - Lobenzarit
  - Actarit
  - Bucillamine
  - > Iguratimod

#### <Other restricted concomitant medications>

For subjects who continue receiving the drugs described below during treatment with the study drug or reference drug, changes to the dosage, administration schedule, or route of administration will not be allowed from 28 days prior to baseline to the end of treatment with the study drug or reference drug, except when the following conditions are satisfied:

- The drugs listed below will be prohibited from 28 days prior to baseline to the end of treatment with the study drug if they are discontinued before the initiation of treatment with the study drug or reference drug [except in cases where NSAIDs and non-NSAID analgesics (e.g., acetaminophen, opioid analgesics, all-in-one flu and cold medications) are used as rescue medication].
- In the case of AEs, administration may be temporarily interrupted, or the dose may be temporarily reduced. The period of interruption is up to 28 days. When resuming administration, the baseline dose is the upper limit.
- From the visit at Week 12, the drugs below may be discontinued, new drugs may be used, and the dosage, administration schedule, or route of administration of the concomitant drugs may be changed. However, with the exception of oral corticosteroids, after changing the conditions, administration must be continued under the same conditions for 12 weeks or longer.
  - NSAIDs (excluding topical drugs)
  - Oral morphine
     (Not more than 30 mg per day, or equivalent doses of other opioid analgesics)
  - Acetaminophen

# Oral corticosteroids (However, at 10 mg per day or less in the prednisolone equivalent and from the visit at Week 12, the dose may be reduced or increased within the range not exceeding the baseline dose.)

#### 3) Rescue medications

The drugs listed below may be used only if they are necessary for treating AEs, comorbid conditions, or acute aggravation of the primary disease during the administration period of the study drug or reference drug. However, these medications may not be taken within 24 hours before joint assessment at each visit.

- NSAIDs: For 3 days or less
- Analgesics other than NSAIDs (acetaminophen, opioid analgesics, all-in-one flu and cold medications, etc.): For 7 consecutive days or less

#### **5.1.3** Treatment Compliance

The investigator, sub-investigator, or study drug storage manager will provide the subjects with an explanation of how to take the study drug or inject the reference drug, paying particular attention to the following points when they hand the study drug or reference drug to each subject.

- Do not take multiple doses all at once if doses of the study drug have been missed.
- Bring any remaining study drug with you to the next scheduled examination.
- Immediately contact the investigator, sub-investigator, or collaborator if there is a shortage of the study drug before the next visit due to the loss of study drugs, etc.
- When you have been assigned to the reference group and are given an injection on an outpatient basis, visit the study site every week for etanercept injection. Record the date and site of injection in source documents.
- When you have been assigned to the reference group and inject etanercept by yourself, record the date and site of injection in the medication diary. Closely monitor your health, particularly on the date of injection, and immediately contact the investigator, sub-investigator, or collaborator if something is wrong with your health. Bring any unused syringes with you to the next scheduled visit. In principle, bring used syringes and needles with you to the next scheduled visit.
- Be sure to avoid an overdose if you have been assigned to the reference group and inject etanercept by yourself.
- If you forget to inject etanercept by yourself, bring unused syringes with you to the next scheduled visit.

The investigator/sub-investigator will confirm each subject's compliance with study and reference treatment and the injection of the reference drug during treatment with the study drug or reference drug on the basis of information given by the subject and the number of tablets (study drugs) or syringes (reference drugs) collected from the subject, and the investigator/sub-investigator will record the number of tablets or syringes prescribed and the number of unused tablets or syringes in the eCRF. If there is judged to be a problem with the

rate of compliance or injection, guidance on patient compliance should be provided to the subject again to improve the rate of compliance or the method of injection after investigating the reasons for the problem.

In addition, each subject should be asked regarding the most recent day on which the study drug was taken and the time at which it was taken, at each scheduled visit at Weeks 4, 8, 12, 28, and 52, and at discontinuation, and information should be recorded in the eCRF. It is not necessary to collect information regarding the time of reference drug injection from subjects in the reference group.

#### **5.1.4** Emergency Procedures and Management of Overdose

If any symptoms have developed as a result of an overdose of ASP015K or etanercept, the investigator/sub-investigator will provide emergency treatment appropriate for each symptom under full monitoring to ensure the safety of the subject.

Experience with administration of ASP015K to humans remains limited, and overdose of ASP015K has not been reported. However, based on data on AEs from previous studies, the first sign of overdose of ASP015K may be nausea, diarrhoea, other GI symptoms, CPK increased, lymphocytes decreased, or neutropenia.

The following information regarding an overdose of etanercept is available in its package insert:

The maximum tolerated dose of etanercept has not been established in humans. Single IV doses up to 60 mg/m² have been administered to healthy volunteers in an endotoxemia study without evidence of dose-limiting toxicities. The highest dose level evaluated in RA patients has been a single IV loading dose of 32 mg/m² followed by SC doses of 16 mg/m² (up to 25 mg/m²) administered twice weekly. There is no known antidote to etanercept.

#### 5.1.5 Criteria for Continuation of Treatment

Subjects in the ASP015K 100 mg, ASP015K 150 mg, or placebo groups who completed the assessment at study visit at Week 52 may participate in an extension study (015K-CL-RAJ2) if they wish to do so. Subjects in the reference group will not be eligible for participation in the open-label extension study. Each subject must provide informed consent for the extension study before completing the assessment at study visit at Week 52.

#### 5.1.6 Compliance Rules to be Observed by Subjects throughout the Study

The investigator, sub-investigator, or collaborator will explain the following to the subjects during the study period.

- In principle, subjects should visit the study center for the study visit on the specified date. The visits may be adjusted within an allowable range, but the visit dates must be adjusted so that the intervals between the specified visits are 5 weeks at most.
- The subject should visit the study center on the day of each study visit without taking the dose of the study drug for that day prior to the visit. The subject in the reference group should also visit the study center on the day of each scheduled study visit without

injecting etanercept if he/she has an injection on that visit day. The subject must also fast for at least 8 hours prior to the blood sampling at the time of the study visit. If a subject must make an unscheduled visit due to adverse events, etc., on the day of taking the study drug, the unscheduled visit will be prioritized regardless of whether the study drug was taken and the timing of meals.

- If a new treatment (starting to take a new drug or use a new therapy, etc.) has been prescribed by another department or another medical institution during the study period, the subject should contact the investigator/sub-investigator before starting to use the new treatment, and follow the instructions given by the investigator/sub-investigator. If it is not possible to contact the investigator/sub-investigator in advance, the subject should contact one of them, or the collaborator, as soon as possible.
- Any subject who wishes to take prescription medication or over-the-counter drugs unconfirmed by the investigator/sub-investigator should confirm with the investigator, sub-investigator, or collaborator in advance whether to take the drug. If it is not possible to contact the investigator/sub-investigator in advance, the subject should contact one of them, or the collaborator, as soon as possible.
- Subjects must practice contraception through 2 or more appropriate contraceptive methods throughout the study period, and for 90 days after the end of treatment with the study drug or reference drug in the case of male subjects and for 60 days after the end of treatment with the study drug or reference drug in the case of female subjects of childbearing potential.
- Female subjects must not breastfeed throughout the study period and for 60 days after the end of treatment with the study drug or reference drug.
- ➤ If another visit is instructed by the investigator/sub-investigator due, for example, to a laboratory finding subject to CPK monitoring and liver function monitoring, the subject must promptly visit the study center.

# 5.2 Demographics and Baseline Characteristics

#### 5.2.1 Demographics

The date of obtaining informed consent, date of birth, sex, and study region will be recorded in the eCRF. In addition, height, history of smoking, and alcohol consumption habits will be confirmed during the screening test period and recorded in the eCRF.

#### 5.2.2 Medical History

Diseases cured before the initiation of treatment with the study drug or reference drug will be regarded as previous diseases, and diseases that remain uncured at the initiation of treatment with the study drug or reference drug will be regarded as concurrent diseases. All concurrent diseases will be investigated, and the name of the diagnosis will be recorded in the medical record or other source documents, as well as in the eCRF. Serious infectious diseases (in the

past 365 days from baseline) and herpes zoster are subjects to investigation, and the history, name of diagnosis, date of onset, and date of recovery will be entered in the eCRF.

#### 5.2.3 Diagnosis of the Target Disease, Severity, and Duration of Disease

Information on following items will be obtained and entered in the eCRF:

- Name of diagnosis, onset date of RA, and criteria for the classification of RA used for the diagnosis (Appendix 5, Appendix 6)
- ACR 1991 revised criteria for the classification of global functional status in RA (Appendix 7) at screening
- Classification of disease stage/progression of RA (Appendix 8) at screening
- History of surgery for RA (name of surgery, joint operated, possibility of joint assessment)
- Names of RA treatment drugs used in the past (DMARD), treatment response, and tolerability
- Names of DMARDs to which subjects are considered to have an inadequate response for this study, doses of DMARDs before 90 days prior to the initiation of screening, timing for the initiation of DMARDs for the treatment of RA, treatment response, and tolerability

# 5.3 Efficacy, Pharmacodynamics, and Pharmacokinetics Assessments

#### **5.3.1** Efficacy Assessments

#### **5.3.1.1** Tender and Swollen Joint Counts

(1) Tender joint count

The investigator/sub-investigator will examine the subject for tender joints, assessing the 68 joints listed below, and confirm the location of each tender joint. The 28 joints subject to assessment will also be examined for tender joints and the location will be confirmed. The number of respective confirmed joints and the date of assessment will be entered in the eCRF.

#### (2) Swollen joint count

The investigator/sub-investigator will examine the subject for swollen joints, assessing the 66 joints listed below, with the exception of the hip joints, and confirm the location of the swollen joints. The 28 joints subject to assessment will also be examined for swollen joints and the location will be confirmed. The number of respective confirmed joints and the date of assessment will be entered in the eCRF.

### Table Joints Subject to Assessment

Temporomandibular joints (2), sternoclavicular joints (2), acromioclavicular joints (2), shoulder joints (2)\*, elbow joints (2)\*, wrist joints (2)\*, DIP joints (8), PIP joints of both hands (10)\*, MCP joints (10)\*, hip joints (2), knee joints (2)\*, ankle joints (2), tarsal bones (2), MTP joints (10), interphalangeal joint joints of toes (2), PIP joints of both feet (8)

#### 5.3.1.2 Assessment of Pain and Overall Assessment of Disease Activity

The following assessments will be performed on the scheduled assessment days from the baseline:

- (1) Subject's assessment of pain: The subject assesses his/her own pain severity on a VAS of 0–100 mm on the questionnaire form. The measured value and the date of assessment will be entered in the eCRF.
- (2) SGA: The subject assesses his/her own disease activity on a VAS of 0–100 mm on the questionnaire form. The measured value and the date of assessment will be entered in the eCRF.
- (3) PGA: The investigator/sub-investigator assesses the subject's disease activity on a VAS of 0–100 mm on the physician assessment table. The measured value and the date of assessment will be entered in the eCRF.

#### 5.3.1.3 Acute Phase Reactants (CRP and ESR)

Only CRP is measured during the screening test period. Blood sampling is performed on the scheduled assessment days from baseline to measure CRP and ESR. The measurement of CRP will be performed by the central laboratory, and the measurement of ESR will be performed by each study center. These results will be used to calculate DAS28, SDAI, and ACR response criteria assessment. One-hour value of ESR will be measured. The measured ESR and the date of measurement will be entered in the eCRF.

#### 5.3.1.4 EULAR Response Criteria

Based on DAS28 scores and changes in DAS28 scores before and after treatment with the study drug or reference drug, EULAR Response Criteria categorize response to treatment as "No response," "Moderate response," or "Good response" according to the definition given in the table below [van Gestel et al, 1996; van Gestel et al, 1998].

<sup>\*:</sup> Joints subject to DAS28 assessment

| DAS28 after treatment | DAS28 response (DAS28 before treatment - DAS28 after treatment) | | |
|---|---|---|---|
| DAS28 after treatment | > 1.2 | $> 0.6$ and $\leq 1.2$ | ≤ 0.6 |
| ≤ 3.2 | Good response | Moderate response | No response |
| $> 3.2 \text{ and } \le 5.1$ | Moderate response | Moderate response | No response |
| > 5.1 | Moderate response | No response | No response |

#### 5.3.1.5 DAS28

The subject's DAS28 will be calculated at the screening visit and on each subsequent assessment day using data from the following assessments, together with the formula shown below [Prevoo et al, 1995; van der Heijde et al, 1990; Fransen et al, 2003; Mallya et al, 1982; Wolfe, 1997].

- TJC (28 joints)
- SJC (28 joints)
- CRP or ESR
- SGA

```
[When CRP is used] DAS28 = 0.56\sqrt{(TJC)} + 0.28\sqrt{(SJC)} + 0.36 \ln{(CRP + 1)} + 0.014 \times SGA + 0.96 [When ESR is used] DAS28 = 0.56\sqrt{(TJC)} + 0.28\sqrt{(SJC)} + 0.70 \ln{ESR} + 0.014 \times SGA
```

DAS28 score is assessed as below.

- High disease activity: DAS28 score of > 5.1
- Moderate disease activity: DAS28 score of > 3.2 and  $\le 5.1$
- Low disease activity: DAS28 score of  $\leq 3.2$

If the DAS28 score is less than 2.6, the subject will be considered to be in DAS28 remission [van Gestel et al, 1998; Fransen and van Riel, 2005].

#### **5.3.1.6 SDAI Score**

The SDAI score at baseline and Week 12 will be calculated using data from the following assessments, together with formula shown below [Smolen et al, 2003; Aletaha and Smolen, 2005; Felson et al, 2011].

- TJC (28 joints)
- SJC (28 joints)
- SGA
- PGA
- CRP (mg/dL)

$$SDAI = TJC + SJC + SGA + PGA + CRP$$

The SDAI score is assessed as below.

- High disease activity: SDAI score exceeding 26
- Moderate disease activity: SDAI score exceeding 11 and not greater than 26

  - Low disease activity: SDAI score exceeding 3.3 and not greater than 11

If the SDAI score is 3.3 or less, the subject will be considered to be in SDAI remission.

#### 5.3.1.7 ACR Response Criteria Assessment

ACR Response Criteria [Felson et al, 1995] measure improvement in TJC, SJC, subject's assessment of pain, SGA, PGA, assessment of physical function using HAQ-DI, and acute phase reactant (CRP or ESR).

The ACR20 response requires that all criteria from (1) to (3) below be met. The ACR50 response indicates a 50% improvement in all criteria from (1) to (3) below, and the ACR70 response similarly indicates a 70% improvement. In this study, [5] is assessed with CRP.

- (1) TJC:  $\geq$  20% reduction compared with baseline
- (2) SJC:  $\geq$  20% reduction compared with baseline
- (3)  $\geq$  20% improvement in 3 or more of the following 5 parameters compared with baseline
  - [1] Subject's assessment of pain
  - [2] SGA
  - [3] PGA
  - [4] Disability Index (HAQ-DI)
  - [5] CRP or ESR

#### **5.3.1.8** Patient Reported Outcomes/Assessments

Subjects will complete the following assessments at baseline and on days specified in the Schedule of Assessments. The outcome of the assessments will be recorded in the eCRF. In principle, the copy of assessment forms will be provided to the sponsor.

- HAQ-DI [Fries et al, 1982; Ramey et al, 1992]
- SF-36v2<sup>®</sup> [Ware, 2004]
- WPAI [Takeuchi T, 2011; Reilly MC, 1993]

#### 5.3.2 Pharmacodynamic Assessments

Blood samples will be collected at baseline and on days specified in the Schedule of Assessments. At the study visit points where blood sample collection for PK assessment is performed, sample collection for PD assessment will be performed before treatment with the study drug or reference drug and at the same time as that for the sampling for PK assessment. These measurements will be performed at the central laboratory, and the results will be reported to the sponsor and the study center after the breaking of the treatment code.

#### 5.3.2.1 Lymphocyte Subsets

Lymphocyte subset quantification of CD3, CD4, CD8, CD16, CD19, CD56, and CD56/16 will be performed, and the changes from baseline will be calculated. The date of blood sampling will be entered in the eCRF.

#### 5.3.2.2 Biomarkers for Efficacy and Safety Assessments

To assess the effects of ASP015K on biomarkers, VEGF and MMP-3 will be measured, and the changes from baseline will be calculated. The date of blood sampling will be entered in the eCRF.

Additional analysis may be performed for biomarkers for efficacy and safety assessments based on study results using blood samples that have been collected during the study and biobanked (i.e., residual sample stored for retrospective analysis). These could include biomarkers of inflammation, bone or cartilage metabolism, or inhibitory activity of JAK, but other biomarkers may also be subject to analysis.

#### **5.3.3** Pharmacokinetic Assessments

The concentration of ASP015K will be measured. If necessary, the concentrations of ASP015K metabolites will also be measured. Subjects in the reference group will be excluded from concentration measurement and will not provide blood samples. Blood samples will be collected at baseline and on the days specified in the Schedule of Assessments. Moreover, the date and time on which the last dose of study drug will be taken just prior to blood sampling will be recorded in the eCRF, together with the date and time of blood sampling.

The sampling for the assessment of post-dose concentrations will be performed as a substudy at study centers approved for the sampling. The sampling for the assessment of post-dose concentrations will be performed at either Week 4 or Week 8, 2 hours after the administration of the study drug (the acceptable time range is from 1 hour to 4 hours post-dose). In addition, the sampling for post-dose concentrations will be performed on the same day as central ECG at Week 4 or Week 8, promptly after the central ECG.

# 5.4 Safety Assessment

The following tests and observations will be made for the purpose of safety assessments at baseline and on the days specified in the Schedule of Assessments. The requirements for reporting and analysis of information on drug-induced liver injury (DILI) are in Appendix 4 "Liver Safety Monitoring and Assessment." If marked liver function abnormal in Appendix 4 is observed, the investigator or the responsible personnel should contact the sponsor or CRO by telephone or fax (within 24 hours of awareness).

#### 5.4.1 Vital Signs

Blood pressure (in the sitting position), pulse rate, and body temperature at rest will be measured at screening and on the days specified in the Schedule of Assessments. The date of measuring and measurements taken (blood pressure and the measuring position, systolic blood pressure, diastolic blood pressure, pulse rate, and body temperature) will be entered in the eCRF.

#### 5.4.2 Body Weight

Body weight will be measured at screening and on the days specified in the Schedule of Assessments. The date of measuring and measurements taken will be entered in the eCRF.

#### **5.4.3** Adverse Events

The survey period for AEs will be from the initiation of treatment with the study drug or reference drug to before the initiation of administration in the extension study or until the end of follow-up.

Events that occurred after treatment with the study drug or reference drug until before the initiation of administration in the extension study or until the end of follow-up will be recorded as AEs. Concurrent diseases that worsened during the study will also be recorded as AEs. AEs that occurred after the subject has completed the study plan or has been discharged from the hospital or the study center will not be recorded.

AEs that have not resolved before the initiation of administration in the extension study or at the end of follow-up must be followed-up until resolved or judged to be no longer clinically significant or until they become chronic to the extent that they can be fully characterized. If the event resolves during the study period, the date of resolution is to be entered in the eCRF.

See Appendix 4 "Liver Safety Monitoring and Assessment" for the assessment of AEs caused by DILI.

Herpes zoster should be entered as an AE information in the eCRF, and also, a separate Herpes Zoster (shingles) Worksheet should be prepared, and a copy should be submitted to the sponsor. If the sponsor considers necessary and requests for submission of forms for the purpose of providing additional information on other AEs, a form must be prepared to report to the sponsor.

#### 5.4.3.1 Adverse Events of Possible Hepatic Origin

Subjects with liver-derived AEs associated with hepatic function abnormal should be monitored carefully.

#### 5.4.4 Laboratory Assessments

The below hematology, biochemistry, fasting lipid profile, and urinalysis will be performed at screening and on each of the days specified in the Schedule of Assessments. These measurements will be performed at the central laboratory. For the period of performing additional laboratory tests for DILI, see Appendix 4 "Liver Safety Monitoring and Assessment."

Additional sampling and tests may be performed if it is considered necessary by the investigator/sub-investigator or if retesting is considered necessary by the investigator/sub-investigator because the results could not be obtained due to defects in the sample. Additional tests and analysis may be performed based on the study results using blood samples for laboratory assessments that have been collected during the study and have been biobanked (i.e., residual samples stored for retrospective analyses).

Hematology, biochemistry (including fasting lipid profile tests), urinalysis
 The following hematology, biochemistry, fasting lipid profile tests, and urinalysis will be performed:

Hematology

Hemoglobin, hematocrit, erythrocytes (RBC), leukocytes (WBC), differential WBC (neutrophils, lymphocytes, monocytes, eosinophils, basophils), platelet count

Each blood cell count will be calculated from the differential WBC.

Biochemistry

Na, K, Ca, Cl, Mg, HCO<sub>3</sub>, BUN, phosphorus, glucose, creatinine, ALP, AST (GOT), ALT (GPT), γ-GTP, total bilirubin, total protein, albumin, uric acid, CPK, LDH, serum amylase, eGFR, β-D-glucan

Fasting lipid profile

Total cholesterol, LDL, HDL, triglycerides

The date of sample collection will be entered in the eCRF.

- ➤ Blood specimens for scheduled fasting lipid profile tests should be drawn after the subject has fasted for at least 8 hours, unless it is at termination or at an unscheduled visit when the subject could not fast.
- Urinalysis

pH, specific gravity, protein (qualitative), glucose (qualitative), keton bodies (qualitative), bilirubin (qualitative), occult blood, sediment

2) Pregnancy test (for females only)

Pregnancy testing will be performed from screening according to the Schedule of Assessments. Serum pregnancy testing is required only at screening, and urine pregnancy testing will be performed after baseline. The serum pregnancy testing will be performed by the central laboratory and the urine pregnancy testing will be performed by the study centers using the kits provided by the central laboratory. If, in the serum pregnancy test, hCG level exceeds ULN, but the possibility of pregnancy can be completely ruled out by another test, the subject is eligible for enrollment. Pregnancy testing is not subject to the safety assessment.

- If a urine pregnancy test is positive at any time, a negative serum pregnancy is required for the subject to continue participation in the study. If the possibility of pregnancy can be completely ruled out by another test, the subject may continue to participate in the study.
- The pregnancy tests need not be performed if the possibility of pregnancy can clearly be ruled out, such as if the woman is postmenopausal and has not had a menstrual period for 1 year or more, or has had a hysterectomy, bilateral oophorectomy, etc.

#### 3) Tuberculosis test

The tuberculosis test will be performed at screening to confirm the eligibility of the subject in accordance with Exclusion Criterion 14. T-SPOT or QuantiFERON Gold test is the preferential test for tuberculosis infection. If T-SPOT or QuantiFERON Gold test cannot be performed, tuberculin skin test may be performed instead. Tuberculin test and QuantiFERON Gold test cannot be performed at the central laboratory in Japan. Tuberculin test and T-SPOT cannot be performed at the central laboratory in Korea and Taiwan. Tuberculosis test is not required at screening provided that there is documentation of a negative tuberculosis test within 90 days prior to baseline.

#### 4) Hepatitis test

Tests for HBs antigens, HBs antibodies, the HBV-DNA assay, HBc antibodies, and HCV antibodies will be performed at the screening visit to confirm the eligibility of the subject. If a subject is positive for either or both HBc antibodies and HBs antibodies, the subject will be monitored during treatment with the study drug or reference drug by performing an HBV-DNA assay at scheduled visits and early termination. Safety analysis will not be performed for the results of HBV-DNA assays from baseline.

#### 5) CPK monitoring

If an increase in CPK is observed, in accordance with Section 5.4.4.1 CPK Monitoring, when CPK is retested, CPK, CK-MB, troponin T, and aldolase should also be tested. Urinalysis (blood and microscopy) will be performed as part of the targeted physical examination.

#### 5.4.4.1 CPK Monitoring

If a CPK elevation is observed after treatment with the study drug or reference drug is initiated, CPK will be monitored as follows:

- If laboratory testing reveals CPK > 3 × ULN, and the subject is asymptomatic, retest CPK preferably within 1 week of previous blood sampling to confirm it. Subsequently, retest CPK weekly (from the date of the initial CPK elevation) until CPK is ≤ 3 × ULN or is stable according to the judgment of the investigator/sub-investigator. If the retest cannot be performed within 1 week of blood sampling, which marks the starting point of CPK monitoring, suspension or interruption of the study drug or reference drug should be considered until the retest results are obtained.
- In subjects whose baseline CPK is already > 3 × ULN, if laboratory testing reveals CPK > 2 × baseline, and the subject is asymptomatic, retest CPK preferably within 1 week of previous blood sampling to confirm it. Subsequently, retest CPK weekly (from the date of CPK elevation to > 2 × baseline) until CPK is ≤ 2 × baseline, or is stable in the judgment of the investigator/sub-investigator. If the retest cannot be performed within 1 week of blood sampling, which marks the starting point of CPK monitoring, suspension or interruption of the study drug or reference drug should be considered until the retest results are obtained.

- If CPK is > 10 × ULN at any time, treatment with the study drug or reference drug will be immediately suspended or interrupted (see Section 3.4 Discontinuation Criteria for Individual Subjects), and retest CPK.
- If there is a symptomatic CPK elevation (CPK elevation > 1.5 × ULN accompanied by severe and unusual episodes of myalgia, muscular weakness, or muscle twitching), as reported by the investigator/sub-investigator, treatment with the study drug or reference drug will be immediately discontinued (see Section 3.4 Discontinuation Criteria for Individual Subjects).

In the retest for CPK monitoring, the following tests will be performed in addition to CPK measurements. The content of the subject questionnaire will be entered in the eCRF.

- ➤ Laboratory tests (Measurement parameters: CK-MB, troponin T, aldolase)
- A targeted physical examination\* and subject questionnaire to assess muscle strength and pain
  - \*: As part of the targeted physical examination, urinalysis (blood and microscopy) will be performed.

#### **5.4.4.2** Hepatic Function Abnormal

If laboratory testing for a subject enrolled in the study and receiving the study drug or reference drug reveals an increase in serum aminotransferase (ALT, AST)  $> 3 \times ULN$  or TBL  $> 2 \times ULN$ , at least 4 parameters (ALT, AST, ALP, and TBL) of the usual hepatic function test parameters should be retested. The retest should be performed between 48 hours and 72 hours after notification of the test results.

For additional information on monitoring and the assessment of the hepatic function test, see Appendix 4 "Liver Safety Monitoring and Assessment."

If laboratory testing for a subject enrolled in the study receiving the study drug or reference drug reveals an increase in serum aminotransferase (ALT, AST)  $> 3 \times \text{ULN}$  and TBL  $> 2 \times \text{ULN}$ , the investigator will determine whether it is an SAE. Even if the abnormality is not considered an SAE by the investigator/sub-investigator, it will be reported to the sponsor or CRO in writing as in the case of SAEs.

### 5.4.5 Physical Examination

A physical examination will be performed at scheduled visits and early termination to confirm physical findings.

Physical findings and RA symptoms will be confirmed at unscheduled visits whenever possible.

#### 5.4.6 12-lead Electrocardiogram (ECG)

A 12-lead ECG will be obtained at screening and on the assessment dates specified in the Schedule of Assessments. The investigator/sub-investigator will confirm the ECG chart, assess the results as "normal," "abnormal but not to a clinically important degree," or

"clinically important abnormality," and record the results of the assessment in the CRF. If the finding is "abnormal but not to a clinically important degree" or "clinically important abnormality," the finding will be recorded in the CRF.

The screening 12-lead ECG must be performed within 4 weeks prior to the first dose of study drug or reference drug. In addition, the clinical interpretation of the results of this examination must be completed prior to the first dose of study drug or reference drug.

#### 5.4.7 Radiography

Chest radiography will be performed at screening and on the assessment dates specified in the Schedule of Assessments. Chest radiography examination will be performed at early termination if it is determined necessary by the investigator/sub-investigator. However, chest radiography at screening is not required provided that there is documentation of a normal chest radiograph within 90 days from baseline. The investigator/sub-investigator will confirm the chest radiographic images, assess the results as "normal," "abnormal but not to a clinically important degree," or "clinically important abnormality," and the investigator/sub-investigator record the results of the assessment in the eCRF.

If the results of chest radiography at screening reveal findings of tuberculosis, the subject's eligibility will be decided in accordance with Exclusion Criterion 14.

#### 5.4.8 Central ECG

Central ECG is conducted as sub-study at the sites which approved blood sampling for post-dose drug concentration. Subjects in the reference group will be excluded from Central ECG. Central ECG is performed at baseline before study drug administration, as well as before study drug administration and 2 hours after study drug administration at Week 4 or Week 8 on the same day as blood sampling for post-dose drug concentration at Week 4 or Week 8. 12-lead ECG is performed as Central ECG. The measurement date and time of central ECG is recorded in the eCRF.

The measuring and transmittal method of central ECG in the handling manual provided by sponsor is followed. The QT interval, QTcF and QTcB will be calculated by the third party using the Central ECG data transmitted and the method of ECG analysis is described in the handling manual prepared by the third party.

# 5.5 Adverse Events and Other Safety Aspects

### 5.5.1 Definition of Adverse Events (AEs)

An AE is defined as any untoward medical occurrence in a subject administered a study drug or reference drug that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study drug or reference drug, whether or not related to the study drug or reference drug.

An abnormality identified during a medical test (e.g., laboratory parameter, vital sign, ECG data, physical examination) should be defined as an AE only if the abnormality meets one of the following criteria:

- Induces clinical signs or symptoms
- Requires active intervention
- Requires suspension, interruption, or discontinuation of the study drug or reference drug
- The abnormality or laboratory test value is clinically significant based on the opinion of the investigator or other responsible personnel

The particulars to be noted with respect to the AE are the name of the event, date of onset, date of disappearance, severity (at peak time), seriousness, treatment of the study drug or reference drug, other treatment, outcome, causal relationship to the study drug or reference drug, and rationale for the assessment of causal relationship. The rationale for the assessment of the causal relationship does not need to be recorded for all AEs but only at the request of the sponsor. The severity of each event should be recorded on a scale of Grade 1 to Grade 5 in the eCRF, and the causal relationship to the study drug should be recorded as "Probable," "Possible," or "Not related" (see Section 5.5.3 Criteria for Causal Relationship to the Study Drug and Section 5.5.4 Criteria for Defining the Severity of an Adverse Event). The treatment of the AE (whether it was treated with pharmacotherapy or by other means) and the treatment of the study drug or reference drug should be recorded in the medical record or other source documents and in the eCRF. The outcome should be recorded in the medical record or other source documents and in the eCRF as "resolved," "alleviated," "unresolved," "resolved but with late effects," "death," or "unknown."

#### 5.5.2 Definition of Serious Adverse Events (SAEs)

An adverse event is considered "serious" if, in the view of either the investigator or Sponsor, it results in any of the following outcomes:

- Results in death
- Is life threatening (an adverse event is considered "life-threatening" if, in the view of either the investigator or Sponsor, its occurrence places the subject at immediate risk of death. It does not include an adverse event that, had it occurred in a more severe form, might have caused death)
- Results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions
- Results in congenital anomaly, or birth defect
- Requires inpatient hospitalization or leads to prolongation of hospitalization (hospitalization for treatment/observation/examination caused by AE is to be considered as serious)
- Other medically important events

Medical and scientific judgment should be exercised in deciding whether expedited reporting is appropriate in other situations, such as important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the

subject or may require intervention to prevent one of the other outcomes listed in the definition above. These events, including those that may result in disability/incapacity, should also usually be considered serious. Examples of such events are intensive treatment in an emergency room or at home for allergic bronchospasm; blood dyscrasias or convulsions that do not result in hospitalization; or development of drug dependency or drug abuse.

In addition, all sponsor's clinical studies have the requirement that all the medical events described in Appendix 3 "Events Always considered to be Serious" and Appendix 4 "Liver Safety Monitoring and Assessment" be reported by the investigator as SAEs even if they do not meet the aforementioned conditions.

#### 5.5.3 Criteria for Causal Relationship to the Study Drug

AEs that fall under either "Possible" or "Probable" should be defined as "AEs whose relationship to the study drug could not be ruled out." This definition also applies to those occurring in the reference group.

| Causal Relationship<br>to Study Drug | Related Assessment Criteria |
|---|---|
| Not related | A clinical event, including laboratory test abnormality, with a temporal relationship to drug administration which makes a causal relationship improbable, and/or in which other drugs or underlying disease provide plausible explanations. |
| Possible | A clinical event with a reasonable time sequence to administration of the drug, to which one of the following applies: • Could also be explained by concurrent/underlying disease or other drugs • Information on drug withdrawal is lacking or unclear |
| Probable | <ul> <li>A clinical event with a reasonable time sequence to administration of the drug, to which one of the following applies:</li> <li>Recurs upon re-administration of the drug, or disappears or is alleviated when the drug is withdrawn.</li> <li>Cannot be explained by concurrent/underlying disease or other drugs or is unlikely to be attributable to them</li> </ul> |

#### 5.5.4 Criteria for Defining the Severity of an Adverse Event

The AE grades will be based on NCI-CTCAE [Japan Clinical Oncology Group (JCOG), 2011]. Items unspecified by these criteria will be assessed according to the following criteria and recorded.

| Grade | Assessment Criteria |
|---|---|
| Grade 1 (Mild) | Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. |
| Grade 2 (Moderate) | Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL. |
| Grade 3 (Severe) | Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL. |
| Grade 4 (Life-threatening or incapacitating) | Life-threatening consequences; urgent intervention indicated. |
| Grade 5 (Death) | Death related to AE. |

#### 5.5.5 Reporting of Serious Adverse Events (SAEs)

In the case of a serious adverse event (SAE), the investigator must contact the Sponsor/delegated CRO by telephone or fax immediately (within 24 hours of awareness) [in case of Japan: in addition to reporting to the head of the study center].

The investigator should complete and submit an SAE report containing all information that is required by the Regulatory Authorities to the Sponsor/delegated CRO [in case of Japan: and to the head of the study center] by fax immediately (within 24 hours of awareness). If the faxing of an SAE report is not possible or is not possible within 24 hours, the investigator should inform the Sponsor or delegated CRO by phone.

SAEs occurring in the reference group should also be reported in the same way as above.

For contact details, see Section II CONTACT DETAILS OF KEY SPONSOR'S PERSONNEL.

Please fax the SAE report to:

Contact Information of the Sponsor

| TEL: | , FAX: |
|-----------------|-------------|
| Contact Informa | tion of CRO |
| Japan: | |
| TEL: | |
| FAX: | |
| Korea: | |
| TEL: | , FAX: |
| Taiwan: | |



#### 5.5.6 Follow-up of Adverse Events

All AEs occurring during or after the subject has discontinued the study are to be followed up until resolved or judged to be no longer clinically significant, or until they become chronic to the extent that they can be fully characterized.

If during AE follow-up, the adverse event progresses to an "SAE", or if a subject experiences a new SAE, the investigator must immediately report the information to the Sponsor/delegated CRO.

Even if the subject does not return to normal or to his/her previous state, follow-up can be considered no longer necessary or finished when the following procedures have been taken:

[1] Follow-up is considered no longer necessary if:

The investigator/sub-investigator judges that follow-up of the subject is no longer necessary because the AE's relationship to the study drug or reference drug could be ruled out, and this judgment is considered appropriate by the sponsor.

[2] Follow-up is considered finished if:

The investigator judges that follow-up of the subject is no longer necessary based on the progression made during follow-up; the reason for such a judgment is entered as a comment in the CRF for follow-up, and the sponsor judges that the reason is acceptable with regard to the safety of the subject concerned.

For details of follow-up of DILI (medical history, concomitant medications, history of alcohol intake and narcotic use), see Appendix 4 "Liver Safety Monitoring and Assessment."

#### 5.5.7 Procedure in Case of Pregnancy

If a woman is proven to be pregnant during treatment with the study drug or reference drug or within 28 days from the end of treatment or early termination, the investigator should report this information to the sponsor/CRO in the same manner as that for an SAE. The expected date of delivery, last menstruation, estimated fertility date, pregnancy result and neonatal data etc., should be included in this information.

The investigator or other responsible personnel will handle the pregnancy in the same manner as an SAE and will follow the medical status of the mother, as well as the fetus, and report the outcome to the sponsor.

When the outcome of the pregnancy falls under the criteria for SAEs [spontaneous abortion, induced abortion, stillbirth, death of newborn, congenital anomaly (including anomaly in a miscarried fetus)] and when information on newborn falls under the criteria for SAEs (including death, congenital anomaly, and other anomalies), the investigator should respond in accordance with the report procedure for SAEs.

Additional information regarding the outcome of a pregnancy (which is categorized as an SAE) is mentioned below.

"Spontaneous abortion" includes abortion and missed abortion.

Death of a newborn within 1 month after birth should be reported as an SAE regardless of its relationship with the study drug.

If a newborn dies more than 1 month after the birth, it should be reported if a relationship between the death and intrauterine exposure to the study drug is judged as "possible" by the investigator or other responsible personnel.

In the case of a delivery of a living newborn, the "normality" of the newborn is evaluated at the birth.

"Normality" of the miscarried fetus is evaluated by visual examination unless test results which indicate a congenital anomaly are obtained prior to miscarriage.

If a male subject impregnates his partner during the conduct of the clinical study, the subject should report the pregnancy to the investigator or other responsible personnel, and the investigator must report the pregnancy to the sponsor/CRO.

# 5.5.8 Supply of New Information Affecting the Conduct of the Study

In Japan:

- 1. When information is obtained regarding serious and unexpected adverse drug reactions (or other) that are specified in Article 80-2 Paragraph 6 and Article 273 of the Law for Ensuring the Quality, Efficacy, and Safety of Drugs and Medical Devices, the Sponsor should inform all the investigators involved in the clinical study, the head of the study site, and the regulatory authorities of such information. The head of the study site who receives such information will decide whether the clinical study should be continued after hearing the opinions of the IRB. The investigator will supply the new information to the subjects, in compliance with Section 8.2.3.3 Supply of New and Important Information Influencing the Subject's Consent and Revision of the Written Information.
- 2. In addition to the above item 1, when the head of the study site receives the revisions of the Investigator's Brochure, protocol, or written information, information on the matters covering the quality of the study drug, efficacy and safety, information necessary for conducting the clinical study properly, or documents to be examined by the IRB should be sent to the IRB.
- 3. According to the Pharmaceutical and Medical Device Safety Information Reporting System, information regarding serious and unexpected adverse drug reactions and others occurring in the reference group will be reported to the regulatory authorities or marketing authorization holders. The sponsor will not report serious and unexpected adverse drug reactions and others that occurred in the reference group because the marketing authorization holder provides such information to medical institutions through revisions to the package inserts.

#### In Korea and Taiwan:

When the sponsor gains new information suggesting adverse impact on the subjects' safety, safe conduct of the clinical study, or the IRB/IEC approval for study continuation, the sponsor will immediately notify all investigators, all study sites, and relevant regulatory authorities.

The sponsor must immediately report SAEs to all participating principal investigators, study sites (and the IRBs/IECs if appropriate) in compliance with local requirements and the relevant regulatory authorities.

When information necessary for conducting the clinical study properly (including "Dear Doctor Letters" but not limited to that) becomes available and leads to a protocol amendment, the sponsor should inform the regulatory authorities, as well as all investigators and medical institutions involved in the clinical study, who will then inform the IRB/IEC of such information, and when needed, should amend the Written Information.

# 5.5.9 Deviations from the Protocol and Other Actions Taken to Avoid Life-Threatening Risks to Subjects

The investigator must not deviate from or amend the protocol without prior written consent of sponsor and prior written approval from IRB/IEC.

In Japan:

When the investigator does not follow the protocol in order to avoid urgent risks for subjects, the investigator should take the following actions.

- 1. Describe the contents of the deviation or amendment and the reasons for it in a written notice, and immediately send the document stating the deviation or amendment and the reasons to the Sponsor and the head of the study site. Keep a copy of the notice.
- 2. Consult with the Sponsor at the earliest possibility for cases in which it is necessary to amend the protocol. Obtain approval for a draft of the amended protocol from the IRB and the head of the study site as well as written approval from the Sponsor.

In Korea and Taiwan:

When the investigator does not follow the protocol in order to avoid urgent risks for subjects, the investigator should report to sponsor, IRB/IEC, and regulatory authority (if applicable) in compliance with local requirements.

# 5.6 Test Drug Concentration

The plasma concentrations of ASP015K will be measured in the samples collected at the time points in Table 1 Schedule of Assessments, except the reference group. The concentrations of ASP015K metabolites H1, H2, and H4 will also be measured if necessary.

In the placebo group, the concentrations of samples collected during the period of the administration of placebo will not be measured, but the concentration of samples collected after switching to ASP015K 100 mg or ASP015K 150 mg will be measured. The concentration of the sample collected on the day of the visit for switching will be measured as baseline.

The subject registration center will provide information on study drug assignment to the institution performing measurements of drug concentrations. The institution performing measurements of drug concentrations will measure the drug concentrations of samples of subjects in the placebo group who switched to ASP015K 100 mg or ASP015K 150 mg.

Concentration measurements will be performed by central laboratory using a validated, established LC-MS/MS method [Test No.: (ASP015K, H2), (H4), (H1)]. The lower limit of quantification is 0.25 ng/mL. Blood samples for drug concentration (2 mL/sample) will be collected into a 2 mL vacutainer tube containing ethylenediamine-tetra-acetic acid (K<sub>3</sub>EDTA-3K). See the written explanation of testing procedure enclosed in the clinical laboratory testing kit for descriptions of the procedure for sampling blood and storing and shipping the blood samples. The central laboratory will not report the results of determinations to the investigator, sub-investigator, sponsor, or other third parties until the breaking of the treatment code.

# 5.7 Other Measurements, Assessments, or Methods

#### 5.7.1 Pharmacodynamic Measurements

In this study, the following will be measured as part of the pharmacodynamic evaluation: biomarkers of bone or cartilage metabolism and lymphocyte subsets (see Section 5.3.2.2 Biomarkers for Efficacy and Safety Assessments).

Blood samples for biomarkers of bone or cartilage metabolism will be collected in a 2 mL sampling tube containing EDTA-2Na, and samples for lymphocyte subsets will be collected in a 2 mL vacutainer tube containing EDTA-2K in Japan, and in a 3 mL vacutainer tube containing EDTA-2K in Korea and Taiwan. See the written explanation of testing procedure enclosed in the clinical laboratory testing kit for descriptions of the procedure for sampling blood and storing and shipping the blood samples.

The central laboratory will not report the results to the investigator, sub-investigator, sponsor, or other third parties until the breaking of the treatment code.

#### **5.7.2** Purposes of Pharmacogenomics

- Pharmacogenomics will only be performed at study centers in Japan and Korea that have approved to the content of the research, and only those study centers will follow the procedures described in Sections 5.7, 8.2, and 8.3.
- To prepare for future research that will analyze the relationship between genes and the efficacy, safety, or pharmacokinetics of the test drug, blood samples will be collected and stored.
- To prepare for future research that will analyze the relationship between genome and the efficacy or safety of the test drug, biological samples will be stored over long-term. Details will be described in the "Bio-Banking Procedures" prepared separately.
- To prepare for future exploratory research on biomarkers that can predict the pharmacologic response [efficacy and toxicity (adverse drug reactions)] through the

- analysis of genetic information from this study or from integration of other studies using this test drug, biological samples will be collected and stored.
- If a serious adverse drug reaction is observed, samples for genomic/genetic analysis will be collected to explore the markers related to the adverse drug reaction.

### 5.7.3 Handling and Storage for Samples Used for Pharmacogenomics

To prepare for future research that will analyze the relationship between genes and the efficacy, safety, or pharmacokinetics of the study drug, blood samples will be collected and stored after obtaining consent from the subject to participate in PGx research and after randomization of blood samples and, whenever possible, before the first dose of the study drug. If it is not possible to take the sample before the first dose, it should be taken by the end of the study. The subject's consent to participate in the PGx research must be obtained after the subject has given consent to participate in the main study and by the time the blood sample for bio-banking is taken.

At study centers in Japan and Korea approved to conduct PGx research, blood samples will be taken from those subjects participating in the main study who have given written consent for the collection and storage of blood samples for use in PGx research. On one occasion during the study period, the investigator, sub-investigator, or collaborator will collect 5 mL of peripheral blood from a forearm vein(s) in a storage tube and store it at the study center at  $4^{\circ}$ C until the time of specimen collection. The date on which informed consent was obtained and the sampling date should be recorded for each subject and entered into the eCRF. The sample collection and shipping agency should then temporarily store the blood sample for PGx research (at  $-20^{\circ}$ C or  $-80^{\circ}$ C) and send it to the prolonged storage laboratory for samples used in PGx research will collect the blood samples and store them at  $-80^{\circ}$ C until it is time to analyze them. All collected PGx samples will be maintained for a period of up to 15 years after database hard lock.

• Sample anonymization: Because the specific content of the analyses to be performed in the PGx research has not yet been determined, the specimens will be double coded and anonymized. After the first code (subject identification code) has been assigned by the study center, the second code will be assigned by the prolonged storage laboratory for samples used in PGx research.

#### 5.7.4 Disposal of Pharmacogenomics Samples

At the conclusion of the retention period, or if the prolonged storage laboratory for samples used in PGx research has been notified by the investigator to the effect that the subject has withdrawn consent for PGx research or that the sponsor has decided to dispose of the stored samples, the prolonged storage laboratory for samples used in PGx research should promptly remove the labels from the tubes holding the subject's samples and dispose of the samples as appropriate. If genome/gene analysis has been performed before the end of the storage period or before consent is withdrawn, the data obtained through that analysis will not be destroyed.

#### 5.7.5 Disclosure of Genetic Information

Even if PGx research is conducted in the future, the research will be exploratory, and since any results obtained from the gene analyses (results of gene assays, relationship between genes and drug response) are expected to be lacking in accuracy and definitiveness, the results of the gene analysis will not be disclosed.

#### 5.8 Total Amount of Blood

The approximate total volume of blood required for tests performed at the central laboratory during the study period is as follows. Blood sampling for the assessment of plasma drug concentrations (trough and post-dose concentrations) will not be performed for the reference group.

Additionally, there will be 16 samplings for ESR at the study center, and the amount will differ between the centers (approximately 1 mL to 2 mL per sampling). The amount of blood required for T-SPOT and Quantiferon Gold test (tuberculosis test) to be performed at the central laboratory is 10 mL and 3 mL respectively.

Subjects who are positive for hepatitis and continuing the study will require a HBV-DNA assay at baseline and each subsequent visit after initiation of study drug or reference drug administration, and the amount of blood required is 5 mL in Japan and Taiwan, and 8.5 mL in Korea per assay respectively.

Moreover, if blood samples are required at unscheduled visits or follow-up, the amount will increase. If CK-MB, troponin T, and aldolase are measured as part of CPK monitoring, the amount of blood required is 4 mL in Japan, and 5 mL in Korea and Taiwan per assessment respectively.

| Assessment | Screening | Baseline | Week 4 | Week 8 | Week 12 | Weeks 16,<br>20, 24, 28,<br>32, 36, 40,<br>44, 48 | Week 52 or<br>at early<br>termination | Follow-<br>up | Volume of sample (mL) |
|---|---|---|---|---|---|---|---|---|---|
| Hematology,<br>biochemistry<br>(including CRP,<br>fasting lipid<br>profile test) | JP:16<br>KR:18.5<br>TW:16.5 | JP:16<br>KR:18.5<br>TW:16.5 | JP:16<br>KR:18.5<br>TW:16.5 | JP:16<br>KR:18.5<br>TW:16.5 | JP:16<br>KR:18.5<br>TW:16.5 | JP:144<br>(16 × 9)<br>KR:166.5<br>(18.5 × 9)<br>TW:148.5<br>(16.5 × 9) | JP:16<br>KR:18.5<br>TW:16.5 | JP:16<br>KR:18.5<br>TW:16.5 | JP:256<br>KR:296<br>TW:264 |
| Hepatitis test | JP:6<br>KR:3.5<br>TW:5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | JP:6<br>KR:3.5<br>TW:5 |
| Hepatitis DNA testing*3 | JP:5<br>KR:8.5<br>TW:5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | JP:5<br>KR:8.5<br>TW:5 |
| Trough concentration*1 | 0 | 2 | 2 | 2 | 2 | 2<br>(Week 28<br>only) | 2 | 0 | 12 |
| PD sampling | 0 | JP:4<br>KR:8.5<br>TW:8.5 | JP:4<br>KR:8.5<br>TW:8.5 | JP:4<br>KR:8.5<br>TW:8.5 | JP:4<br>KR:8.5<br>TW:8.5 | JP:4<br>KR:8.5<br>TW:8.5<br>(Week 28<br>only) | JP:4<br>KR:8.5<br>TW:8.5 | JP:4<br>KR:8.5<br>TW:8.5 | JP:28<br>KR:59.5<br>TW:59.5 |
| PGx*1 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 5 |
| Post-dose<br>concentration<br>(if performed)*1 | | | 2 | 2 | | | | | 2 |
| Total | JP:27<br>KR:30.5<br>TW:26.5 | JP:27<br>KR:34<br>TW:27 | JP:24* <sup>2</sup><br>KR:31<br>TW:29 | JP:22<br>KR:29<br>TW:27 | JP:22<br>KR:29<br>TW:27 | JP:150<br>KR:177<br>TW:159 | JP:22<br>KR:29<br>TW:27 | JP:20<br>KR:27<br>TW:25 | JP:314*4<br>KR:386.5<br>TW:347.5 |

<sup>\*1:</sup> No blood sampling will be performed for the reference group and the subject in Taiwan.

<sup>\*2:</sup> For convenience, the sampling for the assessment of post-dose concentration is summarized at Week 4.

<sup>\*3:</sup> For subjects who are positive for HBs antibody/HBc antibody and require a hepatitis DNA assay at baseline and each subsequent visit, the amount of blood required is 5 mL in Japan and Taiwan, and 8.5 mL in Korea per assay.

<sup>\*4:</sup> In case of reference group, the total blood volume to be collected is 295 mL in Japan, 367 mL in Korea, and 333.5 mL in Taiwan.

#### 6 TERMINATION OF THE CLINICAL STUDY

- 1. When the sponsor is aware of information on matters concerning the quality, efficacy, and safety of the study drugs, as well as other important information that may affect proper conduct of the clinical study, the sponsor may discontinue the clinical study and send a written notice of the discontinuation along with the reasons to the investigator [unique to Japan: and the head of the study center].
- 2. If the investigator wishes to discontinue the study in the particular study center while the study is still in progress, the investigator should contact the sponsor [unique to Japan: and the head of the study center] immediately to inform them of the discontinuation and the reason for it.

3 March 2017 Astellas 

#### 7 STATISTICAL METHODOLOGY

A detailed elaboration of the statistical analysis will be included in a separate statistical analysis plan and PK analysis plan based on the opinions and advice from a medical expert and/or statistical advisor. After review, it will be finalized prior to unblinding.

# 7.1 Sample Size

One hundred subjects per group will receive the study drug and 200 subjects the reference drug (a total of 500 subjects).

[Rationale for the sample size]

Based on 015K-CL-RAJ1 result and efficacy result from other RA drugs [XELJANZ®, tablet, 5 mg, CTD (2013)] [CIMZIA, sc, 200 mg, Syringe, CTD (2012)], 62 subjects per group will provide 90% power to detect a difference assumed in the Step 2 in the closed testing procedure (described in Section 7.4.1.1 Primary Analysis) under the following assumptions. In addition, it is assumed that ACR20 response rate of each country (Japan, Korea and Taiwan) is similar.

- ACR20 response rate at Week 12 in the placebo group: 25%
- ACR20 response rate at Week 12 in the ASP015K 100 mg group: 54.5%
- ACR20 response rate at Week 12 in the ASP015K 150 mg group: 65.5%
- Two-sided significance level of 0.05

On the other hand, according to the Extent of Population Exposure to Assess Clinical Safety for Drugs Intended for Long-term Treatment of Non-life-threatening Conditions (PAB/PCD Notification No.592, dated 24 May 1995), ("the long-term treatment guideline"), a sample size of 300-600 subjects under long-term treatment (6 months) is adequate to observe delayed adverse events at a reasonable frequency (generally, 0.5% to 5%) and to observe whether there is an increase in high-frequency adverse events during the later stage of treatment. For treatment lasting 1 year, 100 subjects is acceptable. It is also described in "Guidelines on methodology for clinical assessment of antirheumatic drugs" (PFSB/ELD Notification No. 0217001, dated 17 February 2006) that 100 subjects for 1 year are necessary.

Therefore, to collect data for 300 subjects for 6 month period, and for 100 subjects for 1 year period in both ASP015K 100 mg and 150 mg groups among 015K-CL-RAJ2/RAJ3/RAJ4 studies as long-term treatment data, approximately 80 subjects per treatment group (400 subjects in total) as a target are necessary to be enrolled in Japan. In addition, the target sample size for Taiwan is set at 10 subjects per treatment group (50 subjects in total) as a target in consideration of the requirement of regulatory authority in Taiwan (10% or more Taiwan subjects) and target sample size for Korea is also set at 10 subjects per treatment group (50 subjects in total) as a target. Therefore, the target sample size per treatment group is set at 100 subjects in total for 3 regions.

[Rationale for the sample size for the reference group]

The target sample size for the reference group was set at 200 subjects, considering the followings:

- Incidence rates for serious infections from post marketing studies for approved biologic drugs: approximately 1.0% to 3.6% reported in post-marketing all-case surveillance [ACTEMRA®, drip infusion, 80 mg, 200 mg, 400 mg, final reports for all patients ] [ORENCIA®, drip infusion, 250 mg, information for appropriate drug usage] [HYUMIRA®, sc, 40 mg, Syringe 0.8 mL, information for appropriate drug usage]; and approximately 2.4% in the 5 mg group and approximately 1.5% in the Adalimumab group, as revealed by pooled analysis of the phase III tofacitinib study [XELJANZ®, tablet, 5 mg, CTD (2013)]
- o Operational feasibility

Setting the sample size of reference group as 200, it can be detectable at least 1 subject with 95% confidence probability for AE which occurs at 1.5% incidence rate.

# 7.2 Analysis Set

The study analyses will be performed on the following analysis sets. Final judgments on inclusion/exclusion of subjects from the analyses will be made at the Case Review based on the opinions and advice from a medical expert and/or statistical advisor.

#### 7.2.1 Full Analysis Set (FAS)

FAS will consist of all subjects who are randomized and receive at least 1 dose of the study drug or reference drug. This will be the primary data set for efficacy analyses.

#### 7.2.2 Per Protocol Set (PPS)

PPS includes all subjects of FAS who meet the following criteria. PPS is defined based on the data up to Week 12.

- Have no violation of inclusion criteria:
- Do not meet any exclusion criteria possibly interfering with the efficacy evaluation;
- Receive study or reference treatment for 8 weeks (56 days) or longer from the initiation of treatment to Week 12\* (those who have discontinued the study drug or reference drug due to the lack of efficacy should be included in PPS);
- Have study or reference treatment compliance of 75% or higher for 12 weeks after treatment;
- Have evaluable primary efficacy variables; and
- Have no major protocol violations after registration.

Subjects who are considered to have no impact on the efficacy evaluation at the Case Review Meeting will also be included in PPS, if they are not satisfying these criteria.

\*: The duration of treatment with the study drug will be calculated by subtracting the first day of study drug treatment from the date of treatment completion plus 1 day, and the

duration of treatment with the reference drug will be calculated by subtracting the first day of reference drug treatment from the date of treatment completion plus 8 days.

#### 7.2.3 Safety Analysis Set (SAF)

SAF is defined as all subjects who received at least 1 dose of the study drug or reference drug.

# 7.2.4 Pharmacokinetic Analysis Set (PKAS)

PKAS will consist of all subjects who receive at least 1 dose of the study drug and who provide samples for drug concentrations for at least 1 time point.

#### 7.2.5 Pharmacodynamics Analysis Set (PDAS)

All subjects who receive at least 1 dose of the study drug or 1 injection of the reference drug and who provide samples for the determination of pharmacodynamic parameters at least 1 time point will be included in PDAS.

# 7.3 Demographics and Other Baseline Characteristics

Demographics and other baseline characteristics will be summarized by treatment group (ASP015K 100 mg, ASP015K 150 mg, placebo, reference groups) for SAF. Descriptive statistics will include sample size, mean, standard deviation, minimum, median and maximum for continuous variables, and frequency and percentage for categorical variables. To detect a possible treatment imbalance among treatment groups, chi-squared test will be used to analyze categorical variables and one-way analysis of variance (ANOVA) will be used to analyze continuous variables. The significance level is set at 0.05.

# 7.4 Analysis of Efficacy

Efficacy analysis will be conducted on FAS and PPS. The interpretation of results from statistical tests will be based on FAS. In the primary analysis of the primary variable, the purpose of using PPS is to assess the robustness of the results from the statistical tests based on FAS. Primary efficacy variable analysis will be performed for the ASP015K 100 mg, ASP015K 150 mg, and placebo groups, and only summary statistics will be calculated for the reference group. Unless otherwise noted, analysis will performed for the treatment groups at allocation (ASP015K 100 mg, ASP015K 150 mg, placebo, reference groups) and, if necessary, for the treatment groups taking into consideration a switch from placebo to active treatment (ASP015K 100 mg, ASP015K 150 mg, placebo—ASP015K 100 mg, placebo—ASP015K 150 mg, reference groups).

# 7.4.1 Analysis of Primary Variable

#### 7.4.1.1 Primary Analysis

Primary analysis will be conducted on FAS. For the ACR20 response at Week 12/ET, pairwise comparisons to placebo will be performed at each ASP015K dose level using

logistic regression model with treatment group (Placebo, ASP015K 100 mg, and ASP015K 150 mg) as the factor and the prior biologic-DMARD-IR, concomitant DMARD use, and study region (Japan, Korea, and Taiwan) as the covariates. For multiplicity adjustment, following closed testing procedure will be done.

- Step 1. ACR20 response at Week 12/ET: ASP015K 150 mg vs. Placebo
- Step 2. ACR20 response at Week 12/ET: ASP015K 100 mg vs. Placebo

The null hypotheses will be tested at a two-sided significance level of 0.05.

For the missing data imputation of ACR20 at Week 12/ET, Last Observation Carried Forward (LOCF) methodology will be used.

#### 7.4.1.2 Secondary Analysis

The same analysis of the primary variable as described in Section 7.4.1.1 will be conducted using PPS. A sensitivity analysis will be conducted to impute the missing data. In addition the same analysis as the primary analysis will be conducted for Japanese subjects. Furthermore, a re-randomization test by the Monte Carlo sampling method will be performed as a sensitivity analysis to evaluate the appropriateness of the results of the dynamic allocation.

#### 7.4.1.3 Subgroup Analysis

Subgroup analyses for sex, age categories, prior biologic-DMARD-IR, concomitant DMARD use during the treatment period with the study drug or reference drug, study region, and others may be explored.

#### 7.4.2 Analysis of Secondary Variables

For secondary efficacy endpoints, binary variables such as Percentage of subjects achieving ACR50 response at Week 12/ET, and Percentage of subjects achieving ACR70 response at Week 12/ET will be analyzed (to Week 12/ET) using logistic regression model as described in the primary analysis with treatment group as the factor and the prior biologic-DMARD-IR, concomitant DMARD use during the study period and study region (Japan, Korea and Taiwan) as the covariates. Continuous variables, such as Change from baseline/Day 1 to Week 12/ET in DAS28-CRP and DAS28-ESR scores, will be analyzed using analysis of covariance (ANCOVA) with treatment group as the factor, and the prior biologic-DMARD-IR, concomitant DMARD use, study region (Japan, Korea, and Taiwan), and baseline value as the covariates. Each ASP015K group will be compared with placebo group (to Week 12/ET) and multiplicity for the secondary efficacy variables will not be adjusted.

# 7.5 Analysis of Safety

The following analyses will be performed on SAF. Unless otherwise noted, analysis will performed for the treatment groups at allocation (ASP015K 100 mg, ASP015K 150 mg, placebo, reference groups) and, if necessary, for the treatment groups after placebo was

switched to active treatment (ASP015K 100 mg, ASP015K 150 mg, placebo–ASP015K 100 mg, placebo–ASP015K 150 mg, reference groups). In addition, analysis will be performed for each study region (Japan, Korea, and Taiwan).

#### 7.5.1 Adverse Events

AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA/J). The incidence of AEs, SAEs, AEs leading to discontinuation, and AEs whose relationship to study drugs or reference drugs could not be ruled out will be summarized by system organ class and preferred term, as well as the treatment group. The incidence of AEs by severity will also be summarized.

### 7.5.2 Laboratory Assessments

Descriptive statistics will be used to summarize clinical laboratory measurements and the change from baseline if quantitative, by time point.

#### 7.5.3 Vital Signs

Descriptive statistics will be used to summarize vital sign measurements and the change from baseline by time point.

#### 7.5.4 12-lead ECG

The frequency of each category of 12-lead ECG results will be summarized by time point.

#### 7.5.5 QT assessment

Descriptive statistics will be used to summarize QT assessment (including QTc assessment) measurements and the change from baseline.

The frequency of each category of QT assessment (including QTc assessment) will be summarized by time point.

In addition, the relationship between quantity of QT change and concentration of ASP015K may be explored.

#### 7.5.6 Body Weight

Descriptive statistics will be used to summarize measurements by time point.

# 7.6 Analysis of Pharmacokinetics

A detailed elaboration of the PK analysis will be included in a separate PK analysis plan. The trough plasma concentrations of ASP015K will be summarized by treatment group and visit. In addition, the same PK analysis will be conducted for each study region (Japan, Korea, and Taiwan). Exploratory population PK analysis may be performed by pooling the results obtained so far.

# 7.7 Other Analyses

# 7.7.1 Analysis of Pharmacodynamics

Analysis will be performed in PDAS. Descriptive statistics will be used to summarize PD measurements and the change from baseline by time point.

### 7.7.2 Analysis of Pharmacogenomics

At present, the content of analysis as part of pharmacogenomic research has not been determined yet. The relationship between the results from genetic analyses and study data (clinical information such as pharmacological activity, toxicity and PK) may be explored in the future. The sponsor can initiate such research once a specific methodology is established. Prior to research, the sponsor will prepare a research plan (including procedures and timing of document disposal) and have appropriateness of conduct of the research reviewed and approved by the sponsor's ethics review committee from ethical and scientific viewpoints.

# 7.8 Interim Analysis (and Early Discontinuation of the Clinical Study)

Not applicable. Review of safety data and safety evaluation will be completed by an independent DSMB [see Section 10.1 Independent Data and Safety Monitoring Board (DSMB)] during the study in accordance with separate SOP.

# 7.9 Handling of Missing Data, Outliers, Visit Windows, and Other Information

Final judgments on handling of missing data, outliers, visit windows, and other information will be made at the Case Review Meeting based on the opinions and advice from a medical expert and/or statistical advisor prior to treatment code breaking and included in the SAP.

The acceptable time ranges for the efficacy and safety examinations and observations from the date of initial study or reference treatment (Day 1) are defined as follows. If there are multiple data available over the same period of time, the data obtained on the date closest to the reference date will be utilized; the later date will be applied if the number of days from the reference date is equal. Subjects who have no evaluable post-dose data on ACR20, ACR50, and ACR70 response rates after initial treatment with the study drug or reference drug will be counted as non-responders and included in the analysis at the end of Week 12 (Week 12 or at early termination before Week 12).

#### 7.9.1 Handling of Schedule of Assessments of Efficacy Variables

For data after the end of study treatment, data obtained within + 2 days after the last dose is taken will be included in analysis. For data after the end of reference treatment, data obtained within + 9 days after the last dose will be included in analysis.

#### (1) TJC (68 joints)/SJC (66 joints), laboratory test (CRP)

| Time points defined in analysis | Reference date* | Acceptable time range |
|---|---|---|
| Screening | Day -28 to Day -1 | Day -28 to Day -1 |
| Baseline | Day 1 | Day 1 |
| Week 4 to Week 48** | Day $7 \times x + 1$ | Day $(7 \times x - 6)$ to Day $(7 \times x + 8)$ and |
| | | before the initiation of treatment with the |
| | | study drug or reference drug on the visit day |
| Week 52 | Day 365 | Day 358 to Day 372 |
| End of Week 12 (Week 12 or at | Day 85 | Day 2 to Day 92 |
| early termination before Week 12) | | |
| End of treatment (Week 52 or at | Day 365 | Day 2 to Day 372 |
| early termination) | | |

<sup>\*:</sup> Day 1 represents the first day of study or reference treatment. The day before the initiation of treatment with the study drug or reference drug is expressed as Day -1.

# (2) PGA and SGA (VAS), subject's assessment of pain (VAS), HAQ-DI, laboratory test (ESR)

| Time points defined in analysis | Reference date* | Acceptable time range |
|---|---|---|
| Baseline | Day 1 | Day 1 |
| Week 4 to Week 48** | Day $7 \times x + 1$ | Day $(7 \times x - 6)$ to Day $(7 \times x + 8)$ and |
| | | before the initiation of treatment with the |
| | | study drug or reference drug on the visit day |
| Week 52 | Day 365 | Day 358 to Day 372 |
| End of Week 12 (Week 12 or at | Day 85 | Day 2 to Day 92 |
| early termination before Week 12) | | |
| End of treatment (Week 52 or at | Day 365 | Day 2 to Day 372 |
| early termination) | | |

<sup>\*:</sup> Day 1 represents the first day of study or reference treatment. The day before the initiation of treatment with the study drug or reference drug is expressed as Day -1.

# (3) SF-36 v2<sup>®</sup>, WPAI

| Time points defined in analysis | Reference date* | Acceptable time range |
|---|---|---|
| Baseline | Day 1 | Day 1 |
| Week 4 to Week 28** | Day $7 \times x + 1$ | Day $(7 \times x - 6)$ to Day $(7 \times x + 8)$ and |
| | | before the initiation of treatment with the |
| | | study drug or reference drug on the visit day |
| Week 52 | Day 365 | Day 358 to Day 372 |
| End of Week 12 (Week 12 or at | Day 85 | Day 2 to Day 92 |
| early termination before Week 12) | | |
| End of treatment (Week 52 or at | Day 365 | Day 2 to Day 372 |
| early termination) | | |

<sup>\*:</sup> Day 1 represents the first day of study or reference treatment. The day before the initiation of treatment with the study drug or reference drug is expressed as Day -1.

#### 7.9.2 Handling of Schedule of Assessments of Safety Variables

For data obtained after the end of study treatment, the data obtained within + 2 days after the last dose is taken will be included in analysis. For data after the end of reference treatment, data obtained within + 9 days after the last dose will be included in analysis.

<sup>\*\*:</sup> Represents the reference date and acceptable time range for Week x.

<sup>\*\*:</sup> Represents the reference date and acceptable time range for Week x.

<sup>\*\*:</sup> Represents the reference date and acceptable time range for Week x.

# (1) Physical examination, vital signs, laboratory test [hematology, biochemistry, urinalysis, and pregnancy test (serum and urine)]

| Time points defined in analysis | Reference date* | Acceptable time range |
|---|---|---|
| Screening | Day -28 to Day -1 | Day -28 to Day -1 |
| Baseline | Day 1 | Day 1 |
| Week 4 to Week 48** | Day $7 \times x + 1$ | Day $(7 \times x - 6)$ to Day $(7 \times x + 8)$ and |
| | | before the initiation of treatment with the |
| | | study drug or reference drug on the visit day |
| Week 52 | Day 365 | Day 358 to Day 372 |
| End of Week 12 (Week 12 or at | Day 85 | Day 2 to Day 92 |
| early termination before Week 12) | | |
| End of treatment (Week 52 or at | Day 365 | Day 2 to Day 372 |
| early termination) | | |

<sup>\*:</sup> Day 1 represents the first day of study or reference treatment. The day before the initiation of treatment with the study drug or reference drug is expressed as Day -1.

#### (2) Laboratory test (fasting lipid profile test)

| Time points defined in analysis | Reference date* | Acceptable time range |
|---|---|---|
| Baseline | Day 1 | Before the initiation of treatment with the |
| | | study drug or reference drug on Day 1 and |
| | | at least 8 hours after the last meal |
| Week 12 | Day 85 | Day 78 to Day 92 |
| Week 28 | Day 197 | Day 190 to Day 204 |
| Week 40 | Day 281 | Day 274 to Day 288 |
| Week 52 | Day 365 | Day 358 to Day 372 |
| End of Week 12 (Week 12 or at | Day 85 | Day 2 to Day 92 |
| early termination before Week 12) | | |
| End of treatment (Week 52 or at | Day 365 | Day 2 to Day 372 |
| early termination) | | |

<sup>\*:</sup> Day 1 represents the first day of study or reference treatment. The day before the initiation of treatment with the study drug or reference drug is expressed as Day -1.

#### (3) 12-lead ECG

| Time points defined in analysis | Reference date* | Acceptable time range |
|---------------------------------|-------------------|-----------------------|
| Screening | Day -28 to Day -1 | Day -28 to Day -1 |
| Week 28 | Day 197 | Day 190 to Day 204 |
| Week 52 | Day 365 | Day 358 to Day 372 |
| End of treatment (Week 52 or at | Day 365 | Day 2 to Day 372 |
| early termination) | - | |

<sup>\*:</sup> Day 1 represents the first day of study or reference treatment. The day before the initiation of treatment with the study drug or reference drug is expressed as Day -1.

<sup>\*\*:</sup> Represents the reference date and acceptable time range for Week x.

# (4) Body weight

| Time points defined in analysis | Reference date* | Acceptable time range |
|---|---|---|
| Screening | Day -28 to Day -1 | Day -28 to Day -1 |
| Week 12 | Day 85 | Day 78 to Day 92 |
| Week 28 | Day 197 | Day 190 to Day 204 |
| Week 40 | Day 281 | Day 274 to Day 288 |
| Week 52 | Day 365 | Day 358 to Day 372 |
| End of Week 12 (Week 12 or at | Day 85 | Day 2 to Day 92 |
| early termination before Week 12) | | |
| End of treatment (Week 52 or at | Day 365 | Day 2 to Day 372 |
| early termination) | | |

<sup>\*:</sup> Day 1 represents the first day of study or reference treatment. The day before the initiation of treatment with the study drug or reference drug is expressed as Day -1.

#### (5) QT assessment (except the reference group)

| Time points defined in analysis | Reference date* | Acceptable time range |
|---|---|---|
| Baseline | Day 1 | Day 1 |
| | | Before the initiation of treatment with the |
| | | study drug |
| Week 4 or 8 | Day 29 or Day 57 | Before the initiation of treatment with the |
| (before study drug administration) | | study drug on Reference date $\pm 7$ |
| Week 4 or 8 | Day 29 or Day 57 | 2 hours post-dose (reference time, but within |
| (after study drug administration) | | the range of 1 hour to 4 hours post-dose is |
| | | acceptable) on Reference date $\pm 7$ |

#### 7.9.3 Handling of Schedule of Assessments of Pharmacodynamic Variables

For data obtained after the end of study treatment, data obtained within + 2 days after the last dose will be included in analysis. For data after the end of reference treatment, data obtained within + 9 days after the last dose will be included in analysis.

#### (1) Biomarkers and lymphocyte subsets

| Time points defined in analysis | Reference date* | Acceptable time range |
|---|---|---|
| Baseline | Day 1 | Before the initiation of treatment with the |
| | | study drug or reference drug on Day 1 |
| Week 4 to Week 28** | Day $7 \times x + 1$ | Day $(7 \times x - 6)$ to Day $(7 \times x + 8)$ and before |
| | | the initiation of treatment with the study |
| | | drug or reference drug on the visit day |
| Week 52 | Day 365 | Day 358 to Day 372 |
| End of Week 12 (Week 12 or at | Day 85 | Day 2 to Day 92 |
| early termination before Week 12) | | |
| End of treatment (Week 52 or at | Day 365 | Day 2 to Day 372 |
| early termination) | | |

<sup>\*:</sup> Day 1 represents the first day of study or reference treatment.

<sup>\*\*:</sup> Represents the reference date and acceptable time range for Week x.
# 7.9.4 Handling of Schedule of Assessments of Pharmacokinetic Variables

# (1) Trough concentration (except the reference group)

| Time points defined in analysis | Reference date* | Acceptable time range |
|---|---|---|
| Baseline | Day 1 Before the initiation of treatment with the | |
| | - | study drug on Day 1 |
| Weeks 4, 8, 12, 28, and 52** | Day $7 \times x + 1$ | Day $(7 \times x - 6)$ to Day $(7 \times x + 8)$ and within |
| | | 19 to 29 hours between the time of treatment |
| | | with the study drug before blood collection |
| | | and the time of blood collection |

<sup>\*:</sup> Day 1 represents the first day of study treatment.

# (2) Post-dose concentration (except the reference group)

| Time points defined in analysis | Reference date* | Acceptable time range |
|---|---|---|
| Week 4 or Week 8** | Day $7 \times x + 1$ | Day $(7 \times x - 6)$ to Day $(7 \times x + 8)$ and |
| | | within 1 to 4 hours between the time of |
| | | treatment with the study drug before blood |
| | | collection and the time of blood collection |

<sup>\*:</sup> Day 1 represents the first day of study treatment.

<sup>\*\*:</sup> Represents the reference date and acceptable time range for Week x.

<sup>\*\*:</sup> Represents the reference date and acceptable time range for Week x.

# 8 OPERATIONAL AND ADMINISTRATIVE CONSIDERATIONS

# 8.1 Procedure for Clinical Study Quality Control

#### 8.1.1 Data Collection

The investigator is responsible to ensure that all data in the eCRFs and queries are accurate and complete and that all entries are verifiable with source documents. These source documents should be appropriately maintained by the study center.

The investigator, sub-investigator, or collaborator will enter data collected using an Electronic Data Capture (EDC) system. The investigator, sub-investigator, or collaborator will enter the data, in principle within 5 working days from the creation of the data (date of visit by the subject, date of obtaining information, etc.).

In principle, the name of AE must be entered within 5 working days of the date of confirming its occurrence. The name of concomitant drug/therapy must also be entered within 5 working days of the awareness of its use. Other information to be entered in the eCRF must be entered immediately on receipt.

The monitor should verify the data in the eCRFs with source documents and confirm that there are no inconsistencies between them.

For screening failures, the minimum demographic data (sex, birth date, study region, and informed consent date) and, if reason for screening failure is to be obtained, the screening failure log (SFL) will be collected.

Measurements of laboratory tests, pharmacodynamic parameters, and plasma drug concentrations will be performed by central laboratory. The Data Science Department of the sponsor will obtain the laboratory test results, pharmacodynamic measurements, and plasma drug concentration measurements in an electronic format from central laboratory at predefined intervals during the study.

| Analysis of Central ECG will be perfor | med by | | The Data Science |
|---|---|---|---|
| Department of the sponsor will obtain t | he quali <mark>ty assu</mark> | red analysis data in | an electronic |
| format from | at predefined | timing. | |
| The central laboratory and | | will provide the spo | onsor with a copy of |
| the complete and clean data, together w | ith the quality | control report. | |

# **8.1.2** Specification of Source Documents

Source data must be available at the study center to document the existence of the study subjects and substantiate the integrity of study data collected. Source data must include the original documents relating to the study as well as those relating to the medical treatment and medical history of the subject.

The following information should be included in the source medical records:

- Demographic data (study region, birth date, sex, height, and body weight)
- Inclusion and exclusion criteria details

- Participation in study and signed and dated informed consent forms
- Visit dates
- Medical history and physical examination details
- Key efficacy and safety data
- AEs and symptomatic treatment
- The results of the relevant examination (e.g., ECG charts, radiographic data, etc.)
- Laboratory test slips/reports
- Details of dispensing and returning the study drug or reference drug
- Reason for premature discontinuation
- Records of RA diagnosis and evaluation, patient questionnaires (e.g., HAQ-DI, SF-36v2<sup>®</sup>, WPAI)
- Subject questionnaire for CPK monitoring
- Herpes Zoster (shingles) Worksheet

If the following data are not included in medical records, the entries in the eCRFs are treated as source data:

- Dates of AE occurrence and resolution, its severity, seriousness, outcome, causality to the study drug, and rationale for the causality
- Route of administration, treatment dates, and reason of use for previous and concomitant drugs
- Type, treatment dates, and reason of use for previous and concomitant therapies
- Presence or absence of abnormal 12-lead ECG readings, abnormal findings
- Date, reason, and background/details for discontinuation
- Other comments

# 8.1.3 Clinical Study Monitoring

The sponsor or delegated CRO is responsible for monitoring the clinical study to ensure that subject's human rights, safety, and well-being are protected, that the study is properly conducted in adherence to the current protocol and GCP, and study data reported by the investigator/sub-investigator are accurate and complete and that they are verifiable with study-related records such as source documents. The sponsor is responsible for assigning study monitor(s) to this study for proper monitoring. They will monitor the study in accordance with planned monitoring procedures.

#### 8.1.4 Direct Access to Source Data/Documents

The investigator and the study site must accept monitoring and auditing by the Sponsor or delegated CRO as well as inspections from the IRB/IEC and relevant regulatory authorities. In these instances, they must provide all study-related records, such as source documents (refer to Section 8.1.2 "Specification of Source Documents") when they are requested by the Sponsor monitors and auditors, the IRB/IEC, or regulatory authorities. The confidentiality of the subject's identities shall be well protected consistent with local and national regulations when the source documents are subject to direct access.

# 8.1.5 Data Management

Data management will be coordinated by the Data Science Department of the sponsor in accordance with SOPs for data management. All study specific processes and definitions will be documented by Data Management. eCRF entry and correction process will be referenced in the CRF instructions. Coding of medical terms will be performed using MedDRA.

# 8.2 Ethics and Protection of Subject Confidentiality

# 8.2.1 Institutional Review Board (IRB)/ Independent Ethic Committee (IEC)

Prior to a conclusion of study contracts for the present study, the protocol and documents used to obtain patient consent shall be reviewed and approved by the IRBs/IECs of each study center in order to ensure that subject's human rights, safety, and well-being are protected.

# 8.2.2 Ethical Conduct of the Study

The investigator(s) and all parties involved in this study should conduct the study in adherence to GCP, ICH Guidelines, and the applicable laws/regulations.

In Japan:

Moreover, PGx research should be conducted consistent with "Ethical Guidelines for Human Genome/Gene Analysis Research" (Notification No. 1 issued by Ministry of Education, Culture, Sports, Science and Technology/Ministry of Health, Labour and Welfare [MHLW]/Ministry of Economy, Trade and Industry in 2004) and "Clinical Trials with Pharmacogenomics Analysis" (Notification from the Director of the Evaluation and Licensing Division, Pharmaceutical and Food Safety Bureau, MHLW, dated 30 September 2008).

## 8.2.3 Informed Consent of Subjects

# 8.2.3.1 Subject Information and Consent

Prior to execution of the clinical study, the investigator should prepare the written informed consent form and other written information in collaboration with the sponsor and revise the information whenever necessary. The investigator should submit the written or revised informed consent form and any other written information to the sponsor to be subject to prior approval by IRB/IEC.

- The investigator or other responsible personnel is responsible for explaining the nature and purpose of the study and other study-related matters to subjects using the written information and for obtaining their full understanding and written consent to participate in the study of their own free will.
- The investigator or other responsible personnel who provided explanations (including collaborators who gave supportive information, if applicable) and the subject should sign, [unique to Japan: seal,] and date the written information.

- Informed consent must be obtained by the time the observations/examinations during the pre-investigational period are performed before treatment with the study drug or reference drug.
- The investigator or other responsible personnel must give a copy of the signed [unique to Japan: or sealed] consent form to the subject with the written information and store the original appropriately in accordance with the rules at the study center concerned.
- The investigator or other responsible personnel should note the following when obtaining consent from subjects:
  - No subject may be subjected to undue influence, such as compulsory enrollment into a study.
  - The language and expressions used in the written information should be as plain and understandable as possible for the subjects. Subjects should be given the opportunity to ask questions and receive satisfactory answers to the inquiry, and should have adequate time to decide whether or not to participate in the study. Written information should not contain any language or contents that causes the subject to waive or appears to waive any legal rights, or that releases/mitigates or appears to release/mitigate the study center, the investigator/sub-investigator, collaborators, or the sponsor from liability for negligence.

The investigator will retain the signed consent forms, which will be made available (for review only) to the study monitor and auditor on request.

# 8.2.3.2 Subject Information and Consent for PGx Research

The study centers in Japan and Korea with approval of the conduct of PGx research should obtain the consent to participate in PGx research in addition to the study entry. Prior to execution of the clinical study, the investigator should prepare the written informed consent form for PGx research in collaboration with the sponsor and revise the information whenever necessary. The written or revised written informed consent form and any other written information should be submitted to the sponsor and be subject to prior approval by the IRB/IEC.

Only subjects who have given consent for the study entry are subject to the consent for PGx research. Subjects can withdraw consent for PGx research only, separately from withdrawal of consent for the study entry. Procedures provided in Section 8.2.3.1 Subject Information and Consent should also be applied when obtaining consent for PGx research.

All of the remaining samples for PGx research obtained from the subject who has withdrawn consent for PGx research should be disposed of, except those anonymized.

The signed consent forms will be retained by the investigator and made available (for review only) to the study monitor and auditor upon request.

# 8.2.3.3 Supply of New and Important Information Influencing the Subject's Consent and Revision of the Written Information

1. The investigator or other responsible personnel will immediately inform the subject orally whenever new information becomes available that may be relevant to the subject's

3 March 2017 Astellas 

consent or may influence the subject's willingness to continue participation in the study (e.g., report of serious adverse drug reactions). The communication should be documented in the subject's medical records, and it should be confirmed whether the subject is willing to remain in the study or not.

- 2. If the investigator recognizes the necessity to revise the written information in the terms and conditions applicable to paragraph 1, the written information should be revised immediately based upon the newly available information, and be re-approved by the IRB/IEC.
- 3. The investigator or other responsible personnel should obtain written informed consent to continue participation in the study with the revised written information defined in paragraph 2, even if subjects are already informed of the relevant information orally. The investigator or other responsible personnel who provided explanations (including collaborators who gave supportive information, if applicable) and the subject should sign and date the informed consent form, or write down his/her name, place a personal seal, and date the form. The investigator or other responsible personnel should give a copy of the signed [unique to Japan: or sealed] informed consent form to the subject who had given consent with the written information and store the original appropriately as done for the previous informed consent.

# 8.2.4 Subject Confidentiality

Medical information of individual subjects obtained as a result of this study is considered confidential, and disclosure to third parties is prohibited. Medical information of individual subjects may be given only after approval of the subject to the subject's physician or to other appropriate medical personnel responsible for the subject's well-being.

The sponsor, its board members or its employee shall not disclose any confidential information on subjects obtained during the performance of their duties in the clinical study without justifiable reasons.

All individuals and organizations involved in the study must pay very careful attention to protect subjects' privacy with appropriate measures, for example, by prohibiting the use of any private information that may identify a subject (e.g., name or address). These details shall be processed in accordance with the applicable laws such as Personal Information Protection Law and regulatory requirement(s).

Even though any individuals involved in the study including the study monitors and auditors, may get to know matters related to subject's privacy due to direct access to source documents, or from other sources, they may not leak the content to third parties.

## **8.3** Administrative Matters

# 8.3.1 Arrangement for Use of Information and Publication of the Clinical Study

Information concerning the study drug, patent applications, processes, unpublished scientific data, the Investigator's Brochure and other pertinent information is confidential and remains

the property of the Sponsor. Details should be disclosed only to the persons involved in the approval or conduct of the study. The investigator may use this information for the purpose of the study only. It is understood by the investigator that the Sponsor will use the information obtained during the clinical study in connection with the development of the drug and therefore may disclose it as required to other clinical investigators or to regulatory agencies. In order to allow for the use of the information derived from this clinical study, the investigator understands that he/she has an obligation to provide the Sponsor with all data obtained during the study.

The study will be considered for publication or presentation at (scientific) symposia and congresses. The investigator or other responsible personnel will be entitled to publish or disclose the data generated at their respective study center only after submitting all transcripts, texts of presentations, and abstracts related to the study to the sponsor at least 90 days prior to the intended submission for publication or any other disclosure. Because such disclosure of study results is presupposed, it is important that the information concerning the invention is protected by a patent, through the preparation and submission of a patent application. Moreover, publication of facts and opinions summarized by the investigator is not restricted. The sponsor will inform the investigator in writing of any objection or question arising within 30 days of receipt of the proposed publication material. After agreement between investigator(s) and sponsor, the manuscript can be submitted for publication.

## 8.3.2 Documents and Records Related to the Clinical Study

The sponsor will provide the investigator or other responsible personnel and/or study center with the following:

- Study protocol (and amendments, where applicable)
- Investigator's Brochure (and amendments, where applicable)
- eCRFs and other related documents, SAE Worksheet
- Study drugs and reference drugs with all necessary documentation
- Study contract

In order to start the study, the investigator and/or study center is required to provide the following documentation to the sponsor:

- Signed Investigator's Statement in this protocol and eCRF
- Current curricula vitae (CVs) of all investigators
- List of sub-investigators and collaborators
- IRB/IEC approval of the protocol, protocol supplement (if applicable) including a membership list with names and qualification (copy)
- Instruction and decision of the head of the study center (if applicable)
- Study contract and memorandum
- Laboratory normal reference ranges (including modification and amendment)

At the end of the study, the sponsor is responsible for the collection of:

- Other study documentation
- Unused study drugs and reference drugs (if applicable)

The investigator will archive all study data (e.g., subject identification code list, source documents, and investigator's file) and relevant correspondence. These documents are to be kept on file for the appropriate term determined by local regulations (for study centers in the US, 2 years from the approval of NDA or termination of IND). The sponsor will archive and retain all documents pertaining to the study according to local regulations.

## In Japan:

The records to be retained at the study sites are the ones listed as essential documents in GCP. These records shall be retained by the head of the study site or the record keeper designated by the head until notice issued by the Sponsor on completion of the retention period is received. These documents are also subject to direct access and should be provided upon request from the Sponsor or regulatory authorities.

The following are the major documents to be retained at the study center.

Source documents (clinical data, documents, and records for preparing the eCRF)

- 1. Hospital records, medical records, test records, memoranda, or check lists for evaluation, administration records, medication diary (for self-administration in the reference group), data recorded by automatic measuring instruments, reproductions or transcripts verified as precise copies, microfiche, negative films, microfilms/magnetic media, radiographic films, subject files and study-related records kept at either a pharmacy, a laboratory, or medical technical office, as well as subject registration forms, laboratory test slips including central measurement, worksheets/forms [e.g., questionnaires at CPK monitoring, Herpes Zoster (shingles) Worksheet] specified by the sponsor, records of clinical coordinators, and records related to the clinical study selected from those verified in other departments or hospitals.
- 2. Contracts, written informed consent forms, written information, and other documents or their copies prepared by the study personnel.
  A letter of request for clinical study (including a request for continuation/amendment), letter of request for review, notice of clinical study contract, clinical study contract, notification of discontinuation or completion of clinical study, written information for informed consent (including revisions), signed and dated written informed consent (including revisions), CVs of investigators, list of sub-investigators and collaborators, list of signatures and print of seals (copy), and electronic media storing the eCRF data,
- 3. Documents obtained related to the adequacy of conducting the clinical study by the head of the study centers and the protocol, documents obtained related to the adequacy of conducting the clinical study whose period exceeds one year or the adequacy of continuously conducting the clinical study from which information on adverse drug

reactions is obtained, and other documents obtained.

An agreed-upon protocol (including revisions), Investigator's Brochure (including revisions), SOP for the investigator, materials and information supplied by the sponsor (e.g., AE report), matters reported by the investigator (revisions of the protocol, AE report, etc.), SOP for the IRB/IEC, the list of names of the IRB/IEC members, material for IRB/IEC review (including continuous deliberation), IRB/IEC review records (including continuous deliberation), and the review result report of the IRB/IEC (including continuous deliberation), etc.

- 4. Records of control for study drugs and other duties related to the clinical study Procedure for controlling the study drugs, drug inventory and accountability record, vouchers for the receipt and return of the study drugs, and other records of the prescriptions for concomitant medications The documents of the Independent DSMB (minutes, SOPs, and others) shall be retained by the sponsor.
- [Unique to Japan and Korea: Records of PGx research samples

The study centers where the conduct of PGx research has been approved should retain the Subject Identification Code List and written informed consent form (including amendments) for PGx research for up to 15 years after the data lock point in order to comply with the subject's consent withdrawal of PGx research and storage of their samples.]

#### In Korea and Taiwan:

The investigator and the study site should archive study-related documents in compliance with applicable regulatory requirements. The investigator and the study site must take measures to prevent accidental or premature destruction of these documents during the required retention period.

#### 8.3.3 Protocol Amendment and/or Revision

Any changes to the study that arise after approval of the protocol must be documented as protocol amendments and/or revisions. Depending on the nature of the amendment and/or revision, either IRB/IEC/regulatory authorities' approval or notification is required. The changes and revisions will become effective only after the approval of the sponsor, the investigator, and the IRB/IEC (if applicable), [Unique to Japan: followed by the approval of the head of the study center.]

# 8.3.4 Insurance of Subjects and Others

If a subject suffers any study-related injury, the Sponsor will compensate appropriately according to the severity and duration of the damage. However, if it was caused intentionally or was due to gross negligence by the study site, the Sponsor will consult with the study site about handling the injury, based on the agreed study contract. Compensation for the study-related injury is provided by the following procedures:

- 1. If a subject incurs an injury as a result of participation in the clinical study, the study site should provide medical treatment and other necessary measures. The Sponsor/delegated CRO should be notified of the injury.
- 2. When the subject claims compensation from the study site for the above study-related injury, or such compensation may be claimed, the study site should immediately communicate the fact to the Sponsor/delegated CRO. Both parties should work together towards compensation settlement.
- 3. The Sponsor shall pay compensation or indemnification and bear expenses necessary for the settlement as provided in the clinical contract.
- 4. The Sponsor shall make an arranging for insurance and take measures necessary to ensure the compensation or indemnification mentioned above.

# 8.3.5 Signatory Investigator for Clinical Study Report

ICH E3 guidelines recommend and EU Directive 2001/83/EC requires that a final study report that forms part of a marketing authorization application be signed by a coordinating or principal investigator. The coordinating investigator will have the responsibility to review the final study results to confirm to the best of his/her knowledge it accurately describes the conduct and results of the study. A coordinating investigator will be selected from the participating investigators by sponsor prior to database lock.

3 March 2017 Astellas 

# 9 QUALITY ASSURANCE

The sponsor is implementing and maintaining quality assurance and quality control systems with written SOPs to ensure that studies are conducted and data are generated, documented (record), and reported in compliance with the protocol, GCP, and applicable regulatory requirement(s).

The Sponsor or Sponsor's designee may arrange to inspect/audit the clinical study at any or all study centers. The auditor is independent from the clinical monitoring and project management team at the Sponsor. The audit may include on-site review of study-related documents/records, eCRF, and source documents. Direct access to these documents will be required by the auditors.

# 10 STUDY ORGANIZATION

# 10.1 Independent Data and Safety Monitoring Board (DSMB)

An independent DSMB will be organized to review the unblinded safety data, to make a decision on whether to continue or stop the study, or modify the protocol with respect to the safety, and to provide the sponsor with recommendations. The DSMB should follow the procedures separately defined in details, including the frequency of meetings, blind-breaking and data review.

# 10.2 Other Evaluation Committee(s)

Not applicable.

# 10.3 Other Study Organization

See Attachment.

# 10.4 Registration of Subjects



<sup>\*</sup> At the Week 12 visit, only subjects in the placebo group will be switched to receiving ASP015K 100 mg or ASP015K 150 mg based on the allocation at baseline.

<sup>\*\*</sup> Only subjects in the ASP015K 100 mg, ASP015K 150 mg, or placebo groups who completed Week 52.

| <subject center="" registration=""></subject> |
|---|
| In Japan: |
| URL: |
| Service available: Everyday (365 days, 24 hours) |
| Help desk TEL: |
| (Monday to Friday: 9:00-18:00, except national holidays, and 29 December to 4 January) |
| In Korea and Taiwan: |
| URL: |
| Service available: Everyday (365 days, 24 hours) |
| Help desk in Korea |
| TEL: FAX: |
| Help desk in Taiwan |
| TEL: FAX: |
| (Monday to Friday: 9:00-18:00 (Japan time), except national holidays in Japan, and 29 |
| December to 4 January) |

The investigator/sub-investigator is responsible for conducting a survey on demographics of the candidate subjects and obtaining their written consent. After obtaining written consent, the investigator/sub-investigator should make necessary entries in the case registration form on the web-based registration system. The subject registration center will notify the preregistration results to the study centers via the web-based registration system.

The investigator/sub-investigator will confirm the inclusion/exclusion criteria at baseline, and the investigator/sub-investigator will make the necessary entries in the case registration form on the web-based registration system. The registration center will confirm the fulfillment of inclusion/exclusion criteria based on the case registration information received and inform the study centers of the case inclusion or exclusion via the web-based registration system. The investigator/sub-investigator will dispense the study drug or reference drug to the subject who is considered "eligible" for study registration.

## 11 REFERENCES

- Aletaha D, Smolen J. The Simplified Disease Activity Index (SDAI) and the Clinical Disease Activity Index (CDAI): A review of their usefulness and validity in rheumatoid arthritis. Clin Exp Rheumatol 2005;23(Suppl. 39):S100-S108.
- Daniel A, Tuhina N, Alan J, et al. 2010 Rheumatoid arthritis classification: An American College of Rheumatology/European League against rhumatism collaborative initiative. Arthritis Rheum 2010; 62:2569-2581.
- Felson DT, Anderson JJ, Boers M, Bobmardier C, Furst D, Goldsmith C, et al. American College of Rheumatology preliminary definition of improvement in rheumatoid arthritis. Arthritis Rheum 1995;38:727-735.
- Felson DT, Smolen JS, Wells G, Zhang B, Tuyl LHD van, Funovitis J, et al. American College of Rheumatology/European League Against Rheumatism Provisional Definition of Remission in Rheumatoid Arthritis for Clinical Trials. Arthritis Rheum 2011;63:573-586.
- Fransen J, Riel PLCM van. The Disease Activity Score and the EULAR response criteria. Clin Exp Rheumatol 2005;23(Suppl 39):S93-9.
- Fransen J, Welsing P, Keijzer Rd, Riel P van. Disease Activity Scores using C-reactive protein: CRP may replace ESR in the assessment of RA disease activity. Ann Rheum 2003;62:151.
- Fries JF, Spitz PW, Young DY. The dimensions of health outcomes: The health assessment questionnaire, disability and pain scales. J Rheumatol 1982;9:789-793.
- Hochberg MC, Chang RW, Dwosh I, Lindsey S, Pincus T, Wolfe F. The American College of Rheumatology 1991 Revised Criteria for the Classification of Global Functional Status in Rheumatoid Arthritis. Arthritis Rheum 1992;35:498-502.
- Kremer JM, Bloom BJ, Breedveld FC, Coombs JH, Fletcher MP, Gruben D, et al. The safety and efficacy of a JAK inhibitor in patients with active rheumatoid arthritis. Arthritis Rheum. 2009;60:1895-1905.
- Mallya RK, de Beer FC, Berry H, Hamilton EDB, Mace BEW, Pepys MB. Correlation of clinical parameters of disease activity in rheumatoid arthritis with serum concentration of C-reactive protein and erythrocyte sedimentation rate. J Rheumatol 1982;9(2):224-8.
- O'Dell JR. Therapeutic strategies for rheumatoid arthritis. N Engl J Med. 2004;350:2591-602.
- Papageorgiou AC, Wikman LEK. Is JAK3 a new drug target for immunomodulation-based therapies? Trends Pharmacol Sci. 2004;25(11):558-62.
- Prevoo MLL, Hof MA van't, Kuper HH, Leeuwen MA van, Putte LBA van de, Riel PLCM van. Modified disease activity scores that include twenty-eight-joint counts. Arthritis Rheum 1995;38:44-48.
- Ramey DR, Raynauld JP, Fries JF. The health assessment questionnaire 1992: status and review. Arthritis Care & Research 1992;5:119-129.

3 March 2017 Astellas 

- Silvia G. Priori, Arthur A.Wilde, et al. HRS/EHRA/APHRS Expert consensus statement on the diagnosis and management of patients with inherited primary arrhythmia syndromes. Heart Rhythm 2013: 10; 1932-1963
- Reilly MC, Zbrozek AS, Dukes EM. The validity and reproducibility of a work productivity and activity impairment instrument. PharmacoEconomics 1993;4(5):353-65
- Smolen JS, Breedveld FC, Schiff MH, Kalden JR, Emery P, Eberl G, et al. A simplified disease activity index for rheumatoid arthritis for use in clinical practice. Rheumatology 2003;42:244-257.
- Steinbrocker O, Traeger CH, Batterman RC. Therapeutic criteria in rheumatoid arthritis. J Am Med Assoc. 1949;140(8):659-62.
- Van Gestel AM, Prevoo MLL, Hoff MA van't, Rijswijk MH van, Putte LBA van de, Riel PLCM van. Development and validation of the European League Against Rheumatism response criteria for rheumatoid arthritis. Arthritis Rheum 1996;39:34-40.
- Van Gestel AM, Haagsma, CJ, Riel PLCM vav. Validation of RA improvement criteria that include simplified joint counts. Arthritis Rheum 1998;41:1845-1850.
- Van der Heijde DM, Hof MA van't, Riel PL van, Theunisse LA, Lubberts EW, Leeuwen MA van, Rijswijk MH van, Putte LB van de. Judging disease activity in clinical practice in rheumatoid arthritis: first step in the development of a disease activity score. Ann Rheum Dis 1990;49:916-920.
- Ware JE. SF-36 Health Survey update. The Use of Psychological Testing for Treatment Planning and Outcomes Assessment. 2004;3:693-718.
- Wolfe F. Comparative usefulness of C-reactive protein and erythrocyte sedimentation rate in patients with rheumatoid arthritis. J Rheumatol 1997;24:1477-85.
- Actemra®, Drip Infusion, 80 mg, 200 mg, 400 mg, final reports on all-case surveillance. "Rheumatoid arthritis" "Active polyarticular juvenile idiopathic arthritis"
- Enbrel®, Drug Interview Form (Revised June 2013 Ver. 21)
- Orencia<sup>®</sup>, Drip Infusion, 250 mg, information regarding appropriate drug usage Vol. 4. Summary of final reports
- Cimzia Subcutaneous Injection 200 mg Syringe CTD, 2.7 Clinical Summary, 2.7.3 Summary of Clinical Efficacy, 2.7.3.2 Summary of Results of Individual Studies, 2.7.3.2.2 Comparison of Efficacy Results of All Studies, 2.7.3.2.2.1 Japanese Studies (1) Study CDP870-041, (2) Study RA0006 22-35 (2012)
- Simponi<sup>®</sup>, Drug Interview Form (September 2013 Ver. 5)
- Xeljanz<sup>®</sup>, Drug Interview Form (Revised July 2013 Ver. 3)
- Xeljanz<sup>®</sup> Tablets, 5 mg CTD, 2.7 Clinical Summary, 2.7.3 Summary of Clinical Efficacy, 2.7.3.3 Comparison of Results in Subpopulations, 2.7.3.3.1 Comparison of Japanese Population and Whole Population in Global Studies (Study No. A3921044) 123-139 (2013)

3 March 2017 Astellas 

- Xeljanz<sup>®</sup> Tablets, 5 mg CTD, 2.7 Clinical Summary, 2.7.4 Summary of Clinical Safety, 2.7.4.2 Adverse Events, 2.7.4.2.1.5.1.6 Serious Infections 150-153 (2013)
- Takeuchi T. [The significance of assessing the work productivity in the practice of rheumatoid arthritis For higher treatment goals–]. Rheumatology. 2011;46:288-296. Japanese.
- Tanaka Y. [New target molecules in treatment for rheumatoid arthritis Will signal-inhibiting low-molecular-weight compounds surpass biologics? –]. Inflammation and Immunity. 2009;17:214-218. Japanese.
- Nakajima A. [Drug therapy for rheumatoid arthritis: Indications, contraindications, and methods of use Antirheumatic drugs (DMARDs)]. Internal Medicine. 2009;103:655-659. Japanese.
- Japan Clinical Oncology Group (JCOG), Japanese Society of Clinical Oncology (JSCO). Common Terminology Criteria for Adverse Events (CTCAE) v4.0, Japanese translation, JCOG/JSCO Version: 1 February 2010. Available from: http://www.jcog.jp/index.htm
- Humira<sup>®</sup>, Drug Interview Form (Revised July 2013 Ver. 12)
- Humira<sup>®</sup>, Subcutaneous Injection, 40 mg, syringe 0.8 mL, information regarding appropriate drug usage Vol. 7. (Summary of final reports from 7,740 patients)
- Yamaoka K, Tanaka Y. [Rheumatoid arthritis treatment with Jak3 inhibitors]. Rheumatology. 2008;40:526-530. Japanese.

3 March 2017 Astellas 

## 12 APPENDICES

# APPENDIX <1>: LIST OF PROHIBITED CONCOMITANT MEDICATION

## ✓ Biologic DMARD (biological drugs for the treatment of RA)

Etanercept (except use as a reference drug), anakinra, adalimumab, golimumab, infliximab, tocilizumab, abatacept, certolizumab pegol, rituximab, denosumab

# ✓ Non-biologic DMARD\*

MTX, hydroxychloroquine, Salazosulfapyridine, gold, *D*-penicillamine, leflunomide, lobenzarit, actarit, tacrolimus, mizoribine, bucillamine, iguratimod, tofacitinib

\*: MTX, hydroxychloroquine, Salazosulfapyridine, gold, *D*-penicillamine, lobenzarit, actarit, bucillamine, or iguratimod can be administered concomitantly when subjects receive the drug at the same dosage and using the same administration schedule from 28 days prior to baseline to the end of treatment with the study drug or reference drug. Topical drugs other than those for the treatment of RA may be used concomitantly.

# ✓ Other drugs used in the treatment of RA

Cyclosporine, cyclophosphamide, azathioprine, minocycline, etc.

#### ✓ Corticosteroids\*\*

Prednisolone, hydrocortisone succinate, methylprednisolone, methylprednisolone succinate, triamcinolone, triamcinolone acetonide, dexamethasone, betamethasone, etc.

\*\*: Administration of corticosteroids at doses exceeding 10 mg/day in prednisolone equivalent is prohibited. Intra-articular, intravenous, intramuscular, or endorectal administration is prohibited. However, suppositories for anal disease may be used concomitantly.

#### ✓ Oral morphine\*\*\*

Morphine hydrochloride, morphine sulfate

\*\*\*: Oral morphine in doses exceeding 30 mg/day (or equivalent amount of opioid analgesic)

## ✓ CYP3A substrates with narrow therapeutic range

Dihydroergotamine, ergotamine, fentanyl, pimozide, quinidine, temsirolimus, disopyramide, etc.

## ✓ Live or live attenuated virus vaccines

Freeze-dried live attenuated measles vaccine, freeze-dried live attenuated mumps vaccine, freeze-dried BCG vaccine, freeze-dried live attenuated varicella vaccine, freeze-dried live attenuated rubella vaccine, live oral poliomyelitis vaccine, etc.

#### ✓ Articular cartilage protective agents

Purified sodium hyaluronate (intra-articular injection), chondroitin sulfate (excluding eye drops)

# APPENDIX <2>: LABORATORY TESTS

| | Visit | Collecting tube* [unique to Japan] | Parameters to be analyzed |
|---|---|---|---|
| Hematology | Screening, Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44, Week 48, Week 52, at early termination, follow-up, unscheduled | 2 mL vacutainer tube containing EDTA-2K | Hemoglobin,<br>hematocrit, RBC,<br>WBC, differential<br>WBC, platelet count |
| Biochemistry | Screening, Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44, Week 48, Week 52, at early termination, follow-up, unscheduled | 9 mL vacutainer tube containing the separating medium For glucose: 2 mL vacutainer tube containing NaF+EDTA-2Na For β-D-glucan: 3 mL container for blood endotoxin/β-D-glucan | Na, K, Ca, Cl, Mg, HCO <sub>3</sub> , BUN, phosphorus, glucose, creatinine, ALP, AST (GOT), ALT (GPT), γ-GTP, TBL, total protein, albumin, uric acid, CPK, LDH, serum amylase, eGFR, β-D-glucan |
| Biochemistry (at CPK monitoring) | At CPK monitoring | 4 mL vacutainer tube containing the separating medium | CK-MB, troponin-T, aldolase |
| Fasting lipid profile test | Baseline, Week 12, Week 20, Week 28, Week 40, Week 52, at early termination, follow-up, unscheduled | (Included among biochemistry tests) | Total cholesterol, LDL,<br>HDL, triglycerides |
| Tuberculosis test (When performed at the central laboratory) | Screening | 10 mL vacutainer tube containing heparin Na | Interferon γ titer |
| Hepatitis test | Screening | 6 mL vacutainer tube containing the separating medium | HBs antigens, HBs antibodies, HBc antibodies, and HCV antibodies |
| Hepatitis DNA test | Screening If a subject is positive for HBc antibodies or HBs antibodies, tests should be performed at the following visits: Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44, Week 48, Week 52, at early termination, follow-up, unscheduled | 5 mL vacutainer tube containing the separating medium | HBV-DNA assay |

| Urinalysis | Screening, Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44, Week 48, Week 52, at early termination, follow-up, unscheduled | For urinalysis: 10 mL light-blocking urine collection tubes For urine microscopic examination: 10 mL urine collection tubes | pH, specific gravity,<br>protein, glucose, keton<br>bodies, bilirubin, occult<br>blood, sediment |
|---|---|---|---|
| Pregnancy testing | Screening, Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44, Week 48, Week 52, at early termination, follow-up, unscheduled | Serum pregnancy test (Included among biochemistry tests) Urine pregnancy test (In-hospital testing) | Human chorionic<br>gonadotropin (hCG) |
| Acute phase reactants | Screening (CRP only), Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44, Week 48, Week 52, at early termination, follow-up, unscheduled | (Included among biochemistry tests) In-hospital testing | CRP<br>ESR |
| PK<br>(Assessment of trough<br>concentration) | Baseline, Week 4, Week<br>8, Week 12, Week 28,<br>Week 52, at early<br>termination | 2 mL vacutainer tubes<br>containing EDTA-3K | Concentrations of<br>ASP015K and its<br>metabolites H1, H2,<br>and H4 |
| Additional PK<br>(for post-dose<br>concentration) | Week 4 or Week 8 | 2 mL vacutainer tubes<br>containing EDTA-3K | Concentrations of<br>ASP015K and its<br>metabolites H1, H2,<br>and H4 |
| PD | Baseline, Week 4, Week 8, Week 12, Week 28, Week 52, at early termination, follow-up, unscheduled | 2 mL vacutainer tubes<br>containing EDTA-2Na<br>(MMP-3 is included<br>among biochemistry<br>tests.) | VEGF<br>MMP-3 |
| | Baseline, Week 4, Week 8, Week 12, Week 28, Week 52, at early termination, follow-up, unscheduled | 2 mL vacutainer tubes<br>containing EDTA-2K | Lymphocyte subset |
| Pharmacogenomics<br>(Only at approved study<br>centers) | After obtaining the subject's consent for PGx | 5 mL vacutainer tubes<br>containing EDTA-2K | PGx analysis |

<sup>\*:</sup> Types of collecting tube used at Korea and Taiwan are described in the laboratory handling manual.

3 March 2017 Astellas 

# APPENDIX <3>: EVENTS ALWAYS CONSIDERED SERIOUS

If any of the following events occurs during the study, it should be regarded as an SAE and must be reported in accordance with Section 5.5.5 Reporting of Serious Adverse Events (SAEs).

- Acute hepatic failure
- Renal failure acute
- Acute respiratory failure
- Agranulocytosis
- Anaphylactic reaction, anaphylactic shock
- Malignant tumor
- Aplastic anaemia
- Endotoxic shock (confirmed or suspected)
- Confirmed or suspected transmission of infectious agents by marketed product
- Congenital anomalies
- Hepatic necrosis
- Malignant hypertension
- Pulmonary fibrosis
- Pulmonary hypertension
- Sclerosing syndromes
- Convulsion (only central neurological seizure)
- Torsades de pointes
- Toxic epidermal necrolysis
- Ventricular fibrillation

Note: Hy's Law cases should be regarded as SAE.

See Appendix 4 "Liver Safety Monitoring and Assessment."

# APPENDIX <4>: LIVER SAFETY MONITORING AND ASSESSMENT

If laboratory testing for a subject enrolled in the study and receiving the study drug or reference drug reveals an increase in serum aminotransferase (ALT, AST)  $> 3 \times \text{ULN}$  or TBL  $> 2 \times \text{ULN}$ , the investigator/sub-investigator should repeat at least 4 parameters (ALT, AST, ALP, and TBL) of the usual hepatic function test parameters. Retesting should be performed between 48 hours and 72 hours after notification of the test results. For studies for which a central laboratory is used, alerts will be generated by the central laboratory regarding moderate and marked liver abnormality to inform the investigator or other responsible personnel and the sponsor. Subjects should be asked if they have any symptoms suggestive of hepatobiliary dysfunction by the investigator/sub-investigator.

# **Definition of Hepatic Function Abnormal**

Confirmed hepatic function abnormal will be characterized as moderate (hepatocellular failure type or cholestasis type) or marked (mixed type) based on the ULN as follows:

| | ALT or AST | | TBL |
|---|---|---|---|
| Moderate Hepatocellular failure type or cholestasis type | > 3 × ULN | or | > 2 × ULN |
| Marked<br>Mixed type | > 3 × ULN | and | > 2 × ULN |

In addition, the subject with any of the following should be considered to have marked (severe) hepatic function abnormal.

ALT or AST  $> 8 \times ULN$ 

ALT or AST  $> 5 \times ULN$  for more than 2 weeks

ALT or AST  $> 3 \times ULN$  and INR > 1.5

ALT or AST  $> 3 \times$  ULN with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, pyrexia, rash and/or eosinophilia (> 5%)

If the investigator/sub-investigator determines that abnormal liver function results, other than as described above, qualify as moderate or marked abnormalities, they should conduct additional monitoring and follow-up.

## **Follow-up Procedures**

Confirmed moderate and marked hepatic function abnormal should be thoroughly characterized by obtaining appropriate expert consultations, detailed pertinent history, physical examination and laboratory tests by the investigator/sub-investigator. The investigator should complete the liver abnormality case report form (LA-CRF) or an appropriate document. Subjects with confirmed abnormal liver function test results should be followed as described below by the investigator/sub-investigator.

If moderate liver abnormality is confirmed, re-testing should be performed every 2 to 3 times a week. If the abnormal test values stabilize or the patient is asymptomatic after the study drug or reference drug is withdrawn, re-testing should be performed at a frequency of once a week or less.

Marked hepatic function abnormal, in the absence of another etiology, may be considered an important medical event and reported as an SAE by the investigator. The sponsor should be contacted and informed of all subjects for whom marked hepatic function abnormal possibly attributable to study drug or reference drug is observed.

To further assess the findings of hepatic function abnormal, the investigator/sub-investigator is expected to:

Obtain a more detailed history of symptoms and prior or concurrent diseases. Symptoms and new onset-diseases should be recorded as "AEs" on the AE page of CRF. Illnesses and conditions such as hypotensive events, and decompensated cardiac disease that may lead to secondary liver abnormalities should be noted. Non-alcoholic steatohepatitis (NASH) is seen in obese hyperlipoproteinemic and/or diabetic patients and may be associated with fluctuating serum aminotransferase (ALT, AST) levels. The investigator/sub-investigator should ensure that the medical history form captures any illness that pre-dates study enrollment that may be relevant in assessing hepatic function.

Obtain a history of concomitant drug use (including non-prescription medication, complementary and alternative medications), alcohol intake, drug abuse, and special diets. Medications, including dose, should be entered on the concomitant medication page of CRF. Information on alcohol, other substance use, and diet should be entered into the LA-CRF or an appropriate document.

Obtain a history of exposure to environmental chemical agents.

Based on the subject's history, other testing may be appropriate including:

- Acute viral hepatitis subtypes (A, B, C, D, E, or other infectious agents)
- Ultrasound or other imaging to assess biliary tract disease
- Other laboratory tests including INR, direct bilirubin

Consider gastroenterology or hepatology consultations

Enter the results for any additional testing and possible etiology into the LA-CRF or an appropriate document.

#### **Study Discontinuation**

In the absence of an explanation for liver function test raised such as viral hepatitis, pre-existing or acute liver disease, or exposure to other agents associated with liver injury or when the investigator/sub-investigator determines that it is not in the subject's best interest to continue study enrollment, the subject may be discontinued from the study by the

#### Sponsor: Astellas Pharma Inc.


investigator/sub-investigator. Discontinuation of treatment with the study drug or reference drug should be considered if any of the following applies:

ALT or AST  $> 8 \times ULN$ 

ALT or AST  $> 5 \times ULN$  for more than 2 weeks

ALT or AST  $> 3 \times ULN$  and (TBL  $> 2 \times ULN$  or INR > 1.5)

ALT or AST  $> 3 \times$  ULN with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia (> 5%)

In addition, if close monitoring for a subject with moderate or marked hepatic function abnormal is not possible, the study drug or reference drug should be discontinued by the investigator.

#### Reference

See "Guidance for Industry on Drug-Induced Liver Injury: Premarketing Clinical Evaluation," published by the FDA in July 2009.

# APPENDIX <5>: 1987 ACR CRITERIA FOR THE CLASSIFICATION OF RA

For classification purposes, a patient shall be said to have RA if he/she has satisfied at least 4 of these 7 criteria. Criteria [1] through [4] must have been present for at least 6 weeks.

| Criterion | Definition |
|---|---|
| [1] Morning stiffness | Morning stiffness in and around the joints, lasting at least 1 hour |
| | before maximal improvement |
| [2] Arthritis of 3 or more joint | At least 3 joint areas simultaneously have had soft tissue swelling |
| areas | or fluid (not bony overgrowth alone) observed by a physician. The |
| | 14 possible areas are right or left PIP, MCP, wrist, elbow, knee, |
| | ankle, and MTP joints. |
| [3] Arthritis of hand joints | At least 1 area swollen (as defined above) in a wrist, MCP, or PIP |
| | joint |
| [4] Symmetric arthritis | Simultaneous involvement of the same joint areas (as defined in |
| | [2]) on both sides of the body (bilateral involvement of PIPs, |
| | MCPs, or MTPs is acceptable without absolute symmetry) |
| [5] Rheumatoid nodules | Subcutaneous nodules, over bony prominences, or extensor |
| | surfaces, or in juxtaarticular regions, observed by a physician |
| [6] Serum rheumatoid factor | Demonstration of abnormal amounts of serum rheumatoid factor by |
| | any method for which the result has been positive in $\leq 5\%$ of |
| | normal control subjects |
| [7] Radiographic changes | Radiographic changes typical of RA on posteroanterior hand and |
| | wrist radiographs, which must include erosions or unequivocal |
| | bony decalcification localized in or most marked adjacent to the |
| | involved joints (osteoarthritis changes alone do not qualify) |

[Armett FC et al, 1988]

3 March 2017 Astellas 

# APPENDIX <6>: 2010 ACR-EULAR CLASSIFICATION CRITERIA FOR RA

1. If a patient has at least 1 joint with synovitis not explained by another disease and scores  $\geq 6$  in the scoring system of 4 categories, he/she is assessed as having "definite RA."

| Joint involvement <sup>a)</sup> | |
|--------------------------------------------|---|
| 1 large joint <sup>b)</sup> | 0 |
| 2–10 large joints | 1 |
| 1–3 small joints <sup>c)</sup> | 2 |
| , | |
| 4–10 small joints | 3 |
| ≥ 11 joints (at least 1 small joint) | 5 |
| Serology | |
| RF8 (-) and anti-CCP antibody (-) | 0 |
| Low positive RF or low positive anti-CCP | 2 |
| antibody | |
| High positive RF or high positive anti-CCP | 3 |
| antibody | |
| (High: $> 3 \times ULN$ ) | |
| Acute phase reactants | |
| Normal CRP and normal ESR | 0 |
| Abnormal CRP or abnormal ESR | 1 |
| Duration of symptoms | |
| < 6 weeks | 0 |
| $\geq$ 6 weeks | 1 |

- a): The distal interphalangeal joints, first CMC joints, and first MTP joints are excluded from assessment.
- b): Large joints: Shoulder, elbow, hip, knee, and ankle joints
- c): Small joints: PIP joints, MCP joints, 2-5 MTP joints, first IP joints, and wrist joints

[Daniel A et al, 2010]

3 March 2017 Astellas 

Sponsor: Astellas Pharma Inc.


# APPENDIX <7>: CRITERIA FOR THE CLASSIFICATION OF GLOBAL FUNCTIONAL STATUS IN RA (1991 REVISED CRITERIA)

[Classification of Global Functional Status in RA: Class]

| Class I | Complete functional capacity with ability to carry on all usual duties without |
|---|---|
| | handicaps |
| Class II | Functional capacity adequate to conduct normal activities despite handicap or |
| | discomfort or limited mobility of one or more joints |
| Class III | Functional capacity adequate to perform only few or none of the duties of usual |
| | occupation or of self-care |
| Class IV | Largely or wholly incapacitated with patient bedridden or confined to wheelchair, |
| | permitting little or no self-care |

[Hochberg et al, 1992]

# APPENDIX <8>: CLASSIFICATION OF DISEASE STAGE/PROGRESSION OF RA

| Stage I: Early | 1 | X-rays show no evidence of bone destruction. |
|---|---|---|
| | 2 | X-rays may show radiological osteoporosis. |
| Stage II: | 1. | X-rays show osteoporosis which may or may not be accompanied |
| Intermediate | | by mild destruction of subchondral bone. Mild bone destruction may be observed. |
| | 2. | Joint mobility may be limited, but there is no joint deformation. |
| | 3. | Muscle atrophy surrounding the joint is present. |
| | 4. | Lesions in extra-articular soft tissue, such as nodules and tenosynovitis, may be present. |
| Stage III: Advanced/<br>Progressive | 1. | In addition to osteoporosis, X-rays show destruction of bone and cartilage. |
| | 2. | Joint deformities such as subluxation, ulnar displacement, or hyperextension are present, unaccompanied by fibrous or bony ankylosis. |
| | 3. | Exaggerated muscle atrophy is present. |
| | 4. | Lesions in extra-articular soft tissue, such as nodules and |
| | | tenosynovitis, may be present. |
| Stage IV: End Stage | 1. | Fibrous or bony ankylosis is present. |
| | 2. | Other symptoms meet criteria for Stage III. |

[Steinbrocker O. 1949]

(GPF 3.03)